

## STATISTICAL ANALYSIS PLAN

| Title | INAS-VIPOS International Active Surveillance Study of Medication Used for the Treatment of Endometriosis: Visanne Post-approval Observational Study |
|---|---|
| Protocol version | VIPOS Study Protocol,<br>2 <sup>nd</sup> revision of Nov. 21, 2011 |
| Active substance | Dienogest |
| Medicinal product | Visanne 2 mg |
| Marketing authorization holder | Bayer AG<br>13342 Berlin<br>Germany |
| Author | Kerstin Becker ZEG – Berlin Center for Epidemiology and Health Research Invalidenstraße 115 10115 Berlin Germany |

Submitted with the final report on June 04, 2019

ClinicalTrials.gov Identifier: NCT01266421

| 1. | INTRODUCTION | 6 |
|-----|-----------------------------------------------------|----|
| 1.1 | RATIONALE AND BACKGROUND | 6 |
| 1.2 | RESEARCH QUESTION AND OBJECTIVE | 6 |
| 1.3 | PROTOCOL VERSION AND AMENDMENTS | 6 |
| 2. | STUDY OBJECTIVES | 6 |
| 3. | STUDY DESIGN | 7 |
| 3.1 | STUDY POPULATION, INCLUSION AND EXCLUSION CRITERIA | 8 |
| 3.2 | STUDY FLOW CHART | 9 |
| 3.3 | STUDY VARIABLES | 10 |
| 4. | POWER AND SAMPLE SIZE | 11 |
| 5. | STATISTICAL METHODOLOGY | 14 |
| 5.1 | Analysis sets | 14 |
| 5.2 | Hypothesis | 15 |
| 5.3 | Analysis of population characteristics | 16 |
| 5.3 | 3.1 Descriptive statistics | 16 |
| 5.3 | 3.2 Stratifying factors | 16 |
| 5.4 | ANALYSIS OF PRIMARY AND SECONDARY OUTCOME VARIABLES | 17 |
| 5.4 | 4.1 Incidence measures | 17 |
| 5.4 | 4.2 Regression models | 18 |
| 5 | 5.4.2.1 Cox Proportional Hazard Model | |
| | 4.3 Definition of primary outcomes | |
| | 4.4 Definition of secondary outcomes | |
| | 4.5 Definition of other safety outcomes | |
| | 4.6 Definition of other outcomes of interest | |
| 5.5 | MISSING DATA | |
| 6. | DATA HANDLING | |
| 6.1 | | |
| | Variable definitions | |
| | 2.1 Definition of derived variables | |
| 6.2 | 2.2 Definition of subgroups | 21 |
| 7. | INTERIM ANALYSES AND DATA MONITORING | 22 |
| 7.1 | Data Monitoring | 22 |
| 7.2 | INTERIM ANALYSIS | 22 |
| 8. | STRUCTURE OF THE ANALYSIS TABLES | 22 |
| 9. | REFERENCES | 26 |
| 10. | APPENDIX | 27 |
| I E | BASELINE QUESTIONNAIRE | 27 |



Supporting document SOP BMT 01.09 – Doc 5002.02 – Effective date 21.03.2017

| II | FOLLOW-UP QUESTIONNAIRE | . 31 |
|-----|-----------------------------------------------------------|------|
| Ш | LIST OF POTENTIAL PROGNOSTIC FACTORS FOR PRIMARY OUTCOMES | . 33 |
| IV | LIST OF DERIVED VARIABLES | . 34 |
| Mod | CK TABLES | . 35 |



Supporting document SOP BMT 01.09 – Doc 5002.02 – Effective date 21.03.2017

#### **Abbreviations**

| ADB | Administrative Database |
|---|---|
| ADR | Adverse Drug Reaction |
| AT | As Treated |
| ATE | Arterial Thromboembolism |
| ATC | Anatomical Therapeutic Chemical Classification System |
| СНС | Combined Hormonal Contraceptives |
| CI | Confidence Interval |
| DIMDI | German Institute for Medical Documentation and Information |
| EMT | Endometriosis treatment |
| EURAS | EURopean Active Surveillance (study) |
| FU | Follow-up |
| GP | General Practitioner |
| НСР | Health Care Professional |
| HR | Hazard Ratio |
| ICD-10 | International Classification of Diseases, 10th revision |
| IP | Incidence Proportion |
| IR | Incidence Rate |
| IRR | Incidence Rate Ratio |
| ITT | Intention to Treat |
| LOCF | Last observation carrying forward |
| NAED | Not approved hormonal medications for the treatment of endometriosis |
| OAED | Other approved hormonal medications for the treatment of endometriosis |
| OR | Odds Ratio |
| Р | Prevalence |
| SAE | Serious Adverse Event |
| SAP | Statistical Analysis Plan |
| SDB | Study Database |
| SMAC | Safety Monitoring and Advisory Council |
| VTE | Venous Thromboembolism |
| WHO | World Health Organization |
| WY | Women years |
| ZEG | Berlin Center for Epidemiology & Health Research (acronym for the German term 'Zentrum für Epidemiologie & Gesundheitsforschung Berlin') |



Supporting document SOP BMT 01.09 - Doc 5002.02 - Effective date 21.03.2017

#### 1. Introduction

This document describes the Statistical Analysis Plan (SAP) for the "International Active Surveillance Study of Medication Used for the Treatment of Endometriosis, the **Vi**sanne **P**ost-approval **O**bservational **S**tudy". To enhance understanding and to follow the guidelines proposed by the European Network of Centers for Pharmacoepidemiology and Pharmacovigilance (ENCePP), this SAP will also reflect parts of the study protocol.

#### 1.1 Rationale and background

Dienogest (DNG) is a 19-nortestosterone derivative progestogen that is highly selective for progesterone receptors [1]. As a progestin in DNG/EE, DNG is known for having strong endometrial effects that improve dysmenorrhea and decrease the duration of menstrual bleeding [2]. In addition, progestogens may also modulate pain associated with endometriosis by dampening neuronal activity [3]. It is not known what influence DNG will have on bleeding disturbances associated with endometriosis over a longer time frame or the potential influence of DNG on mood disturbance and depression in endometriosis patients.

#### 1.2 Research question and objective

The primary objective of the study is to assess safety aspects of Dienogest 2 mg/day (Visanne®) used as endometriosis therapy and of other hormonal treatments for endometriosis in a study population that is representative for the actual users of the individual preparations. This includes an estimate of the absolute risk of rare serious adverse outcomes.

#### 1.3 Protocol version and amendments

INAS-VIPOS – Final study protocol, 2<sup>nd</sup> revision of Nov. 21, 2011.

Study Protocol, Amendment of September 30, 2017.

#### 2. Study Objectives

The main clinical outcomes of interest for the short and long-term follow-up are:

- Medical intervention for anemia induced by cyclical bleeding disturbances (anemia)<sup>1</sup>
- · First-time occurrence of clinically relevant depression, or worsening of existing depression
- To analyze discontinuation patterns of DNG and other endometriosis treatments due to treatment failure<sup>2</sup>.

<sup>1</sup> For the purposes of this SAP, this will be referred to as "anemia" for the remainder of the document. The definition for validation of "anemia" is given in Section 5.4.3

<sup>2 &#</sup>x27;Treatment failure' is defined as cessation of treatment caused by lack of efficacy, loss of efficacy or an adverse drug reaction and does not include women who stop treatment after pre-defined treatment periods (e.g. after six months for GnRH agonists). In addition, combined



Supporting document SOP BMT 01.09 – Doc 5002.02 – Effective date 21.03.2017

#### Secondary objectives are:

- To characterize the baseline risk of users of the individual formulations (lifetime history of co-morbidity, risk markers, co-medication, socio-demographic and lifestyle data).
- To analyze the drug utilization pattern of DNG and other endometriosis treatments in a study population that is representative for typical use of the individual preparations under routine medical conditions.
- To investigate the risks of short and long-term use of DNG and of established endometriosis treatments in adolescent women.

#### 3. Study Design

This is a large, prospective, controlled, non-interventional, long-term cohort study which follows two cohorts, users of DNG and users of other medications used for the treatment of endometriosis<sup>3</sup>. The cohorts consist of new users (starter<sup>4</sup> and restarter<sup>5</sup>) or switcher<sup>6</sup> of a hormonal endometriosis treatment. A "non-interference" approach will be used to provide standardized, comprehensive, reliable information on endometriosis treatment patterns.

A follow-up assessment for each woman is scheduled 6, 12, 24, 36 and depending on the date of enrollment 48, 60, 72 and 84 months after baseline. Women will be followed-up for at least 2 years. Women recruited in the early phase of the study will be followed-up until study endpoint [max. 7 years]<sup>7</sup>. By means of these contacts, almost all relevant clinical outcomes will be captured.

However, during the first year of the study, less than 15% of the planned recruitment target within that time frame was achieved (i.e. 1,191 women were recruited rather than the anticipated 8,334 women). As a consequence, the overall recruitment phase was longer (and therefore the observation time was less) than we had expected. In order to achieve the envisaged total observation time of 84,000 women years, the follow-up period will be prolonged by one year (until end of QII 2018)<sup>6</sup>.

All clinically relevant serious adverse events will be verified by ZEG through contact with the relevant physicians and by reviewing pertinent source documentation. A standard algorithm will be used to classify 'clinically relevant depression' and 'medically treated anemia' as 'confirmed' or 'not confirmed'. At the end of the study, this classification will be verified by blinded independent adjudication

treatment with GnRH, an estrogen and/or a progestogen (add-back therapy) will be considered as a single treatment regimen. In cases where add-back therapy is used the predefined end-point is the cessation of the add-back therapy.

<sup>3</sup> Users of non-approved hormonal medications prescribed for endometriosis treatment are additionally followed up and included in the analysis.

<sup>4</sup> First ever user of EMT

<sup>5</sup> EMT use after intake break (>= 4 weeks)

<sup>6</sup> Switching from another EMT

<sup>7</sup> According Study Protocol, Amendment of September 30, 2017



Supporting document SOP BMT 01.09 - Doc 5002.02 - Effective date 21.03.2017

#### 3.1 Study population, inclusion and exclusion criteria

It was planned to implement the study in several European countries including, but not necessarily limited to, Germany, Austria, France, and Poland. However, the study was initiated in Germany in 2010, and in Hungary and Poland in early 2011. Because of recruitment problems, additional countries were included to broaden the recruitment base: Ukraine, Russia, and Switzerland started recruitment in 2012.

Recruitment of the cohort members will be conducted via a network of approximately 1,000 physicians (study centers) managing women with a diagnosis of endometriosis. The combined cohort will include 25,000 women <sup>8</sup>.

At the participating centers, all women prescribed a new treatment for endometriosis are to be asked by their physician if they are willing to participate. The physician is to explain the nature of the study, its purpose and associated procedures, and the expected duration of follow-up for each woman prior to her study entry. Each woman is to have ample opportunity to ask questions and must be informed about her right to withdraw from the study at any time without disadvantage and without having to provide reasons for her decision. This information will be provided on an informed consent and data privacy form which must be signed by all study participants. These documents are to be approved by the relevant local Ethics Committees and the relevant Data Privacy Office, if applicable.

Once enrolled, a subject may discontinue use of the relevant medication at any time. However, subjects will continue to be followed whether or not they remain on their treatment for endometriosis, provided that they do not withdraw their consent. During the follow-up phase, subjects will be asked whether they have discontinued their treatment or whether they have switched to another medication or received surgical treatment to manage their endometriosis. Information on the date and reason for discontinuation or switching during the follow-up phase will also be collected.

The study participants are women who

- are users of a newly prescribed regimen for endometriosis (starter, switcher or restarter)
- are willing to participate in this long-term follow-up study.

There are no specific medical inclusion or exclusion criteria. However, women

- who are not cooperative/available for follow-up may be excluded from study participation
- women with a language barrier will not be eligible for study inclusion.

The study flowchart (section 3.2) provides an overview of all study phases.

<sup>8</sup> At the end of recruitment in June 2014 the number of OED patients was much lower than the anticipated share of 10% of the study population. The SMAC recommend therefore to re-start recruitment for 2,000 OAED patients.



Supporting document SOP BMT 01.09 - Doc 5002.02 - Effective date 21.03.2017

#### 3.2 Study Flow Chart

Recruitment: 6 European countries (Germany, Poland, Russia, Hungary, Switzerland, Ukraine)

Indication: Starter, restarter and switcher initiating a new treatment for endometriosis and

willing to participate

Recruitment time: approx. 58 months (end of 2010 – June 2014; spring 2015 – June 2016)

Phase I: BASELINE SURVEY

Baseline Questionnaire:

Physician/Patient

DNG

(DNG 2mg/day)

OAED

- 1) GnRH-a
- 2) Danazol

NAED

- 1) Combined contraceptives (CC)
- 2) Other progestins
- 3) Any other non-approved hormonal medication for endometriosis or those approved only in some participating countries

Phase II: FOLLOW-UP

FU-Questionnaire: Patient

FU 1: 6 months
FU 2 up to FU 8: on annual basis

Sample: AT/ITT

Objectives: Primary and secondary outcomes

Validation of *self-reported* outcomes of interest:

- 1. Contact treating HCP, review relevant source documents
- 2. Classification: confirmed / not confirmed by ZEG physicians
- 3. Verification by blinded independent adjudication (anemia/depression)

#### **END OF OBSERVATION**

- 1. End of FU (i.e. end of study)
- 2. Drop-out (e.g., withdrawal of informed consent)
- 3. Loss to Follow-up

Supporting document SOP BMT 01.09 – Doc 5002.02 – Effective date 21.03.2017

## 3.3 Study variables

Table 1: Schedule of assessments and variables obtained during study phases.

| | Ph | ase I | Phase II |
|---|---|---|---|
| | Baseline | | FU 1 |
| | Dd | seille | up to FU 8 |
| | Physician | Patient | Patient |
| Informed consent | | Before any procedure | |
| Patient characteristics | | | |
| - Age of women | | x | |
| - Height | | | |
| - Weight | | v | v |
| - BMI | | X | X |
| Socio-economic characteristics | | | |
| - Education | | x | |
| - Smoking | | | |
| Endometriosis treatment | X | | |
| - Diagnosis classification | ^ | | |
| <ul> <li>Prescribed medication</li> </ul> | | | |
| <ul> <li>Number of surgical procedures (related to</li> </ul> | x | | x |
| endometriosis) | | | |
| <ul> <li>Reasons for switching / stopping treatment</li> </ul> | | | х |
| Endometriosis characteristics | | | |
| <ul> <li>Endometriosis pattern (symptoms, first</li> </ul> | | x | |
| diagnosis, treatment history, pain) | | | |
| <ul> <li>Surgical procedures related to endometriosis</li> </ul> | | Х | Х |
| Gynecological History | | | |
| <ul> <li>Age at first menarche</li> </ul> | | x | |
| <ul> <li>Pregnancies/deliveries</li> </ul> | | | |
| Medical history | | | |
| - Diseases / conditions | | v | |
| <ul> <li>Surgical procedures (other than</li> </ul> | | X | |
| endometriosis-related) | | | |
| Family history | | v | |
| (Endometriosis, Depression, VTE) | | Х | |
| Medication | | х | Х |
| Anemia | | х | Х |
| Depression | | х | Х |
| Mood | | Х | Х |
| Serious Adverse events | | | Х |

### 4. Power and Sample Size

The 2 to 7-year follow-up of more than 25,000 women should result in approximately 89,000 documented women-years. This estimate is based on the assumptions that (1) ZEG's physicians' network could recruit 25,000 women within three years, and (2) the annual drop-out rate is 10% (based on the EURAS-OC [4] and LASS studies). Details are provided in Table 1 and are based on the assumption that the follow-up period is a maximum of 6 years<sup>9</sup>.

**Table 1:** Expected observation time (max. 6 years follow-up): Patient recruitment within 3 years (annual recruitment rate = 8,334 women)

| | Sub-cohorts recruited during the | | | | | |
|---|---|---|---|---|---|---|
| | 1 <sup>st</sup> study year | | 2 <sup>nd</sup> study year | | 3 <sup>rd</sup> study year | |
| Time (y)* | No. of women | Time of observation | No. of<br>women | Time of observation | No. of<br>women | Time of observation |
| 1 | 7,910 | 4,035 | | | | |
| 2 | 7,119 | 7,515 | 7,910 | 4,035 | | |
| 3 | 6,407 | 6,763 | 7,119 | 7,515 | 7,910 | 4,035 |
| 4 | 5,766 | 6,087 | 6,407 | 6,763 | 7,119 | 7,515 |
| 5 | 5,190 | 5,478 | 5,766 | 6,087 | 6,407 | 6,763 |
| 6 | 4,671 | 4,930 | 5,190 | 5,478 | 5,766 | 6,087 |
| WY (total) | | 34,808 | | 29,878 | | 24,400 |
| WY<br>(grand total) | 89,086 | | | | | |

<sup>\*</sup> Time after start of recruitment

The study was designed to analyze rare events (according to the CIOMS classification 1-10 and less than 1 event(s) per 10,000 women-years, respectively). The adverse events of particular interest for the sample size calculations are anemia, clinically relevant depression and treatment failure.

The background prevalence of anemia in premenopausal European women is approximately 10-15% [5]. Based on this high prevalence and the fluctuating character of the disease the investigators anticipate an incidence of new or recurrent anemia in an active surveillance study of 0.01-0.02. The sample size calculation is based on a conservative estimate of 0.01 (or 1 event per 100 WY).

A conservative estimate of the prevalence rate for depression in women with endometriosis is 20%. This figure is based on a systematic literature review of the available evidence and an analysis of EURAS/INAS results. For newly diagnosed or worsening depression the expected incidence rate is at least 0.01. Based on this incidence, the sample size outlined below was calculated; in case the study

11

<sup>\*\*</sup> The number of recruited women equals 8,334. However, the number of women at the end of the first year is lower because some women will drop out during the first year (daily drop-out rate is ~ 0.029%).

 $<sup>{\</sup>bf 9}$  According Study Protocol, Amendment of September 30, 2017



Supporting document SOP BMT 01.09 – Doc 5002.02 – Effective date 21.03.2017

shows other incidence rates at a later point in time, a re-calculation may be necessary and will be discussed with the Safety Monitoring and Advisory Council if required.

Based on the natural history of endometriosis treatment, we anticipate that the majority of women will stop or change treatment regimen during the course of this study. We expect an incidence rate of women ceasing or changing treatment ('treatment failure') for other endometriosis medications due to lack of efficacy, loss of efficacy or an adverse drug reaction of at least 0.3. For the DNG cohort, a proportion of 0.25 of the total study population seems to be realistic.

Overall, 3 hypotheses will be tested (cf. section 11). The problem of <u>multiple comparisons</u> is addressed by using Bonferroni-Holm correction to maintain the <u>overall</u> error rate by testing each individual hypothesis at a <u>statistical significance</u> level of 1/3 times what it would be if only one hypothesis were tested (i.e., the individual tests will be based on an  $\alpha$  level of 0.0167 instead of 0.05).

Power calculations based on the incidences given above showed that approximately 84,000 womenyears would be needed to show non-inferiority of DNG versus other endometriosis medications for anemia. The calculations for anemia are based on the assumptions given in Table 2. In essence, the study is powered to exclude a two-fold risk of anemia for the DNG with at least 10% of the total exposure – if the true risk of anemia is not different for the relevant sub-cohorts.

**Table 2:** Power calculation [6] for anemia based on the assumption that the true incidence of DNG cohort is not different from other endometriosis medications (reference cohort)

| Test significance level, α (one-sided) | 0.0083 (= 0.0167 two-sided) |
|---|---|
| Anemia Incidence for reference cohort | 0.01 |
| Non-inferiority margin | 0.01 (equal to the anemia incidence for the reference cohort) |
| Expected anemia incidence for DNG cohort | 0.01 |
| Power (%) | 90 |
| Proportion of DNG users (% of study population) | 10 |
| Proportion of reference users (% of study population) | 5 |
| Required women-years in DNG cohort | 8,400 |
| Required women-years in reference cohort | 4,200 |
| Total women years | 84,000 |

Furthermore, 84,000 WY would be sufficient to also exclude a two-fold risk of clinically relevant depression (cf. Table 3), assuming that DNG accounts for at least 10% of the total exposure.



Supporting document SOP BMT 01.09 – Doc 5002.02 – Effective date 21.03.2017

For 'treatment failure' approximately 29,500WY will be required to show that DNG is superior to other endometriosis medications (cf. Table 4), assuming that the proportion of DNG, danazol, and GnRH agonists users each account for 10% of the total exposure.

**Table 3:** Power calculation [6] for depression based on the assumption that the true incidence in the DNG cohort is not different from the reference cohort

| Test significance level, $\alpha$ (one-sided) | 0.0083 (= 0.0167 two-sided) |
|---|---|
| Depression Incidence for reference cohort | 0.01 |
| Non-inferiority margin | 0.01 (equal to the depression incidence for the reference cohort) |
| Expected depression incidence for DNG cohort | 0.01 |
| Power (%) | 90 |
| Proportion of DNG users (% of study population) | 10 |
| Proportion of reference users (% of study population) | 5 |
| Required women-years in DNG cohort | 8,400 |
| Required women-years in reference cohort | 4,200 |
| Total women years | 84,000 |



Supporting document SOP BMT 01.09 – Doc 5002.02 – Effective date 21.03.2017

**Table 4:** Power calculation [6] for 'treatment failure' based on the assumption that the true incidence in the DNG cohort is ~ 2,500/10,000 compared to ~ 3,000/10,000 in the other endometriosis medications cohort.

| Test significance level, α (one-sided) | 0.0167 |
|---|---|
| Incidence of treatment failure for other endometriosis medications cohort | 0.30 |
| Clinically relevant difference | 0.05 |
| Expected incidence of treatment failure for DNG cohort | 0.25 |
| Power (%) | 90 |
| Proportion of DNG users (% of study population) | 10 |
| Proportion of reference users (% of study population) | 5 |
| Required women-years in DNG cohort | 2,950 |
| Required women-years in other endometriosis medications cohort | 1,475 |
| Total women years | 29,500 |

These power calculations suggest that this study is sufficiently powered to show non-inferiority of DNG compared to established endometriosis treatments with regard to anemia and clinically relevant depression, as well as superiority with regards to 'treatment failure'.

### 5. Statistical Methodology

Three primary outcomes of interest, anemia, depression and treatment failure, will be analyzed using inferential statistics. Statistical evaluation will be performed with the most current release version of the software package SAS® [7]

#### 5.1 Analysis sets

There are no specific inclusion or exclusion criteria. However, women with a language barrier, a non-hormonal or not newly prescribed baseline medication or women who are pregnant at study enrollment will be excluded from the analysis. The final analyses will include both an "as treated" (AT) and an "intention-to-treat" (ITT) analysis. All women who are not excluded from the analysis will be assigned to the ITT and AT population at baseline. Only women with follow up information will be considered for longitudinal analysis (e.g. distribution of outcomes over time, incidence rates, regression). Women who never started their prescribed baseline medication will be considered in the ITT analysis, but excluded from the AT analysis. The safety conclusions of the study will be based on the AT analysis.



Supporting document SOP BMT 01.09 – Doc 5002.02 – Effective date 21.03.2017

This study follows three cohorts: users of Visanne (DNG), users of other medication approved for the treatment of endometriosis (OAED) and users of non-approved hormonal medications prescribed for endometriosis treatment or those approved only in some participating countries (NAED).

Distribution of women, population characteristics (baseline and follow up) as well as clinical outcomes will be presented for the following cohorts and sub-categories.

| Cohort Sub-category for presentation | |
|---|---|
| DNG | Complete cohort |
| OAED | GnRH-a, Danazol, complete cohort |
| NAED | Combined hormonal contraceptives, other progestins, complete |

The cohorts consist of new users (starter and restarter) or switcher of a hormonal endometriosis treatment. For the primary analysis, outcomes of interest or adverse events will be assigned to the treatment at the time the outcome or the event occurred. Women with multiple exposure or unspecific treatment will be specified as "Allocation unknown". Women who stopped their treatment will be assigned to an "Ex-use" cohort.

### 5.2 Hypothesis

Based on available data and pharmacological/pharmacokinetic considerations the a priori assumption is that use of DNG is not associated with an increased risk of anemia compared to approved hormonal medications used in the treatment of endometriosis ("endometriosis medications"). It is probable that statistical comparisons of DNG vs. other endometriosis medications will not show a difference. Therefore, a non-inferiority design to investigate the anemia risk of DNG had been chosen. The analysis will be based on the comparison of the upper confidence limit for the point estimate of the anemia hazard ratio with the predefined non-inferiority margin (cf. section 4).

 $H_0$  and  $H_A$  denote the null and alternative hypotheses, respectively.  $HR_{Anemia}$  is defined as the hazard ratio for anemia for DNG vs. OAED.

$$H_0: HR_{Anemia} \geq 2$$

$$H_A$$
:  $HR_{Anemia} < 2$ 

For clinically relevant depression (first episode or worsening), the a priori assumption is that no approved treatment for endometriosis is associated with a higher risk of depression compared with untreated endometriosis. A non-inferiority design has been chosen, with primary analysis based on the comparison of the upper confidence limit for the point estimate of the depression hazard ratio with the predefined non-inferiority limit (cf. section 4).  $HR_{Depression}$  is defined as the hazard ratio for depression (newly diagnosed or worsening) for DNG vs. OAED

$$H_0: HR_{Depression} \geq 2$$

$$H_A: HR_{Depression} < 2$$



Supporting document SOP BMT 01.09 – Doc 5002.02 – Effective date 21.03.2017

There are both pharmacological and clinical indications that suggest that DNG may be superior to other endometriosis medications as a long-term treatment for endometriosis. That is, a statistical comparison of DNG vs. other endometriosis medications may show a difference in 'treatment failure', with DNG users continuing on treatment for longer periods of time. 'Treatment failure' is defined as cessation of treatment caused by lack of efficacy, loss of efficacy or an adverse drug reaction and does not include women who stop treatment after pre-defined treatment periods (e.g. after six months for GnRH agonists). In addition, combined treatment with GnRH, an estrogen and/or a progestogen (add-back therapy) will be considered as a single treatment regimen. In cases where add-back therapy is used the predefined end-point is the cessation of the add-back therapy. A superiority design to investigate 'treatment failure' for DNG has been chosen. The analysis will be based on a 5%-point difference (difference of 0.05) of DNG vs. other endometriosis medications.  $OR_{TreatmentFailure}$  is defined as the odds ratio for 'treatment failure' for DNG vs. OAED.

 $H_0: OR_{TreatmentFailure} \ge 1$ 

 $H_A: OR_{Treatmentfailure} < 1$ 

#### 5.3 Analysis of population characteristics

#### 5.3.1 Descriptive statistics

All background data such as patient characteristics, socio-economic characteristics, endometriosis pattern and gynecological history, family and medical history, concomitant medication as well as mood will be described by presenting frequency distributions and/or basic summary statistics (number of patients with an observation [n], mean, standard deviation [SD], median, 25th [Q1] and 75th [Q3] percentiles, minimum [Min] and maximum [Max]). Unless otherwise specified, the mean and median for a continuous variable will be listed to 1 more decimal place than the original (raw) values and the SD will be listed to 2 more decimal places than the original values. The minimum and maximum will be listed to the same number of decimal places as the original values.

Categorical variables will be summarized using frequencies and percentages. Each table will list both absolute and relative numbers (%), providing the total amount of available data for each variable. Total number of women (100%) for the presented (sub-) population is given in the first line of each table. Additional categories may be derived from data and are denoted by <<CATEGORY>> in the table templates. Percentages will be listed to 2 decimal places. In cases where the percentage calculated is > 0% and < 0.01%, three decimal places will be listed with the absolute value.

In addition, age-standardized proportions are presented for selected baseline characteristics, history of co-morbidity, risk markers and co-medication. Therefore, the most represented cohort will used as the referenced standard population.

#### 5.3.2 Stratifying factors

The numbers of patients enrolled and included in the analysis populations will be tabulated by defined stratifying variables for the AT and ITT population, if appropriate.

Baseline and follow-up population characteristics will be presented for the AT and ITT population and stratified by



Supporting document SOP BMT 01.09 - Doc 5002.02 - Effective date 21.03.2017

- (1) Country
- (2) EMT user type: starter vs. switcher vs. restarter
- (3) Diagnostic classification: Diagnosis confirmed by surgery vs. diagnosis based on clinical symptoms,

if not otherwise specified.

The analysis of the primary and secondary outcomes will be presented for the AT population, anemia and depression additionally for the ITT population. Primary and secondary outcomes are stratified by subgroups if appropriate:

- (1) Country
- (2) EMT user type: starter vs. switcher vs. restarter
- (3) Diagnostic classification: Diagnosis confirmed by surgery vs. diagnosis based on clinical symptoms

Selected outcomes regarding the baseline risk (lifetime history of co-morbidity, risk markers, co-medication, socio-demographic and lifestyle data), will be additionally displayed by subgroups as follows:

- (1) Age categories: < 20 vs. 20 to < 30 vs. 30 to < 40 vs. >= 40
- (2) Age standardized

Additional subgroups will be added for selected outcomes if appropriate.

#### 5.4 Analysis of primary and secondary outcome variables

The primary outcome (anemia, depression, treatment failure), secondary outcomes (risk factors, treatment pattern) as well as other safety outcomes (SAEs) and other outcomes of interest (surgeries) associated with the use of DNG, OAED and NAED will be assessed using different measurements as defined by Rothman et al. [8].

#### 5.4.1 Incidence measures

The *incidence rate* (IR) measures the occurrence of new cases per unit of person-time.

$$IR = \frac{Number\ of\ new\ cases}{Total\ follow - up\ time}$$

The incidence rate takes into consideration the patient-specific follow-up time and it assumes a constant hazard rate. For each of n subjects the time  $t_k (k=1,...,K)$  to: (1) the end of the risk period, if recurrent events are allowed or (2) to the first occurrence of a certain event is observed. If the event was not experienced, the (censored) time to the end of the risk period is observed.

In the present study, women-years are conducted as a unit of person-time. Incidence rates are shown per 10<sup>4</sup> women-years (WY) unless otherwise specified.

The *incidence rate ratio* (IRR) is the proportion of two incidence rate estimates.

$$IRR = \frac{Incidence\ rate\ of\ treatment\ group}{Incidence\ rate\ of\ control\ group}$$



Supporting document SOP BMT 01.09 - Doc 5002.02 - Effective date 21.03.2017

The incidence rate ratio gives a measure of how much more likely an event occurs in subjects under exposure (treatment group) than in subjects who were not exposed (control group).

The *incidence proportion* (IP) measures the occurrence of new cases in relation to the size of the population at risk within a given period of time (cumulative incidence).

$$IP = \frac{Number\ of\ new\ cases}{Size\ of\ population\ at\ risk}$$

Exact 95% confidence intervals for prevalence, incidence proportion, incidence rate, and incidence rate ratio will be calculated in accordance with Clopper and Pearson[9].

#### 5.4.2 Regression models

Regression analysis will be performed if a sufficient number of confirmed events are available for estimation, i.e. n≥5 confirmed events in each of the comparison groups.

Potential confounders such as

- age, personal and family history of depression, history of anemia, history of bleeding disorders and severity of pain will be included as time-invariant cofactors.
- EMT user type at follow up, use of Antidepressants/SSRI and current or worsening depression (primary outcome) will be included as time-dependent cofactors.

For each primary outcome, a summary table with predefined potential prognostic factors and the corresponding relative risk estimators is provided.

The final decision on the confounding variables will be made by the Safety Monitoring and Advisory Council:

| Primary outcome variable | Predefined Prognostic Factors <sup>10</sup> |
|---|---|
| Anemia | Age, history of anemia, history of bleeding disorders |
| Depression | Age, family and personal history of depression, use of Antidepressants/SSRI |
| Treatment Failure | Age, family and personal history of depression, severity of pain |

#### 5.4.2.1 Cox Proportional Hazard Model

Time-to-event (survival) analyses will be undertaken using Cox proportional hazard models (Cox model) to describe how the hazard increases for each unit increase of the regressor variables. Crude and adjusted hazard ratios (HR) comparing subpopulations under study will be calculated for all primary outcomes and 95% HR confidence limits (Wald) are provided. The crude model refers to a univariable model which includes exposure as the only explanatory factor. Potential predefined event-specific prognostic factors (section 5.4.2) are included in multiple models. In the Cox model, recurrent events are included.

18

<sup>10</sup> See Appendix III for all potential prognostic factors for each primary and secondary outcome.



Supporting document SOP BMT 01.09 - Doc 5002.02 - Effective date 21.03.2017

#### 5.4.3 Definition of primary outcomes

#### Anemia

Confirmed cases of anemia (clinically relevant) is defined as:

- 1. Confirmed by a repeated reliable laboratory test (e.g. hemoglobin, packed cell volume), plus pertinent therapy (blood or iron transfusion, iron tablets) or
- 2. No reliable laboratory data available, but clinical diagnosis stated by a physician, followed by pertinent therapy (see above) and
- 3. No obvious explanation (such as gastrointestinal bleeding, trauma, major surgery) or no explanation other than endometriosis-related bleeding.

#### **Depression**

Confirmed cases of clinically relevant depression or worsening of existing depression is defined as:

- 1. Diagnosis is confirmed by a physician specialized in psychiatry using validated instruments (e.g. HAM-D, BECK depression inventory)<sup>11</sup>
- 2. Confirmed suicide or attempted suicide in a participant with a past history of depression
- 3. Clinical diagnosis confirmed by a physician specialized in psychiatry without the use of validated instruments (see above)<sup>11</sup>
- 4. Confirmed (attempted) suicide without a previous psychiatric diagnosis

#### <u>Treatment Failure</u>

Treatment failure is defined as:

- 1. Medication ineffective given as a reason for stopping or switching treatment
- 2. Side effects of medication given as a reason for stopping or switching treatment

#### 5.4.4 Definition of secondary outcomes

#### Treatment pattern

Treatment pattern is defined as:

- 1. Treatment discontinuation not related to treatment failure (treatment duration over, trying to become pregnant, other reasons)
- 2. Cohort status/switch of women during follow-up, considering the first treatment switch after baseline

#### <u>Selected Baseline characteristics</u>

1. Age, BMI, education, co-morbidity, risk markers, co-medication

#### Risk in adolescence

- 1. Selected baseline characteristics in adolescence
- 2. Anemia (primary outcome) in adolescence
- 3. Depression (primary outcome) in adolescence

<sup>11</sup> Bipolar disorders and schizoaffective disorders are excluded. This specification was added on request of the Safety Monitoring and Advisory Council.



Supporting document SOP BMT 01.09 - Doc 5002.02 - Effective date 21.03.2017

#### Risk of long-term use

- 1. Selected baseline characteristics in long-term user
- 2. Anemia (primary outcome) in long-term user
- 3. Depression (primary outcome) in long-term user
- 4. SAEs in long-term user
- 5.4.5 Definition of other safety outcomes

#### <u>SAEs</u>

SAEs are defined as any adverse event that results in death, a life-threatening experience, inpatient hospitalization, persistent or significant disability/incapacity, or requires medical/surgical intervention to prevent one of the said outcomes. The following items were shown in detail:

- 1. VTE/ATE
- 2. Death
- 3. SAEs by organ system
- 4. Malignant neoplasms
- 5. Malformation of the newborn child

#### 5.4.6 Definition of other outcomes of interest

#### Surgery because of endometriosis symptoms

#### Is defined as:

- 1. Diagnostic surgical intervention
- 2. Any therapeutic surgery related to endometriosis

#### 5.5 Missing data

The investigators were instructed to obtain complete information on primary and secondary outcome variables and primary risk factors. In case of missing data, numbers will be presented in the respective table categories in the descriptive analysis. However, for certain variables (e.g. Mood Score), the last value is carried forward to replace missing items and calculate the related score (as defined in Appendix IV).

Women with multiple exposure or unspecific treatment will be specified as "Allocation unknown".

#### 6. **Data Handling**

Two different databases are used for data collection: the administrative database (ADB) for physician and study participant details and the study database (SDB) for all questionnaire data (baseline and all subsequent follow-ups as well as data gathered during validation of self-reported events).

For each interim analysis and for the final analysis the database is frozen at a predefined time point. The database will be 'cleaned' within 4 weeks of the database freeze. After the final freeze approximately 4 months after the last follow-up questionnaires have been sent to the study participants), no additional incoming data is entered in the database – this database will represent



Supporting document SOP BMT 01.09 - Doc 5002.02 - Effective date 21.03.2017

the final data source for all analyses. Safety copies are made of each database so that all calculations can be repeated if necessary.

#### 6.1 Data coding

Disease diagnoses are coded using the  $ICD10^{12}$  (International Classification of Diseases). Additional codes are used for the coding of events that are of specific interest.

Concomitant medication is coded using WHO ATC-Codes<sup>13</sup>. Surgical procedures are coded using the modified operation and procedure coding list (OPS<sup>14</sup>) provided by DIMDI (German Institute for Medical Documentation and Information). All other relevant information will be coded by a ZEG specific, highly standardized coding system (ZEG Coding Dictionary). All outcomes of interest are additionally described in a case narrative, the "case summary".

#### 6.2 Variable definitions

All time-related variables (age, first diagnosis, first symptoms) are calculated in relation to the study entry date.

#### 6.2.1 Definition of derived variables

The definition of derived or calculated variables from observed items for display in the analysis tables will be described in Appendix IV.

#### 6.2.2 Definition of subgroups

| Variable label | Definition |
|---|---|
| Country | Germany vs. Poland vs. Hungary vs. Switzerland vs. Russia vs. Ukraine |
| Long-term user | 15 months or more of continuous EMT intake |
| EMT user type | Starter vs. restarter vs. switcher |
| Diagnosis classification | Diagnosis of endometriosis confirmed via surgery / laparoscopy vs. diagnosis based on clinical symptoms |
| Age categories | < 20 vs. 20 to < 30 vs. 30 to < 40 vs. >= 40 |
| Age-standardization | Referenced population: NAED cohort |

12 ICD10-Codes Version 2009

13 ATC-Codes Version 2010

14 OPS-Codes Version 2009

Supporting document SOP BMT 01.09 - Doc 5002.02 - Effective date 21.03.2017

#### 7. Interim Analyses and Data Monitoring

#### 7.1 Data Monitoring

This study will maintain scientific independence and will be governed by an independent Safety Monitoring and Advisory Council (SMAC). Bayer Schering Pharma AG Berlin will provide an unconditional grant. The Berlin Center for Epidemiology and Health Research (ZEG), Germany and its research team will be accountable to SMAC in all scientific matters.

The SMAC members will be international experts in relevant scientific fields (e.g., epidemiology, gynecology, psychiatry and internal medicine). The council is responsible for regular review and evaluation of safety data during study conduct as well as for review and approval of the study protocol, statistical analysis plan, interim results, and final study report.

#### 7.2 Interim Analysis

Biannual interim reports will be provided to the funder following the release of the interim analyses results by the independent Safety Monitoring and Advisory Council.

#### 8. Structure of the Analysis Tables

The analysis will be divided in to four sections: Section A – Population Distribution, Section B – Population Characteristics, Section C – Clinical Outcome, and Section D - Comparisons and Inferential statistics.

Baseline characteristics and follow up-characteristics will be displayed for the AT and ITT population. Clinical outcome will be displayed for the AT population, if not otherwise specified.

#### <u>Section A – Population Distribution</u>

Section A overviews the validity and distribution of women. The analysis is stratified by country, EMT user type, and diagnosis classification whenever reasonable.

Section A-1 Eligibility status (enrollment, exclusions)

Study status of women at follow-up, AT and ITT population

Section A-2 Distribution of women, ITT population

Regional distribution

EMT user type at study entry (starter/switcher/restarter)

Diagnosis classification (endometriosis diagnosis based on surgical procedures or

clinical symptoms)

#### Section B – Population Characteristics

Section B summarizes population characteristics of the participating women derived from baseline and follow-up data. The analysis is stratified by country, EMT user type and diagnosis classification.

Section B-1 Age, height, weight and BMI

Section B-2 Socio-economic characteristics and lifestyle factors

Smoking, education level



Supporting document SOP BMT 01.09 - Doc 5002.02 - Effective date 21.03.2017

Section B-3 Gynecological history

Age at menarche, pregnancies, live births, miscarriages, abortions

and/or stillbirths

Section B-4 Endometriosis characteristics

History of EMT use, time since first diagnosis/ first symptoms, surgical procedures,

endometriosis symptoms

Section B-5 Medical History.

Family history of Anemia, Depression,

History of VTE/ATE

Self-reported history of selected cardiovascular risk factors, treated depression and

diseases, presence of mood symptoms

Section B-6 Medication

Regular use of medication, previous medication

Section B-7 Characteristics of Visanne long-term user, Baseline, and Follow-up

Regional distribution, diagnosis classification, age, BMI, endometriosis symptoms

Section B-8 Follow-up characteristics

Mood symptoms and change to baseline, frequencies and timespan of the first switch

after baseline prescription.

Section B-9 Summary tables of selected baseline characteristics

Frequencies of selected baseline characteristics, additionally shown by age categories

and age-standardized and for women with treatment failure and women who

stopped/switched their treatment

#### Section C - Clinical Outcome

Section C provides incidence rates of primary (Section C1), secondary (Section C2) and safety outcomes (Section C3) and other outcomes of interest (Section C4).

Section C-1 Primary outcomes

The analysis of the primary outcomes (Section C1) is stratified by country, EMT user type and diagnosis classification.

Anemia

Incidence rate of Anemia

<u>Depression</u>

Incidence rate of Depression

Treatment failure

Incidence proportion of treatment failure

Section C-2 Secondary Outcomes

The analysis of the secondary outcomes (Section C2) is stratified by country, EMT user type and diagnosis classification.



Supporting document SOP BMT 01.09 - Doc 5002.02 - Effective date 21.03.2017

#### Treatment discontinuation

Incidence proportion if treatment discontinuation reasons unrelated to treatment

#### failure

#### <u>Depression</u>, <u>Anemia and treatment discontinuation in adolescence</u>

Incidence rates of anemia, depression and incidence proportion of treatment discontinuation in adolescence

#### Depression, Anemia and treatment discontinuation for long-term user

Incidence rates of anemia, depression and incidence proportion of treatment discontinuation in long-term user.

#### Section C-3 Other Safety Outcomes

The analysis of other safety outcomes (Section C3) is stratified by country, EMT user type and diagnosis classification.

#### TE (VTE+ATE)

Incidence rate of confirmed TE (VTE+ATE), TIAs

#### Fatal cases

Incidence rate of all death cases

#### Serious adverse events

Incidence rate of SAEs by organ system (complete cohort and long-term user)

#### Malignant neoplasms

Incidence rate of malignant neoplasms by organ system

#### Malformations of the newborn child

Incidence proportion of all reported deliveries and malformations

#### Section C-4 Other Outcomes of Interest

The analysis of other outcomes of interest (Section C4) is stratified by country, EMT user type and diagnosis classification.

#### <u>Surgery / laparoscopy because of endometriosis</u>

Incidence rate of all reported surgeries / laparoscopies

#### Self-reported anemia

Incidence rate of self-reported anemia

#### Self-reported depression

Incidence rate of self-reported depression

#### Section D – Comparisons and Inferential Statistics of Primary Outcomes

Section D consists of tables regarding comparisons between main EMT user groups and inferential statistics, i.e. incidence rate ratios (IRR) and multiple regression analysis of primary outcomes (section D1, D2, D3).



Supporting document SOP BMT 01.09 – Doc 5002.02 – Effective date 21.03.2017

#### Section D-1 Anemia

- Incidence Rate Ratio of Anemia between EMT user cohorts (IRR)
- Risk of Anemia measured as HR (Cox model)
   Crude and adjusted HR

#### Section D-2 Depression

- Incidence Rate Ratio of Depression between EMT user cohorts (IRR)
- Risk of Depression measured as HR (Cox model)
   Crude and adjusted HR

#### Section D-3 Treatment Failure

- Incidence Rate Ratio of Treatment Failure between EMT user cohorts (IRR)
- Risk of Treatment Failure measured as HR (Cox model)
   Crude and adjusted HR



Supporting document SOP BMT 01.09 - Doc 5002.02 - Effective date 21.03.2017

#### 9. **References**

- [1] Nobukata H, Katsuki Y, Ishikawa T, Inokuma M, Shibutani Y. Effect of dienogest on bleeding time, coagulation, fibrinolysis, and platelet aggregation in female rats. Toxicol Lett 1999; 104(1-2):93–101.
- [2] Pérez-Campos EF. Ethinylestradiol/dienogest in oral contraception. Drugs 2010; 70(6):681–9.
- [3] Treatment of pelvic pain associated with endometriosis: A committee opinion. Fertil Steril 2014; 101(4):927–35.
- [4] Dinger JC, Heinemann LAJ, Kühl-Habich D. The safety of a drospirenone-containing oral contraceptive: Final results from the European Active Surveillance Study on oral contraceptives based on 142,475 women-years of observation. Contraception 2007; 75(5):344–54.
- [5] Fischbacher C, Bhopal R, Patel S, White M, Unwin N, Alberti KG. Anaemia in Chinese, South Asian, and European populations in Newcastle upon Tyne: Cross sectional study. BMJ 2001; 322(7292):958–9.
- [6] van Houwelingen H. Modelling Survival Data in Medical Research. D. Collett, Chapman & Hall, London, 1994. No of pages: XVII + 347. Price: E19.99. ISBN 0-41 2-44890-4. Statist. Med. 1995; 14(9):1147–8.
- [7] SAS: The SAS system for Windows, Cary, NC: 2013: SAS Institute Inc.; 2013.
- [8] Rothman KJ, Greenland S, Lash TL. Modern epidemiology. 3rd ed. Philadelphia, Pa., London: Lippincott Williams & Wilkins; 2008. Available from: URL: http://www.loc.gov/catdir/enhancements/fy0743/2007036316-d.html.
- [9] Clopper CJ, Pearson ES. The Use of Confidence or Fiducial Limits Illustrated in the Case of the Binomial. Biometrika 1934; 26(4):404.



Supporting document SOP BMT 01.09 – Doc 5002.02 – Effective date 21.03.2017

## 10. Appendix

### I Baseline questionnaire





#### **INAS-VIPOS**

International Active Surveillance Study of Medication Used for the Treatment of Endometriosis:  $\underline{V} is anne \ \underline{P} ost-approval \ \underline{O} bservational \ \underline{S} tudy$ 

| | <ul> <li>Baseline Questionnaire –</li> </ul> |
|---|---|
| | Country Physician no. Patient no. ID |
| If you h | have any questions, please call our toll-free number: [telephone number]. |
| , , , , , | To be filled in by the physician! |
| _ | TO SECONDARY SECONDARY OF THE PROPERTY OF THE |
| | What is the name of the medication for endometriosis that you prescribed to your patient today? |
| 1a. | If you prescribed an oral contraceptive today, have you prescribed an extended regimen? 2 |
| | □ No □ Yes |
| 2. | Please tick the appropriate box to describe today's prescription: 3 |
| | ☐ First-time hormonal prescription/no previous hormonal treatment |
| | ☐ Repeat of the same hormonal treatment after a medication break of at least 4 weeks |
| | ☐ Switching from another hormonal treatment without a relevant break (< 4 weeks) |
| | ☐ Switching from another hormonal treatment after a break of at least 4 weeks |
| 3. | How would you classify your patient's endometriosis? |
| | □ Diagnosis based only on clinical symptoms |
| | □ Endometriosis confirmed via surgery / laparoscopy |
| 4. | In the last 2 years, how many surgical procedures (diagnostic and/or therapeutical) has your patient received for the management of her endometriosis? |
| | Number of surgical procedures: |
| | The principal of the second of |
| | To be filled in by the study participant! |
| Pers | onal Data |
| 5. | Please give your date of birth: D D 6 M M 7 Y Y Y Y Y 8 |
| 6. | What is your height? cm |
| 7. | What is your weight?kg |
| Gyne | ecological History |
| 8. | How old were you when you had your first menstrual bleeding? |
| 9. | Have you ever been pregnant? 12 |
| | □ No → go to question 10 □ Yes |
| | 22 11 FB 71 ASSOCIES FOR BUILDING |
| 9a. | If <u>ves</u> , when did you last give birth? |
| 9b. | How many live births have you had? |
| 9c. | How many abortions/miscarriages/still births have you had? |
| Endo | ometriosis |
| 10a. | When did you first experience endometriosis symptoms? |
| 10b. | When were you first diagnosed with endometriosis by a physician? \[ \begin{array}{c} \begi |
| | monu yedi |



Supporting document SOP BMT 01.09 – Doc 5002.02 – Effective date 21.03.2017

| 11. | What symptoms do you have associated wit | th your end | ometriosis | ? (plea | ase tick all that apply) |
|---|---|---|---|---|---|
| | $\Box$ Pelvic pain unrelated to period pain $_{\rm 22}$ | vhen pa | assing urine 27 | | |
| | ☐ Experienced pain during or after sexual inter | course 23 | ☐ Pain d | luring b | owel movement 28 |
| | ☐ Difficulty conceiving/infertility 24 | | ☐ Constipation or diarrhoea 29 | | |
| | ☐ Painful periods 25 | | ☐ Tiredn | iess / V | Veakness 30 |
| | $\square$ Heavy or irregular bleeding $_{26}$ | | ☐ Other; | which | 31 32 |
| 12. | Have you had disabling pain associated with events on least two days in the last 4 weeks | | metriosis | preve | nting you from working or attending social |
| | □ No □ Yes | | | | |
| 13. | Please rate the pain associated with your er last 4 weeks, with 0 being no pain and 10 be | | | | box that best describes your pain over the |
| | no pain 0 1 2 3 4 5 | 6 | 7 | 9 | unbearable pain |
| 14. | Have you had an operation to diagnose and | | ur endome | triosis | <b>?</b> 35 |
| | □ No → go on to question 15 | ☐ Yes | | | |
| | If yes, please list the operation (if known) and t<br>removal of ovarian cyst, hysterectomy, colonos<br>For additional space, use comment section on page 4. | | | | |
| | Operation 36 | | | | Date |
| | | | | | M M J <sub>37</sub> Y Y Y Y 38 |
| | | | | | M M Y Y Y Y |
| | | | | | M M Y Y Y Y Y |
| | | | | | M M Y Y Y Y Y |
| 15. | Before today's prescription, have you been | prescribed | any other | medic | |
| | □ No → go on to question 16 | ☐ Yes | | | |
| | If <b>yes</b> , please list <u>all the prescribed medication</u> contraceptive, IUD, progestine, GnRH). Also give section on page 4. | | | | |
| Na | me (type) of medication 40 | | from | | to |
| | | M M 41 | Y Y Y | Y J <sub>42</sub> | M M 43 Y Y Y Y Y 44 □ ongoing 45 |
| | | M M month | Y Y Y year | Y | M,M, Y,Y,Y,Y ☐ ongoing |
| | | M M L | Y Y Y | Υ | M,M, (Y, Y, Y, Y) ☐ ongoing |
| | | M M L | Y Y Y Y | Υ | M M Y Y Y Y Y ☐ ongoing |
| Med | lication | | | | |
| 16. | Are you taking any other medication on a re | gular basis | ? (EXCLU | DING t | oday's prescription) 48 |
| | ☐ No ☐ Yes, which one(s)? (please use Trade Name if known) | | | | |
| | | | | | 47 |
| 17. | Beyond today's prescribed medication, wha | t are you cu | irrently do | ing to | alleviate your endometriosis symptoms? |
| | $\square$ Non-prescription pain killers $_{^{48}}$ | | Massage/ | manual | therapy 52 |
| | ☐ Natural/herbal products ₄9 | | Home rem | nedies ( | (eg. hot water bottle) 53 |
| | ☐ Acupuncture 50 | | Nothing el | se <sub>54</sub> | |
| | ☐ Dietary modification ₅1 | | Other; ple | ase spe | ecify 55 56 |

2



Supporting document SOP BMT 01.09 – Doc 5002.02 – Effective date 21.03.2017

| Medical History 18. Have you ever been told | by a physic | an that you had or have any of the following diseases or conditions? Please |
|---|---|---|
| | | condition was treated by a physician. |
| Deep venous thrombosis 57 (blood clot in the deep veins e.g. legs/arms) | □ No | ☐ Yes, in MMM Self Y Y Y Y Y Self |
| logarams/ | | I was treated by a physician ₀ □ Yes □ No |
| | | I was treated with blood-thinning drugs ₅₁ ☐ Yes ☐ No |
| Pulmonary embolism 62 (blood clot in the lung) | □ No | Yes, in M, M, Y, Y, Y, Y, month 63 year 64 |
| | | I was treated by a physician ⊕5 ☐ Yes ☐ No |
| | | I was treated with blood-thinning drugs ₅ □ Yes □ No |
| Myocardial infarction 67 (heart attack) | □ No | Yes, in |
| | | I was treated by a physician 70 ☐ Yes ☐ No |
| | | If yes, was an ECG performed? ₁₁ ☐ Yes ☐ No |
| | | Was the infarction confirmed by an ECG? ₁₂ ☐ Yes ☐ No |
| Stroke 73 | □ No | Yes, in M M 74 Y Y Y Y 75 |
| | | I was treated by a physician 76 ☐ Yes ☐ No |
| Anemia 77 | □ No | Yes, diagnosed in worth 78 year 79 |
| | | I was treated by a physician <sub>80</sub> □ Yes □ No |
| | | I received a blood or iron trans-/infusion 81 ☐ Yes ☐ No |
| | | I took iron tablets 82 ☐ Yes ☐ No |
| Depression requiring treatment 83 | □ No | ☐ Yes, diagnosed in [M N set Y Y Y Y Y Y Set Y year Y Set Y year Y Set Y Y Y Y Y Y Set Y Y Y Y Y Y Y Y Y Y Y Y Y Y Y Y Y Y Y |
| | | I was treated by a general practitioner 86 ☐ Yes ☐ No |
| | | I was treated by a psychiatrist 87 ☐ Yes ☐ No |
| | | I was admitted to hospital 88 ☐ Yes ☐ No |
| | | There was a suicide attempt № □ Yes □ No |
| Cancer 90<br>(e.g. Breast cancer) | □No | ☐ Yes, diagnosed in [M, M] [Y, Y, Y, Y] [92] year |
| | | What kind of cancer? |
| | | I was treated by a physician 94 ☐ Yes ☐ No |
| Other serious diseases 95<br>(e.g. hypertension, diabetes, benign | □ No | ☐ Yes, which? |
| tumor) | | 1 |
| | | I was treated by a physician ₅ □ Yes □ No |
| | | 2 When? M.M. Y.Y.Y.Y.Y. |
| | | I was treated by a physician ☐ Yes ☐ No |
| | | If you have had more than 2 serious diseases, please use the space in the comment section on page 4. |
| Operations 100 | □ No | ☐ Yes, I had operation(s), which? |
| (excluding those listed in Q14) | | 1 |
| | | 2 When? |
| | | If you have had more than 2 operations, please use the space in the comment section on page 4. |

3



Supporting document SOP BMT 01.09 – Doc 5002.02 – Effective date 21.03.2017

| Relat | tives | | | | |
|---|---|---|---|---|---|
| 19. | - | or sister(s) been diagnosed | d with endometriosis? | | |
| | □ None 104 | ☐ Mother 105 | ☐ Sister | . , | |
| 20. | | parent(s) or sibling(s) beer | | | 1 P |
| | □ None 107 | ☐ Mother 108 | ☐ Fathe | | bling(s) 110 |
| 21. | (blood clot in the I | • | • | , , | |
| Mood | □ None 111 | ☐ Mother 112 | ☐ Fathe | r <sub>113</sub> | bling(s) 114 |
| | We are interested | in finding out about the in changes over the course one of the course of | | | |
| 22a | ı. Have you been fe | eling down, depressed or l | hopeless? 115 | | |
| | ☐ Never | ☐ Rarely | □ Sometimes | ☐ Often | ☐ Always |
| 22b | . Have you been fe | eling like you are a failure | and have let down your | friends and/or family | <b>?</b> <sub>116</sub> |
| | □ Never | □ Rarely | □ Sometimes | ☐ Often | ☐ Always |
| 220 | . Have you felt hap | py or optimistic about the | future? 117 | | |
| | □ Never | □ Rarely | □ Sometimes | ☐ Often | ☐ Always |
| Lifes | tyle | | | | |
| 23. | Do you <u>regularly</u> s | smoke cigarettes (at least | one cigarette a day)? 118 | | |
| | □ Yes | On average | e, how many cigarettes p | er day? | Cigarettes |
| | □ No, stopped sm | oking On average<br>smoke in the | e, how many cigarettes a<br>ne past? | day did you | Cigarettes |
| | ☐ No, never smok | ed regularly | • | 119 | · · |
| Educ | ation | | | | |
| 24. | What is your mos | t advanced school or colle | ege degree? <sub>120</sub> | | |
| | ☐ No school-lea | aving certificate | | | |
| | ☐ High school of | diploma | | | |
| | ☐ Community of | ollege | | | |
| | ☐ University / te | echnical college | | | |
| | Please fill in to | day's date: | 21 month 122 year 123 | | |
| | nment | | | | |
| Ple | ase tell us anything | g else you'd like us to know | <b>W</b> : 124 | | |

Thanks a lot for your help!



Supporting document SOP BMT 01.09 – Doc 5002.02 – Effective date 21.03.2017

## II Follow-up questionnaire

| | LOGO<br>FIELD ORGANIZAT | ION | | | | | ZEG | |
|---|---|---|---|---|---|---|---|---|
| | | | | <b>INAS-VIPOS</b> | | | | |
| | | | - Follow- | up Questionnaire l | No. [N] – | | | |
| | | | | | بينال | | | |
| If voi | ı have any questions, pleas | e call our fre | ee phone numbe | Count | ry Physician | no. Patient r | no. ID | |
| _ | ometriosis Treatment | o our our m | oc priorio riamo | or. [terepriene namber] | | | | |
| 1. | Have you used any ho | ormonal tr | eatment for y | our endometriosis since | we last heard | from you in [mo | onth/year]?₁ | |
| | ☐ Yes → Please fill in a | all medicatio | ns with dates a | nd reasons for stopping / switc | 1 | | | e below |
| Brar | nd name of medication 2 | F | rom | То | (Please tick appro | | ng | |
| | | month 3 | year 4 | ongoing <sub>7</sub> | ☐ Trying to beco☐ Treatment dur☐ Medication ine☐ Side-effects of☐ Which: | ration finished<br>effective<br>f medication | | 9 |
| | | M M L | Y Y Y Y Y year | month year ongoing | Other (e.g. sympto | ome pregnant<br>ration finished<br>effective<br>f medication | | 10 |
| | | M M L | Y 1 Y 1 Y 1 Y 1 | W_M Y_Y_Y_Y Wear ongoing | Other (e.g. symptotics) Trying to become treatment dure Medication ine Side-effects of Which: Other (e.g. symptotics) | ome pregnant<br>ration finished<br>effective<br>f medication | | |
| | | M_M_L | Y I Y I Y I Y I Y I Y I | month year ongoing | ☐ Trying to beco☐ Treatment dur☐ Medication ine☐ Side-effects of Which: | ome pregnant<br>ration finished<br>effective<br>f medication | | |
| | | | | | Other (e.g. sympto | | | |
| | <ul> <li>No, I have not use [month/year] until the provide the medication(s) by</li> </ul> | today.<br>e reason fo | r not using the p | | ☐ Trying to beco<br>☐ Treatment dur<br>☐ Medication ine<br>☐ Side-effects of<br>Which: | ration finished<br>effective<br>f medication | | |
| 2. | Since we last heard fro | m vou in | [month/year] | , have you had surgery/la | Other (e.g. sympto | | ndometrics | |
| | □ No → Go to ques<br>If yes, please specify to | tion 3<br>he type an | ☐ Yes Id date of surg | ery (if known) in the table lery, diagnostic laparoscop | below (i.e. excis | ion of lesions, re | emoval of ova | |
| | Operation 12 | | | | | Date | | |
| | | | | | | M_M_13_Y_Y<br>month 13_y | year 14 | |
| | | | | | | M_M Y_Y | year | |
| Medi<br>3. | cal History We last heard from yo | u in [mon | th/year]. Sind | ce then, have you had an | v of the followi | ng diseases? | | |
| Ane | emia <sub>15</sub> | □ No | ☐ Yes, dia | | Y Y Y Y Y 17 | | | |
| 7 | | | I was | treated by a physician 66 treated with iron tablets 18 | year 17 | □ Yes | □ No | |
| | | | | treated with an iron infusion | Lan | □ Yes | □ No<br>□ No | |
| | | | | treated with a blood transfus | | □ Yes | □ No | |
| | | | | r treatment?. 21 | | □ Yes | □ No | |
| | | | If yes | , which? | | | | _ 22 |
| | p venous thrombosis | □ No | ☐ Yes, in | month 24 | year 25 | | | |
| | Pulmonary embolism 23<br>ad clot in the deep veins e.g. | 3 | I was | treated by a physician 26 | , | □ Yes | □ No | |
| | arms or blood clots in the lung) | | I was | treated with blood-thinning | drugs 27 | □ Yes | □ No | |
| | | | If yes | s which drugs? | | | | 28 |
| | | | | <u> </u> | | | | |



Supporting document SOP BMT 01.09 – Doc 5002.02 – Effective date 21.03.2017

| Dep | ression requiring | □ No | ☐ Yes, diagn | osed in | M 30 Y Y Y | <sub>31</sub> | | |
|---|---|---|---|---|---|---|---|---|
| treatment 29 | | | | eated by a gener | al practitioner 32 | | Yes | □ No |
| | | | l . | eated by a psych<br>Imitted to hospita | | | ∃ Yes<br>∃ Yes | □ No<br>□ No |
| | | | l | ed Suicide 35 | 11 34 | | Yes | □ No |
| Oth | er serious diseases / | □ No | ☐ Yes, which | | | | | |
| ope | rations <sub>36</sub> | | 1 | | 37 | When? | M M 38 Y | Y . Y . Y J |
| | gynecological diseases,<br>rtension, diabetes and cancer) | | l was | treated by a phy | sician 40 | | Yes | □ No |
| | | | 2 | | | When? | MMIY | Y , Y , Y . |
| | | | l was | treated by a phy | sician | | M_M LY_<br>month<br>Yes | year<br>□ No |
| Modi | cations | | If you have | had more than 2 seriou | s diseases/operations, p | lease use the | comment field. | |
| 4. | Are you taking any oth | er medica | tion on a requ | lar basis? (NOT | including the med | tication(s) | listed in guestion | 1) |
| <b>-</b> | | er medica | don on a regu | | one(s)? (please | | | - |
| | | | | L 103, Willott | one(s): (picase | aso brain | a name ii knewi | '' |
| | 14-1141 | | | | | | | 42 |
| | oitalization | ما الما المانية | mr have ver | been admitted | to a boonital (fo | r of loop | t ana niaht\ air | |
| oa. | With the exception of c<br>[month/year]? <sub>43</sub> | iniia aeiive | ery, nave you | been admitted | | | | |
| | □ No → Go to ques | stion 6 | | ☐ Yes | When | was it? | month 44 | year 45 |
| | If yes, was the hosp ☐ No | oital stay pl | anned? <sub>46</sub> | □ Yes | | | | |
| 5b. | What was the reason for | or this hos | pital stay? (PI | | ic as possible) | | | |
| | | | | | . , | | | 47 |
| 50 | Was an operation perfo | ormed? | | | | | | 47 |
| 36. | | Jilleu : 48 | | □Yes | When | was it? | M M 49 | Y . Y . Y I |
| | | | | L 103 | WITCH | was it: | month 49 | year 50 |
| | it ves inlease specif | fy the type | of operation: | | | | | |
| Weig | If yes, please specif | fy the type | of operation: | | | | | . 51 |
| Weig | | | | | | | | |
| 6. | ht | fy the type | | | | | | 51 |
| 6.<br>Preg | ht What is your weight? | <u> </u> | kg | | | | | 51 |
| 6.<br>Preg | ht<br>What is your weight?<br>nancy<br>Have you had a baby s | ince [mon | kg | □ Yes W | hen was the deli | iverv? I | D,D][M,M] | 51 |
| 6.<br>Preg<br>7a. | what is your weight? nancy Have you had a baby s □ No → Go to ques | ince [mon | Lighth/year]? 53 | | | | day s4 M , M | 51<br>55 <u>Year</u> 56 |
| 6.<br>Preg<br>7a. | what is your weight? nancy Have you had a baby s □ No → Go to ques Have there been any se | ince [mon | Lighth/year]? 53 | problems with t | | | D_D_S4 M_M_M<br>day 54 month | 51<br>55 <u>year</u> 56 |
| 6.<br>Preg<br>7a. | what is your weight? nancy Have you had a baby s □ No → Go to ques □ No | ince [mon<br>stion 8a<br>erious hea | th/year]? 53 | | | | D D S4 M M M day 54 month | |
| 6. Preg 7a. 7b. | what is your weight? nancy Have you had a baby si □ No → Go to quest Have there been any se □ No If yes, please specif | ince [mon<br>stion 8a<br>erious hea | th/year]? 53 | problems with t | | | D D S4 M M M day 54 month | 51 51 55 7 7 7 7 7 7 7 7 7 7 7 7 |
| 6. Preg 7a. 7b. | what is your weight? nancy Have you had a baby s □ No → Go to ques Have there been any se □ No □ No □ If yes, please specif | ince [mon<br>stion 8a<br>erious hea | th/year]? 53 Ith issues or p | oroblems with t<br>☐ Yes | the newborn? 57 | | | 58 |
| 6. Preg 7a. 7b. | what is your weight? nancy Have you had a baby s □ No → Go to quest □ No □ No □ If yes, please specificate are interested in the imp | ince [mon stion 8a erious hea | th/year]? 53 Ith issues or particular of problems: | Yes | the newborn? 57 | ı your mo | ood and wheth | er this changes |
| 6. Preg 7a. 7b. Mood We ove | what is your weight? nancy Have you had a baby si □ No → Go to quest Have there been any se □ No □ fyes, please specified are interested in the improve the course of the study | ince [mon stion 8a erious hear fy the types pact of endy. Please | th/year]? 53 Ith issues or problems: | roblems with to<br>☐ Yes ——————————————————————————————————— | the newborn? 57 | ı your mo | ood and wheth | er this changes |
| 6. Preg 7a. 7b. Mood We ove | What is your weight? nancy Have you had a baby s □ No → Go to ques □ No □ No □ If yes, please specificate are interested in the improvement of the study. Have you been feeling | ince [mon<br>stion 8a<br>erious hea<br>fy the types<br>pact of end<br>y. Please<br>down, dep | th/year]? 53 Ith issues or page of problems: Idometriosis all answer these pressed or hope | Yes dendometrios questions base peless? 59 | sis treatment or | ı your mo<br>ve felt ov | ood and wheth<br>er the <u>last 4 w</u> | er this changes |
| 6. Preg 7a. 7b. Mood We ove 8a. | What is your weight? nancy Have you had a baby si □ No → Go to quest □ No □ No □ If yes, please specificat are interested in the improvement of the study Have you been feeling □ Never | ince [mon stion 8a erious hear fy the types pact of endy. Please down, dep | th/year]? 53 Ith issues or problems: Ith issues or problems: Ith issues or problems: | oroblems with to Yes | sis treatment or<br>ed on how you' | ı your move felt ov | ood and wheth<br>er the <u>last 4 w</u><br>□ Alway | er this changes |
| 6. Preg 7a. 7b. Mood We ove 8a. | What is your weight? nancy Have you had a baby s □ No → Go to ques □ No □ No □ If yes, please specificate are interested in the improvement of the study. Have you been feeling | ince [mon stion 8a erious hear fy the types pact of endy. Please down, dep | th/year]? 53 Ith issues or problems: Ith issues or problems: Ith issues or problems: | oroblems with to Yes | sis treatment or<br>ed on how you' | ı your move felt ov | ood and wheth<br>er the <u>last 4 w</u><br>□ Alway | er this changes |
| 6. Preg 7a. 7b. Mood We ove 8a. | What is your weight? nancy Have you had a baby si □ No → Go to quest □ No □ No □ If yes, please specificat are interested in the improvement of the study Have you been feeling □ Never | ince [mon stion 8a erious hear fy the types pact of endy. Please down, dep | th/year]? 53 Ith issues or particles of problems: Idometriosis alanswer these pressed or hopely The a failure an | oroblems with to Yes | sis treatment or<br>ed on how you' | your move felt over ten | ood and wheth<br>er the <u>last 4 w</u><br>□ Alway | er this changes<br>eeks. |
| 6. Preg 7a. 7b. Mooo We ove 8a. | What is your weight? nancy Have you had a baby s □ No → Go to quest Have there been any se □ No If yes, please specificate are interested in the imprime the course of the study Have you been feeling □ Never Have you been feeling | ince [mon stion 8a erious hear fy the types oact of endy. Please down, dep | th/year]? 53 Ith issues or particles of problems: Ith issues or particles are answer these pressed or hopely are a failure and the state of the st | oroblems with to Yes Ind endometrios questions base peless? 59 Sometimes d have let down | sis treatment or<br>ed on how you'd | your move felt over ten | ood and wheth<br>er the <u>last 4 w</u><br>□ Alway<br>nily? ₅₀ | er this changes<br>eeks. |
| 6. Preg 7a. 7b. Mooo We ove 8a. | What is your weight? nancy Have you had a baby s □ No → Go to quest □ No □ If yes, please specificate are interested in the improvement of the study. Have you been feeling □ Never Have you been feeling □ Never | ince [mon stion 8a erious hear fy the types oact of endy. Please down, dep | th/year]? 53 Ith issues or passed of problems: Idometriosis alanswer these pressed or hopely The a failure analy Each about the fut | oroblems with to Yes Ind endometrios questions base peless? 59 Sometimes d have let down | sis treatment or<br>ed on how you'd | your move felt ov<br>ten<br>nd/or far | ood and wheth<br>er the <u>last 4 w</u><br>□ Alway<br>nily? ₅₀ | er this changes<br>eeks. |
| 6. Preg 7a. 7b. Mooo We ove 8a. | What is your weight? nancy Have you had a baby s □ No → Go to quest Have there been any se □ No □ If yes, please specificat are interested in the imprice the course of the study Have you been feeling □ Never Have you been feeling □ Never Have you felt happy or | ince [mon stion 8a erious hear fy the types oact of endy. Please down, dep like you are represented as Rare | th/year]? 53 Ith issues or problems: Ith iss | oroblems with to Yes Ind endometrios questions base peless? 59 Sometimes d have let down Sometimes cure? 61 Sometimes | sis treatment or ed on how you' Of n your friends a | your move felt ov<br>ten<br>nd/or far | ood and wheth<br>rer the <u>last 4 w</u><br>□ Alway<br>nil <b>y?</b> ₅₀<br>□ Alway | er this changes<br>eeks. |
| 6. Preg 7a. 7b. Mood We ove 8a. 8b. | What is your weight? nancy Have you had a baby s □ No → Go to quest Have there been any se □ No □ If yes, please specificat are interested in the impriment of the study. Have you been feeling □ Never Have you been feeling □ Never Have you felt happy or □ Never | ince [mon stion 8a erious hear fy the types oact of endy. Please down, dep like you are represented as Rare | th/year]? 53 Ith issues or passed of problems: Idometriosis alanswer these pressed or hopely The a failure analy Each about the fut | oroblems with to Yes Independent of the Yes | sis treatment or ed on how you' Of n your friends a | your move felt ov<br>ten<br>nd/or far | ood and wheth<br>rer the <u>last 4 w</u><br>□ Alway<br>nil <b>y?</b> ₅₀<br>□ Alway | er this changes<br>eeks. |
| 6. Preg 7a. 7b. Mood We ove 8a. 8b. | What is your weight? nancy Have you had a baby si □ No → Go to quest □ No □ If yes, please specified are interested in the imprime the course of the study Have you been feeling □ Never Have you been feeling □ Never Have you felt happy or □ Never Please fill in today's dament | ince [mon stion 8a erious hear fy the types oact of endy. Please down, dep Rare optimistic Rare | th/year]? 53 Ith issues or problems: Ith iss | oroblems with to Yes Independent of the Yes | sis treatment or ed on how you' Of n your friends a | your move felt ov<br>ten<br>nd/or far | ood and wheth<br>rer the <u>last 4 w</u><br>□ Alway<br>nil <b>y?</b> ₅₀<br>□ Alway | er this changes<br>eeks. |
| 6. Preg 7a. 7b. Mood We ove 8a. 8b. 8c. | What is your weight? nancy Have you had a baby s □ No → Go to quest Have there been any se □ No □ If yes, please specificat are interested in the impriment of the study. Have you been feeling □ Never Have you been feeling □ Never Have you felt happy or □ Never | ince [mon stion 8a erious hear fy the types oact of endy. Please down, dep Rare optimistic Rare | th/year]? 53 Ith issues or problems: Ith iss | oroblems with to Yes Independent of the Yes | sis treatment or ed on how you' Of n your friends a | your move felt ov<br>ten<br>nd/or far | ood and wheth<br>rer the <u>last 4 w</u><br>□ Alway<br>nil <b>y?</b> ₅₀<br>□ Alway | er this changes<br>eeks. |

Thank you for your help with this study!

2

F4



Supporting document SOP BMT 01.09 – Doc 5002.02 – Effective date 21.03.2017

## III List of potential prognostic factors for primary outcomes

| Primary Outcome | Predefined Potential Prognostic Factors |
|---|---|
| Anemia | EMT user type at follow-up, age, history of anemia, history of bleeding disorders |
| Depression | EMT user type at follow-up, age, family and personal history of depression, use of Antidepressants/SSRI, severity of pain |
| Treatment Failure | EMT user type at follow-up, age, family and personal history of depression, current/worsening depression, severity of pain |



Supporting document SOP BMT 01.09 – Doc 5002.02 – Effective date 21.03.2017

## IV List of derived variables

| Variable Label | Definition |
|---|---|
| BMI | Weight (kg) / ( Height(cm) / 100 ) <sup>2</sup> |
| BMI categories | < 20, 20 to <25, 25 to < 30, 30 to < 35, >=35 |
| Age categories | < 20 years, 20 to < 30 years, 30 to < 40 years, >= 40 years |
| Feeling like a failure | Never = 4, Rarely = 3, Sometimes = 2, Often = 1, Always = 0 |
| Felling down, depressed or hopeless | Never = 4, Rarely = 3, Sometimes = 2, Often = 1, Always = 0 |
| Feeling happy or optimistic about the future | Never = 0, Rarely = 1, Sometimes = 2, Often = 3, Always = 4 |
| Mood Score | The response to the three mood-related questions ("Feeling like a failure", "Felling down, depressed or hopeless" and "Feeling happy or optimistic about the future") is scored from 0 to 4, with 4 representing the most positive mental state. The scores of the responses to the three mood questions are then summarized into a single comprehensive Mood Score and transformed to a 0 to 100-point scale. A higher score indicates a better mood. Missing scores for a single mood question are replaced by last observation carried forward (LOCF). |
| Time since first endometriosis symptoms | < 6 months, 6 months to < 1 year, 1 to < 2 years, 2 to < 5 years, 5 to < 10 years, >= 10 years |
| Time since first diagnosis of endometriosis | < 6 months, 6 months to < 1 year, 1 to < 2 years, 2 to < 5 years, 5 to < 10 years, >= 10 years |
| Time span between first endometriosis symptoms and diagnosis | < 6 months, 6 months to < 1 year, 1 to < 2 years, 2 to < 5 years, 5 to < 10 years, >= 10 years |
| Pain severity score | 0 to 3 (mild), 4 to 7 (moderate), 8 to 10 (severe) |



Supporting document SOP BMT 01.09 – Doc 5002.02 – Effective date 21.03.2017

#### **Mock Tables**

#### Volume of Tables:

| Section A | Population Distribution | 66 |
|---|---|---|
| Section A | | 66 |
| Section A | A-1.1 Eligibility Status (all recruited women) | 66 |
| Table A-1 | 1.1.1 Eligibility Status (all recruited women) | 66 |
| Section A | A-1.2 Study status of women at follow-up | 67 |
| Table A-1 | 1.2.1 Study status of women at follow-up, ITT population, Complete cohort | 67 |
| Table A-1 | 1.2.2 Study status of women at follow-up, AT population, Complete cohort | 67 |
| Section A | | |
| Section A | | |
| Table A-2 | , | |
| Section A | A-2.2 EMT user type at study entry | 69 |
| Table A-2 | H | |
| Table A-2 | 2.2.2 EMT user type at study entry, ITT population, Germany | 69 |
| Table A-2 | 2.2.3 EMT user type at study entry, ITT population, Poland | 69 |
| Table A-2 | 2.2.4 EMT user type at study entry, ITT population, Hungary | 69 |
| Table A-2 | 2.2.5 EMT user type at study entry, ITT population, Switzerland | 69 |
| Table A-2 | 2.2.6 EMT user type at study entry, ITT population, Russia | 69 |
| Table A-2 | 2.2.7 EMT user type at study entry, ITT population, Ukraine | 69 |
| Section A | A-2.3 Classification of endometriosis diagnosis at study entry | 70 |
| Table A-2 | 2.3.1 Classification of endometriosis diagnosis at study entry, ITT population, Complete cohort | 70 |
| Table A-2 | 2.3.2 Classification of endometriosis diagnosis at study entry, ITT population, Starter | 70 |
| Table A-2 | 2.3.3 Classification of endometriosis diagnosis at study entry, ITT population, ITT, Switcher | 70 |
| Table A-2 | 2.3.4 Classification of endometriosis diagnosis at study entry, ITT population, Restarter | 70 |
| Table A-2 | 2.3.5 Classification of endometriosis diagnosis at study entry, ITT population, Germany | 70 |
| Table A-2 | 2.3.6 Classification of endometriosis diagnosis at study entry, ITT population, Poland | 70 |



Supporting document SOP BMT 01.09 – Doc 5002.02 – Effective date 21.03.2017

| Table A-2.3.7 | Classification of endometriosis diagnosis at study entry, ITT population, Hungary | 70 |
|---|---|---|
| Table A-2.3.8 | Classification of endometriosis diagnosis at study entry, ITT population, Switzerland | 70 |
| Table A-2.3.9 | Classification of endometriosis diagnosis at study entry, ITT population, Russia | 70 |
| Table A-2.3.10 | Classification of endometriosis diagnosis at study entry, ITT population, Ukraine | 70 |
| Section B Population | n Characteristics | 71 |
| Section B-1 Age ar | nd body measurements | 71 |
| Section B-1.1 | Age at study entry | 71 |
| Table B-1.1.1 | Age (years) at study entry, ITT population, Complete cohort | 71 |
| Table B-1.1.2 | Age (years) at study entry, AT population, Complete cohort | 72 |
| Table B-1.1.3 | Age (years) at study entry, AT population, Starter | 72 |
| Table B-1.1.4 | Age (years) at study entry, AT population, Switcher | 72 |
| Table B-1.1.5 | Age (years) at study entry, AT population, Restarter | 72 |
| Table B-1.1.6 | Age (years) at study entry, AT population, Diagnosis confirmed by surgery | 72 |
| Table B-1.1.7 | Age (years) at study entry, AT population, Diagnosis based on clinical symptoms | 72 |
| Table B-1.1.8 | Age (years) at study entry, AT population, Germany | 72 |
| Table B-1.1.9 | Age (years) at study entry, AT population, Poland | 72 |
| Table B-1.1.10 | Age (years) at study entry, AT population, Hungary | 72 |
| Table B-1.1.11 | Age (years) at study entry, AT population, Switzerland | 72 |
| Table B-1.1.12 | Age (years) at study entry, AT population, Russia | 72 |
| Table B-1.1.13 | Age (years) at study entry, AT population, Ukraine | |
| Section B-1.2 | Height (cm) and Weight (kg) at study entry | 73 |
| Table B-1.2.1 | Height (cm) and Weight (kg) at study entry, ITT population, Complete cohort | 73 |
| Table B-1.2.2 | Height (cm) and Weight (kg) at study entry, AT population, Complete cohort | 74 |
| Table B-1.2.3 | Height (cm) and Weight (kg) at study entry, AT population, Starter | 74 |
| Table B-1.2.4 | Height (cm) and Weight (kg) at study entry, AT population, Switcher | 74 |
| Table B-1.2.5 | Height (cm) and Weight (kg) at study entry, AT population, Restarter | 74 |
| Table B-1.2.6 | Height (cm) and Weight (kg) at study entry, AT population, Diagnosis confirmed by surgery | 74 |
| Table B-1.2.7 | Height (cm) and Weight (kg) at study entry, AT population, Diagnosis based on clinical symptoms | 74 |
| Table B-1.2.8 | Height (cm) and Weight (kg) at study entry, AT population, Germany | 74 |
| Table B-1.2.9 | Height (cm) and Weight (kg) at study entry, AT population, Poland | 74 |



Supporting document SOP BMT 01.09 – Doc 5002.02 – Effective date 21.03.2017

| Table B-1.2.10 | Height (cm) and Weight (kg) at study entry, AT population, Hungary | |
|---|---|---|
| Table B-1.2.11 | Height (cm) and Weight (kg) at study entry, AT population, Switzerland | 74 |
| Table B-1.2.12 | Height (cm) and Weight (kg) at study entry, AT population, Russia | 74 |
| Table B-1.2.13 | Height (cm) and Weight (kg) at study entry, AT population, Ukraine | 74 |
| Section B-1.3 | Body Mass Index (BMI) at study entry | 75 |
| Table B-1.3.1 | Body Mass Index (BMI) at study entry, ITT population, Complete Cohort | 75 |
| Table B-1.3.2 | Body Mass Index (BMI) at study entry, AT population, Complete cohort | 76 |
| Table B-1.3.3 | Body Mass Index (BMI) at study entry, AT population, Starter | 76 |
| Table B-1.3.4 | Body Mass Index (BMI) at study entry, AT population, Switcher | 76 |
| Table B-1.3.5 | Body Mass Index (BMI) at study entry, AT population, Restarter | |
| Table B-1.3.6 | Body Mass Index (BMI) at study entry, AT population, Diagnosis confirmed by surgery | 76 |
| Table B-1.3.7 | Body Mass Index (BMI) at study entry, AT population, Diagnosis based on clinical symptoms | 76 |
| Table B-1.3.8 | Body Mass Index (BMI) at study entry, AT population, Germany | 76 |
| Table B-1.3.9 | Body Mass Index (BMI) at study entry, AT population, Poland | 76 |
| Table B-1.3.10 | Body Mass Index (BMI) at study entry, AT population, Hungary | 76 |
| Table B-1.3.11 | Body Mass Index (BMI) at study entry, AT population, Switzerland | 76 |
| Table B-1.3.12 | Body Mass Index (BMI) at study entry, AT population, Russia | 76 |
| Table B-1.3.13 | Body Mass Index (BMI) at study entry, AT population, Ukraine | 76 |
| Section B-2 Socio | p-economic characteristics and lifestyle factors | 77 |
| Section B-2.1 | Status of cigarette smoking at study entry | 77 |
| Table B-2.1.1 | Status of cigarette smoking at study entry, ITT population, Complete cohort | 77 |
| Table B-2.1.2 | Status of cigarette smoking at study entry, AT population, Complete cohort | 78 |
| Table B-2.1.3 | Status of cigarette smoking at study entry, AT population, Starter | 78 |
| Table B-2.1.4 | Status of cigarette smoking at study entry, AT population, Switcher | 78 |
| Table B-2.1.5 | Status of cigarette smoking at study entry, AT population, Restarter | 78 |
| Table B-2.1.6 | Status of cigarette smoking at study entry, AT population, Diagnosis confirmed by surgery | 78 |
| Table B-2.1.7 | Status of cigarette smoking at study entry, AT population, Diagnosis based on clinical symptoms | 78 |
| Table B-2.1.8 | Status of cigarette smoking at study entry, AT population, Germany | 78 |
| Table B-2.1.9 | Status of cigarette smoking at study entry, AT population, Poland | 78 |
| Table B-2.1.10 | Status of cigarette smoking at study entry, AT population, Hungary | 78 |


| Table B-2.1.11 | Status of cigarette smoking at study entry, AT population, Switzerland | 78 |
|---|---|---|
| Table B-2.1.12 | Status of cigarette smoking at study entry, AT population, Russia | 78 |
| Table B-2.1.13 | Status of cigarette smoking at study entry, AT population, Ukraine | 78 |
| Section B-2.2 | Educational level at study entry | 79 |
| Table B-2.2.1 | Educational level at study entry, ITT population, Complete cohort | 79 |
| Table B-2.2.2 | Educational level at study entry, AT population, Complete cohort | 80 |
| Table B-2.2.3 | Educational level at study entry, AT population, Starter | 80 |
| Table B-2.2.4 | Educational level at study entry, AT population, Switcher | 80 |
| Table B-2.2.5 | Educational level at study entry, AT population, Restarter | 80 |
| Table B-2.2.6 | Educational level at study entry, AT population, Diagnosis confirmed by surgery | 80 |
| Table B-2.2.7 | Educational level at study entry, AT population, Diagnosis based on clinical symptoms | 80 |
| Table B-2.2.8 | Educational level at study entry, AT population, Germany | 80 |
| Table B-2.2.9 | Educational level at study entry, AT population, Poland | 80 |
| Table B-2.2.10 | Educational level at study entry, AT population, Hungary | 80 |
| Table B-2.2.11 | Educational level at study entry, AT population, Switzerland | 80 |
| Table B-2.2.12 | Educational level at study entry, AT population, Russia | 80 |
| Table B-2.2.13 | Educational level at study entry, AT population, Ukraine | 80 |
| Section B-3 Gyne | ecological history | 81 |
| Section B-3.1 | Age (years) at menarche at study entry | 81 |
| Table B-3.1.1 | Age (years) at menarche at study entry, ITT population, Complete cohort | 81 |
| Table B-3.1.2 | Age (years) at menarche at study entry, AT population, Complete cohort | 82 |
| Table B-3.1.3 | Age (years) at menarche at study entry, AT population, Starter | 82 |
| Table B-3.1.4 | Age (years) at menarche at study entry, AT population, Switcher | 82 |
| Table B-3.1.5 | Age (years) at menarche at study entry, AT population, Restarter | 82 |
| Table B-3.1.6 | Age (years) at menarche at study entry, AT population, Diagnosis confirmed by surgery | 82 |
| Table B-3.1.7 | Age (years) at menarche at study entry, AT population, Diagnosis based on clinical symptoms | 82 |
| Table B-3.1.8 | Age (years) at menarche at study entry, AT population, Germany | 82 |
| Table B-3.1.9 | Age (years) at menarche at study entry, AT population, Poland | 82 |
| Table B-3.1.10 | Age (years) at menarche at study entry, AT population, Hungary | 82 |
| Table B-3.1.11 | Age (years) at menarche at study entry, AT population, Switzerland | 82 |



| Table B-3.1.12 | Age (years) at menarche at study entry, AT population, Russia | 82 |
|---|---|---|
| Table B-3.1.13 | Age (years) at menarche at study entry, AT population, Ukraine | 82 |
| Section B-3.2 | Pregnancy status at study entry | 83 |
| Table B-3.2.1 | Pregnancy status at study entry, ITT population, Complete cohort | 83 |
| Table B-3.2.2 | Pregnancy status at study entry, AT population, Complete cohort | 84 |
| Table B-3.2.3 | Pregnancy status at study entry, AT population, Starter | 84 |
| Table B-3.2.4 | Pregnancy status at study entry, AT population, Switcher | 84 |
| Table B-3.2.5 | Pregnancy status at study entry, AT population, Restarter | 84 |
| Table B-3.2.6 | Pregnancy status at study entry, AT population, Diagnosis confirmed by surgery | 84 |
| Table B-3.2.7 | Pregnancy status at study entry, AT population, Diagnosis based on clinical symptoms | 84 |
| Table B-3.2.8 | Pregnancy status at study entry, AT population, Germany | 84 |
| Table B-3.2.9 | Pregnancy status at study entry, AT population, Poland | 84 |
| Table B-3.2.10 | Pregnancy status at study entry, AT population, Hungary | 84 |
| Table B-3.2.11 | Pregnancy status at study entry, AT population, Switzerland | 84 |
| Table B-3.2.12 | Pregnancy status at study entry, AT population, Russia | 84 |
| Table B-3.2.13 | Pregnancy status at study entry, AT population, Ukraine | 84 |
| Section B-3.3 | Number of live births, abortions, miscarriages and/or still births at study entry | 85 |
| Table B-3.3.1 | Number of live births, abortions, miscarriages and/or still births at study entry, ITT population, Complete cohort | 85 |
| Table B-3.3.2 | Number of live births, miscarriages, abortions and/or still births at study entry, AT population, Complete cohort | 86 |
| Table B-3.3.3 | Number of live births, miscarriages, abortions and/or still births at study entry, AT population, Starter | 86 |
| Table B-3.3.4 | Number of live births, miscarriages, abortions and/or still births at study entry, AT population, Switcher | 86 |
| Table B-3.3.5 | Number of live births, miscarriages, abortions and/or still births at study entry, AT population, Restarter | 86 |
| Table B-3.3.6 | Number of live births, miscarriages, abortions and/or still births at study entry, AT population, Diagnosis confirmed by surgery | 86 |
| Table B-3.3.7 | Number of live births, miscarriages, abortions and/or still births at study entry, AT population, Diagnosis based on clinical symptoms | 86 |
| Table B-3.3.8 | Number of live births, miscarriages, abortions and/or still births at study entry, AT population, Germany | 86 |
| Table B-3.3.9 | Number of live births, miscarriages, abortions and/or still births at study entry, AT population, Poland | 86 |
| Table B-3.3.10 | Number of live births, miscarriages, abortions and/or still births at study entry, AT population, Hungary | 86 |
| Table B-3.3.11 | Number of live births, miscarriages, abortions and/or still births at study entry, AT population, Switzerland | 86 |
| Table B-3.3.12 | Number of live births, miscarriages, abortions and/or still births at study entry, AT population, Russia | 86 |
| Table B-3.3.13 | Number of live births, miscarriages, abortions and/or still births at study entry, AT population, Ukraine | 86 |



| Section B-4 | Endometriosis characteristics | 87 |
|---|---|---|
| Section B-4.1 | Time since first endometriosis symptoms at study entry | 87 |
| Table B-4.1.1 | Time since first endometriosis symptoms at study entry, ITT population, Complete cohort | 87 |
| Table B-4.1.2 | Time since first endometriosis symptoms at study entry, ITT population, Complete cohort | 88 |
| Table B-4.1.3 | Time since first endometriosis symptoms at study entry, AT population, Starter | 88 |
| Table B-4.1.4 | Time since first endometriosis symptoms at study entry, AT population, Switcher | 88 |
| Table B-4.1.5 | Time since first endometriosis symptoms at study entry, AT population, Restarter | 88 |
| Table B-4.1.6 | Time since first endometriosis symptoms at study entry, AT population, Diagnosis confirmed by surgery | 88 |
| Table B-4.1.7 | Time since first endometriosis symptoms at study entry, AT population, Diagnosis based on clinical symptoms | 88 |
| Table B-4.1.8 | Time since first endometriosis symptoms at study entry, AT population, Germany | 88 |
| Table B-4.1.9 | Time since first endometriosis symptoms at study entry, AT population, Poland | 88 |
| Table B-4.1.1 | Time since first endometriosis symptoms at study entry, AT population, Hungary | 88 |
| Table B-4.1.1 | Time since first endometriosis symptoms at study entry, AT population, Switzerland | 88 |
| Table B-4.1.1 | 2 Time since first endometriosis symptoms at study entry, AT population, Russia | 88 |
| Table B-4.1.1 | Time since first endometriosis symptoms at study entry, AT population, Ukraine | 88 |
| Section B-4.2 | Time since first diagnosis of endometriosis at study entry | 89 |
| Table B-4.2.1 | Time since first diagnosis of endometriosis at study entry, ITT population, Complete cohort | 89 |
| Table B-4.2.2 | Time since first diagnosis of endometriosis at study entry, AT population, Complete cohort | 90 |
| Table B-4.2.3 | Time since first diagnosis of endometriosis at study entry, AT population, Starter | 90 |
| Table B-4.2.4 | Time since first diagnosis of endometriosis at study entry, AT population, Switcher | 90 |
| Table B-4.2.5 | Time since first diagnosis of endometriosis at study entry, AT population, Restarter | 90 |
| Table B-4.2.6 | Time since first diagnosis of endometriosis at study entry, AT population, Diagnosis confirmed by surgery | 90 |
| Table B-4.2.7 | Time since first diagnosis of endometriosis at study entry, AT population, Diagnosis based on clinical symptoms | 90 |
| Table B-4.2.8 | Time since first diagnosis of endometriosis at study entry, AT population, Germany | 90 |
| Table B-4.2.9 | Time since first diagnosis of endometriosis at study entry, AT population, Poland | 90 |
| Table B-4.2.1 | Time since first diagnosis of endometriosis at study entry, AT population, Hungary | 90 |
| Table B-4.2.1 | Time since first diagnosis of endometriosis at study entry, AT population, Switzerland | 90 |
| Table B-4.2.1 | 2 Time since first diagnosis of endometriosis at study entry, AT population, Russia | 90 |
| Table B-4.2.1 | Time since first diagnosis of endometriosis at study entry, AT population, Ukraine | 90 |
| Section B-4.3 | Time span between occurrence of endometriosis symptoms and diagnosis | 91 |



## INAS-VIPOS Statistical Analysis Plan V02-00

| Table B-4.3.1 | Time span between occurrence of endometriosis symptoms and diagnosis, ITT population, Complete cohort | 91 |
|---|---|---|
| Table B-4.3.2 | Time span between occurrence of endometriosis symptoms and diagnosis, AT population, Complete cohort | 92 |
| Table B-4.3.3 | Time span between occurrence of endometriosis symptoms and diagnosis, AT population, Starter | 92 |
| Table B-4.3.4 | Time span between occurrence of endometriosis symptoms and diagnosis, AT population, Switcher | 92 |
| Table B-4.3.5 | Time span between occurrence of endometriosis symptoms and diagnosis, AT population, Restarter | 92 |
| Table B-4.3.6 | Time span between occurrence of endometriosis symptoms and diagnosis, AT population, Diagnosis confirmed by surgery | 92 |
| Table B-4.3.7 | Time span between occurrence of endometriosis symptoms and diagnosis, AT population, Diagnosis based on clinical symptoms | 92 |
| Table B-4.3.8 | Time span between occurrence of endometriosis symptoms and diagnosis, AT population, Germany | 92 |
| Table B-4.3.9 | Time span between occurrence of endometriosis symptoms and diagnosis, AT population, Poland | 92 |
| Table B-4.3.10 | Time span between occurrence of endometriosis symptoms and diagnosis, AT population, Hungary | 92 |
| Table B-4.3.11 | Time span between occurrence of endometriosis symptoms and diagnosis, AT population, Switzerland | 92 |
| Table B-4.3.12 | Time span between occurrence of endometriosis symptoms and diagnosis, AT population, Russia | 92 |
| Table B-4.3.13 | Time span between occurrence of endometriosis symptoms and diagnosis, AT population, Ukraine | 92 |
| Section B-4.4 | Surgical procedures for the management of endometriosis during the past two years | 93 |
| Table B-4.4.1 | Surgical procedures for the management of endometriosis during the past two years, ITT population, Complete cohort | 93 |
| Table B-4.4.2 | Surgical procedures for the management of endometriosis during the past two years, AT population, Complete cohort | 94 |
| Table B-4.4.3 | Surgical procedures for the management of endometriosis during the past two years, AT population, Starter | 94 |
| Table B-4.4.4 | Surgical procedures for the management of endometriosis during the past two years, AT population, Switcher | 94 |
| Table B-4.4.5 | Surgical procedures for the management of endometriosis during the past two years, AT population, Restarter | 94 |
| Table B-4.4.6 | Surgical procedures for the management of endometriosis during the past two years, AT population, Diagnosis confirmed by surgery | 94 |
| Table B-4.4.7 | Surgical procedures for the management of endometriosis during the past two years, AT population, Diagnosis based on clinical sympt | oms 94 |
| Table B-4.4.8 | Surgical procedures for the management of endometriosis during the past two years, AT population, Germany | 94 |
| Table B-4.4.9 | Surgical procedures for the management of endometriosis during the past two years, AT population, Poland | 94 |
| Table B-4.4.10 | Surgical procedures for the management of endometriosis during the past two years, AT population, Hungary | 94 |
| Table B-4.4.11 | Surgical procedures for the management of endometriosis during the past two years, AT population, Switzerland | 94 |
| Table B-4.4.12 | Surgical procedures for the management of endometriosis during the past two years, AT population, Russia | 94 |
| Table B-4.4.13 | Surgical procedures for the management of endometriosis during the past two years, AT population, Ukraine | 94 |
| Section B-4.5 | Self-reported surgical procedures related to endometriosis at study entry, | 95 |
| Table B-4.5.1 | Self-reported surgical procedures related to endometriosis at study entry, ITT population, Complete cohort | 95 |
| Table B-4.5.2 | Self-reported surgical procedures related to endometriosis at study entry, AT population, Complete cohort | 97 |



| Table B-4.5.3 | Self-reported surgical procedures related to endometriosis at study entry, AT population, Starter | 97 |
|---|---|---|
| Table B-4.5.4 | Self-reported surgical procedures related to endometriosis at study entry, AT population, Switcher | 97 |
| Table B-4.5.5 | Self-reported surgical procedures related to endometriosis at study entry, AT population, Restarter | 97 |
| Table B-4.5.6 | Self-reported surgical procedures related to endometriosis at study entry, AT population, Diagnosis confirmed by surgery | 97 |
| Table B-4.5.7 | Self-reported surgical procedures related to endometriosis at study entry, AT population, Diagnosis based on clinical symptoms | 97 |
| Table B-4.5.8 | Self-reported surgical procedures related to endometriosis at study entry, AT population, Germany | 97 |
| Table B-4.5.9 | Self-reported surgical procedures related to endometriosis at study entry, AT population, Poland | 97 |
| Table B-4.5.10 | Self-reported surgical procedures related to endometriosis at study entry, AT population, Hungary | 97 |
| Table B-4.5.11 | Self-reported surgical procedures related to endometriosis at study entry, AT population, Switzerland | 97 |
| Table B-4.5.12 | Self-reported surgical procedures related to endometriosis at study entry, AT population, Russia | 97 |
| Table B-4.5.13 | Self-reported surgical procedures related to endometriosis at study entry, AT population, Ukraine | 97 |
| Section B-4.6 | Endometriosis associated symptoms at study entry | 98 |
| Table B-4.6.1 | Endometriosis associated symptoms at study entry, ITT population, Complete cohort | 98 |
| Table B-4.6.2 | Endometriosis associated symptoms at study entry, AT population, Complete cohort | 99 |
| Table B-4.6.3 | Endometriosis associated symptoms at study entry, AT population, Starter | 99 |
| Table B-4.6.4 | Endometriosis associated symptoms at study entry, AT population, Switcher | 99 |
| Table B-4.6.5 | Endometriosis associated symptoms at study entry, AT population, Restarter | 99 |
| Table B-4.6.6 | Endometriosis associated symptoms at study entry, AT population, Diagnosis confirmed by surgery | 99 |
| Table B-4.6.7 | Endometriosis associated symptoms at study entry, AT population, Diagnosis based on clinical symptoms | 99 |
| Table B-4.6.8 | Endometriosis associated symptoms at study entry, AT population, Germany | 99 |
| Table B-4.6.9 | Endometriosis associated symptoms at study entry, AT population, Poland | 99 |
| Table B-4.6.10 | Endometriosis associated symptoms at study entry, AT population, Hungary | 99 |
| Table B-4.6.11 | Endometriosis associated symptoms at study entry, AT population, Switzerland | 99 |
| Table B-4.6.12 | Endometriosis associated symptoms at study entry, AT population, Russia | 99 |
| Table B-4.6.13 | Endometriosis associated symptoms at study entry, AT population, Ukraine | 99 |
| Section B-4.7 | Disabling endometriosis associated pain preventing the woman from working or attending social events at study entry | 100 |
| Table B-4.7.1 | Disabling endometriosis associated pain preventing the woman from working or attending social events at study entry, ITT population | on, |
| Complete cohort | 100 | |
| Table B-4.7.2 | Disabling endometriosis associated pain preventing the woman from working or attending social events at study entry, AT population | on, |
| Complete cohort | 101 | |



| Table B-4.7.3 | Disabling endometriosis associated pain preventing the woman from working or attending social events at study entry, AT population, | Starter |
|---|---|---|
| | 101 | |
| Table B-4.7.4 | Disabling endometriosis associated pain preventing the woman from working or attending social events at study entry, AT population, | |
| Switcher | 101 | |
| Table B-4.7.5 | Disabling endometriosis associated pain preventing the woman from working or attending social events at study entry, AT population, | |
| Restarter | 101 | |
| Table B-4.7.6 | Disabling endometriosis associated pain preventing the woman from working or attending social events at study entry, AT population, | |
| Diagnosis confirmed | l by surgery | 101 |
| Table B-4.7.7 | Disabling endometriosis associated pain preventing the woman from working or attending social events at study entry, AT population, | |
| Diagnosis based on o | clinical symptoms | 101 |
| Table B-4.7.8 | Disabling endometriosis associated pain preventing the woman from working or attending social events at study entry, AT population, | |
| Germany | 101 | |
| Table B-4.7.9 | Disabling endometriosis associated pain preventing the woman from working or attending social events at study entry, AT population, | Poland |
| | 101 | |
| Table B-4.7.10 | Disabling endometriosis associated pain preventing the woman from working or attending social events at study entry, AT population, | |
| Hungary | 101 | |
| Table B-4.7.11 | Disabling endometriosis associated pain preventing the woman from working or attending social events at study entry, AT population, | |
| Switzerland | 101 | |
| Table B-4.7.12 | Disabling endometriosis associated pain preventing the woman from working or attending social events at study entry, AT population, | Russia |
| | 101 | |
| Table B-4.7.13 | Disabling endometriosis associated pain preventing the woman from working or attending social events at study entry, AT population, | |
| Ukraine | 101 | |
| Section B-4.8 | Severity of endometriosis associated pain at study entry | 102 |
| Table B-4.8.1 | Severity of endometriosis associated pain at study entry, ITT population, Complete cohort | 102 |
| Table B-4.8.2 | Severity of endometriosis associated pain at study entry, AT population, Complete cohort | 103 |
| Table B-4.8.3 | Severity of endometriosis associated pain at study entry, AT population, Starter | 103 |
| Table B-4.8.4 | Severity of endometriosis associated pain at study entry, AT population, Switcher | 103 |
| Table B-4.8.5 | Severity of endometriosis associated pain at study entry, AT population, Restarter | 103 |
| Table B-4.8.6 | Severity of endometriosis associated pain at study entry, AT population, Diagnosis confirmed by surgery | 103 |
| Table B-4.8.7 | Severity of endometriosis associated pain at study entry, AT population, Diagnosis based on clinical symptoms | 103 |



| Table B-4.8.8 | Severity of endometriosis associated pain at study entry, AT population, Germany | 103 |
|---|---|---|
| Table B-4.8.9 | Severity of endometriosis associated pain at study entry, AT population, Poland | 103 |
| Table B-4.8.10 | Severity of endometriosis associated pain at study entry, AT population, Hungary | 103 |
| Table B-4.8.11 | Severity of endometriosis associated pain at study entry, AT population, Switzerland | 103 |
| Table B-4.8.12 | Severity of endometriosis associated pain at study entry, AT population, Russia | 103 |
| Table B-4.8.13 | Severity of endometriosis associated pain at study entry, AT population, Ukraine | 103 |
| Section B-5 Medi | cal history | 104 |
| Section B-5.1 | Self-reported history of selected risk factors at study entry | 104 |
| Table B-5.1.1 | Self-reported history of selected risk factors at study entry, ITT population, Complete cohort | 104 |
| Table B-5.1.2 | Self-reported history of selected risk factors at study entry, AT population, Complete cohort | 105 |
| Table B-5.1.3 | Self-reported history of selected risk factors at study entry, AT population, Starter | 105 |
| Table B-5.1.4 | Self-reported history of selected risk factors at study entry, AT population, Switcher | 105 |
| Table B-5.1.5 | Self-reported history of selected risk factors at study entry, AT population, Restarter | 105 |
| Table B-5.1.6 | Self-reported history of selected risk factors at study entry, AT population, Diagnosis confirmed by surgery | 105 |
| Table B-5.1.7 | Self-reported history of selected risk factors at study entry, AT population, Diagnosis based on clinical symptoms | 105 |
| Table B-5.1.8 | Self-reported history of selected risk factors at study entry, AT population, Germany | 105 |
| Table B-5.1.9 | Self-reported history of selected risk factors at study entry, AT population, Poland | 105 |
| Table B-5.1.10 | Self-reported history of selected risk factors at study entry, AT population, Hungary | 105 |
| Table B-5.1.11 | Self-reported history of selected risk factors at study entry, AT population, Switzerland | 105 |
| Table B-5.1.12 | Self-reported history of selected risk factors at study entry, AT population, Russia | 105 |
| Table B-5.1.13 | Self-reported history of selected risk factors at study entry, AT population, Ukraine | 105 |
| Section B-5.2 | Self-reported history of selected diseases at study entry | 106 |
| Table B-5.2.1 | Self-reported history of selected diseases at study entry, ITT population, Complete cohort | 106 |
| Table B-5.2.2 | Self-reported history of selected diseases at study entry, AT population, Complete cohort | 107 |
| Table B-5.2.3 | Self-reported history of selected diseases at study entry, AT population, Starter | 107 |
| Table B-5.2.4 | Self-reported history of selected diseases at study entry, AT population, Switcher | 107 |
| Table B-5.2.5 | Self-reported history of selected diseases at study entry, AT population, Restarter | 107 |
| Table B-5.2.6 | Self-reported history of selected diseases at study entry, AT population, Diagnosis confirmed by surgery | 107 |
| Table B-5.2.7 | Self-reported history of selected diseases at study entry, AT population, Diagnosis based on clinical symptoms | 107 |
| Table B-5.2.8 | Self-reported history of selected diseases at study entry, AT population, Germany | 107 |



| Table B-5.2.9 | Self-reported history of selected diseases at study entry, AT population, Poland | 107 |
|---|---|---|
| Table B-5.2.10 | Self-reported history of selected diseases at study entry, AT population, Hungary | 107 |
| Table B-5.2.11 | Self-reported history of selected diseases at study entry, AT population, Switzerland | 107 |
| Table B-5.2.12 | Self-reported history of selected diseases at study entry, AT population, Russia | 107 |
| Table B-5.2.13 | Self-reported history of selected diseases at study entry, AT population, Ukraine | 107 |
| Section B-6 Medica | ation and other procedures for endometriosis treatment | 108 |
| Section B-6.1 | Medication prescribed for the treatment of endometriosis during the past two years before study entry | 108 |
| Table B-6.1.1 | Medication prescribed for the treatment of endometriosis during the past two years before study entry, ITT population, Complete co | hort 108 |
| Table B-6.1.2 | Medication prescribed for the treatment of endometriosis during the past two years before study entry, AT population, Complete col | hort 109 |
| Table B-6.1.3 | Medication prescribed for the treatment of endometriosis during the past two years before study entry, AT population, Starter | 109 |
| Table B-6.1.4 | Medication prescribed for the treatment of endometriosis during the past two years before study entry, AT population, Switcher | 109 |
| Table B-6.1.5 | Medication prescribed for the treatment of endometriosis during the past two years before study entry, AT population, Restarter | 109 |
| Table B-6.1.6 | Medication prescribed for the treatment of endometriosis during the past two years before study entry, AT population, Diagnosis cor | nfirmed |
| by surgery | 109 | |
| Table B-6.1.7 | Medication prescribed for the treatment of endometriosis during the past two years before study entry, AT population, Diagnosis based | sed on |
| clinical symptoms | 109 | |
| Table B-6.1.8 | Medication prescribed for the treatment of endometriosis during the past two years before study entry, AT population, Germany | 109 |
| Table B-6.1.9 | Medication prescribed for the treatment of endometriosis during the past two years before study entry, AT population, Poland | 109 |
| Table B-6.1.10 | Medication prescribed for the treatment of endometriosis during the past two years before study entry, AT population, Hungary | 109 |
| Table B-6.1.11 | Medication prescribed for the treatment of endometriosis during the past two years before study entry, AT population, Switzerland | 109 |
| Table B-6.1.12 | Medication prescribed for the treatment of endometriosis during the past two years before study entry, AT population, Russia | 109 |
| Table B-6.1.13 | Medication prescribed for the treatment of endometriosis during the past two years before study entry, AT population, Ukraine | 109 |
| Section B-6.2 | Medication and other procedures for endometriosis treatment at study entry | 110 |
| Table B-6.2.1 | Medication and other procedures for endometriosis treatment at study entry, ITT population, Complete cohort | 110 |
| Table B-6.2.2 | Medication and other procedures for endometriosis treatment at study entry, AT population, Complete cohort | 111 |
| Table B-6.2.3 | Medication and other procedures for endometriosis treatment at study entry, AT population, Starter | 111 |
| Table B-6.2.4 | Medication and other procedures for endometriosis treatment at study entry, AT population, Switcher | 111 |
| Table B-6.2.5 | Medication and other procedures for endometriosis treatment at study entry, AT population, Restarter | 111 |
| Table B-6.2.6 | Medication and other procedures for endometriosis treatment at study entry, AT population, Diagnosis confirmed by surgery | 111 |
| Table B-6.2.7 | Medication and other procedures for endometriosis treatment at study entry, AT population, Diagnosis based on clinical symptoms | 111 |



| Table B-6.2.8 | Medication and other procedures for endometriosis treatment at study entry, AT population, Germany | 111 |
|---|---|---|
| Table B-6.2.9 | Medication and other procedures for endometriosis treatment at study entry, AT population, Poland | 111 |
| Table B-6.2.10 | Medication and other procedures for endometriosis treatment at study entry, AT population, Hungary | 111 |
| Table B-6.2.11 | Medication and other procedures for endometriosis treatment at study entry, AT population, Switzerland | 111 |
| Table B-6.2.12 | Medication and other procedures for endometriosis treatment at study entry, AT population, Russia | 111 |
| Table B-6.2.13 | Medication and other procedures for endometriosis treatment at study entry, AT population, Ukraine | 111 |
| Section B-6.3 | Regular use of other than endometriosis treatment medication at study entry | 112 |
| Table B-6.3.1 | Regular use of other than endometriosis treatment medication at study entry, ITT population, Complete cohort | 112 |
| Table B-6.3.2 | Regular use of other than endometriosis treatment medication at study entry, AT population, Complete cohort | 113 |
| Table B-6.3.3 | Regular use of other than endometriosis treatment medication at study entry, AT population, Starter | 113 |
| Table B-6.3.4 | Regular use of other than endometriosis treatment medication at study entry, AT population, Switcher | 113 |
| Table B-6.3.5 | Regular use of other than endometriosis treatment medication at study entry, AT population, Restarter | 113 |
| Table B-6.3.6 | Regular use of other than endometriosis treatment medication at study entry, AT population, Diagnosis confirmed by surgery | 113 |
| Table B-6.3.7 | Regular use of other than endometriosis treatment medication at study entry, AT population, Diagnosis based on clinical symptoms | 113 |
| Table B-6.3.8 | Regular use of other than endometriosis treatment medication at study entry, AT population, Germany | 113 |
| Table B-6.3.9 | Regular use of other than endometriosis treatment medication at study entry, AT population, Poland | 113 |
| Table B-6.3.10 | Regular use of other than endometriosis treatment medication at study entry, AT population, Hungary | 113 |
| Table B-6.3.11 | Regular use of other than endometriosis treatment medication at study entry, AT population, Switzerland | 113 |
| Table B-6.3.12 | Regular use of other than endometriosis treatment medication at study entry, AT population, Russia | 113 |
| Table B-6.3.13 | Regular use of other than endometriosis treatment medication at study entry, AT population, Ukraine | |
| Section B-6.4 | Psychotropic medication at study entry | 114 |
| Table B-6.4.1 | Psychotropic medication at study entry, ITT population, Complete cohort | 114 |
| Table B-6.4.2 | Psychotropic medication at study entry, AT population, Complete cohort | 115 |
| Table B-6.4.3 | Psychotropic medication at study entry, AT population, Starter | 115 |
| Table B-6.4.4 | Psychotropic medication at study entry, AT population, Switcher | 115 |
| Table B-6.4.5 | Psychotropic medication at study entry, AT population, Restarter | 115 |
| Table B-6.4.6 | Psychotropic medication at study entry, AT population, Diagnosis confirmed by surgery | 115 |
| Table B-6.4.7 | Psychotropic medication at study entry, AT population, Diagnosis based on clinical symptoms | 115 |
| Table B-6.4.8 | Psychotropic medication at study entry, AT population, Germany | 115 |
| Table B-6.4.9 | Psychotropic medication at study entry, AT population, Poland | 115 |



| Table B-6.4.10 | Psychotropic medication at study entry, AT population, Hungary | 115 |
|---|---|---|
| Table B-6.4.11 | Psychotropic medication at study entry, AT population, Switzerland | 115 |
| Table B-6.4.12 | Psychotropic medication at study entry, AT population, Russia | 115 |
| Table B-6.4.13 | Psychotropic medication at study entry, AT population, Ukraine | 115 |
| Section B-7 Distri | ibution and selected baseline characteristics of Visanne long-term useruser | 116 |
| Section B-7.1 | Duration of Visanne use | 116 |
| Table B-7.1.1 | Duration of Visanne use | 116 |
| Table B-7.1.2 | Duration of Visanne use, Starter | 117 |
| Table B-7.1.3 | Duration of Visanne use, Switcher | 117 |
| Table B-7.1.4 | Duration of Visanne use, Restarter | 117 |
| Table B-7.1.5 | Duration of Visanne use, Diagnosis confirmed by surgery | 117 |
| Table B-7.1.6 | Duration of Visanne use, Diagnosis based on clinical symptoms | 117 |
| Table B-7.1.7 | Duration of Visanne use, Germany | 117 |
| Table B-7.1.8 | Duration of Visanne use, Poland | 117 |
| Table B-7.1.9 | Duration of Visanne use, Hungary | 117 |
| Table B-7.1.10 | Duration of Visanne use, Switzerland | 117 |
| Table B-7.1.11 | Duration of Visanne use, Russia | 117 |
| Table B-7.1.12 | Duration of Visanne use, Ukraine | 11 |
| Section B-7.2 | Regional distribution | 118 |
| Table B-7.2.1 | Regional distribution | 118 |
| Table B-7.2.2 | Regional distribution, Starter | 119 |
| Table B-7.2.3 | Regional distribution, Switcher | 119 |
| Table B-7.2.4 | Regional distribution, Restarter | 119 |
| Table B-7.2.5 | Regional distribution, Diagnosis confirmed by surgery | 119 |
| Table B-7.2.6 | Regional distribution, Diagnosis based on clinical symptoms | 119 |
| Section B-7.3 | Diagnosis classification at study entry | 120 |
| Table B-7.3.1 | Diagnosis classification at study entry | |
| Table B-7.3.2 | Diagnosis classification at study entry, Starter | |
| Table B-7.3.3 | Diagnosis classification at study entry, Switcher | 122 |
| Table B-7.3.4 | Diagnosis classification at study entry, Restarter | |



| Table B-7.3.5 | Diagnosis classification at study entry, Germany | |
|---|---|---|
| Table B-7.3.6 | Diagnosis classification at study entry, Poland | 121 |
| Table B-7.3.7 | Diagnosis classification at study entry, Hungary | 121 |
| Table B-7.3.8 | Diagnosis classification at study entry, Switzerland | 121 |
| Table B-7.3.9 | Diagnosis classification at study entry, Russia | 121 |
| Table B-7.3.10 | Diagnosis classification at study entry, Ukraine | 121 |
| Section B-7.4 | Age (years) at study entry | 122 |
| Table B-7.4.1 | Age (years) at study entry | 122 |
| Table B-7.4.2 | Age (years) at study entry, Starter | 123 |
| Table B-7.4.3 | Age (years) at study entry, Switcher | 123 |
| Table B-7.4.4 | Age (years) at study entry, Restarter | 123 |
| Table B-7.4.5 | Age (years) at study entry, Diagnosis confirmed by surgery | 123 |
| Table B-7.4.6 | Age (years) at study entry, Diagnosis based on clinical symptoms | 123 |
| Table B-7.4.7 | Age (years) at study entry, Germany | 123 |
| Table B-7.4.8 | Age (years) at study entry, Poland | 123 |
| Table B-7.4.9 | Age (years) at study entry, Hungary | 123 |
| Table B-7.4.10 | Age (years) at study entry, Switzerland | 123 |
| Table B-7.4.11 | Age (years) at study entry, Russia | 123 |
| Table B-7.4.12 | Age (years) at study entry, Ukraine | 123 |
| Section B-7.5 | Body Mass Index (BMI) at study entry | 124 |
| Table B-7.5.1 | Body Mass Index (BMI) at study entry | 124 |
| Table B-7.5.2 | Body Mass Index (BMI) at study entry, Starter | 125 |
| Table B-7.5.3 | Body Mass Index (BMI) at study entry, Switcher | 125 |
| Table B-7.5.4 | Body Mass Index (BMI) at study entry, Restarter | 125 |
| Table B-7.5.5 | Body Mass Index (BMI) at study entry, Diagnosis confirmed by surgery | 125 |
| Table B-7.5.6 | Body Mass Index (BMI) at study entry, Diagnosis based on clinical symptoms | 125 |
| Table B-7.5.7 | Body Mass Index (BMI) at study entry, Germany | 125 |
| Table B-7.5.8 | Body Mass Index (BMI) at study entry, Poland | 125 |
| Table B-7.5.9 | Body Mass Index (BMI) at study entry, Hungary | 125 |
| Table B-7.5.10 | Body Mass Index (BMI) at study entry, Switzerland | 125 |



| Table B-7.5.11 | Body Mass Index (BMI) at study entry, Russia | 125 |
|---|---|---|
| Table B-7.5.12 | Body Mass Index (BMI) at study entry, Ukraine | 125 |
| Section B-7.6 | Endometriosis associated symptoms at study entry | 126 |
| Table B-7.6.1 | Endometriosis associated symptoms at study entry | 126 |
| Table B-7.6.2 | Endometriosis associated symptoms at study entry, Starter | 127 |
| Table B-7.6.3 | Endometriosis associated symptoms at study entry, Switcher | 127 |
| Table B-7.6.4 | Endometriosis associated symptoms at study entry, Restarter | 127 |
| Table B-7.6.5 | Endometriosis associated symptoms at study entry, Diagnosis confirmed by surgery | 127 |
| Table B-7.6.6 | Endometriosis associated symptoms at study entry, Diagnosis based on clinical symptoms | 127 |
| Table B-7.6.7 | Endometriosis associated symptoms at study entry, Germany | 127 |
| Table B-7.6.8 | Endometriosis associated symptoms at study entry, Poland | 127 |
| Table B-7.6.9 | Endometriosis associated symptoms at study entry, Hungary | 127 |
| Table B-7.6.10 | Endometriosis associated symptoms at study entry, Switzerland | 127 |
| Table B-7.6.11 | Endometriosis associated symptoms at study entry, Russia | 127 |
| Table B-7.6.12 | Endometriosis associated symptoms at study entry, Ukraine | 127 |
| Section B-7.7 | Endometriosis associated pain severity score at study entry | 128 |
| Table B-7.7.1 | Endometriosis associated pain severity score at study entry | 128 |
| Table B-7.7.2 | Endometriosis associated pain severity score at study entry, Starter | 129 |
| Table B-7.7.3 | Endometriosis associated pain severity score at study entry, Switcher | |
| Table B-7.7.4 | Endometriosis associated pain severity score at study entry, Restarter | 129 |
| Table B-7.7.5 | Endometriosis associated pain severity score at study entry, Diagnosis confirmed by surgery | 129 |
| Table B-7.7.6 | Endometriosis associated pain severity score at study entry, Diagnosis based on clinical symptoms | 129 |
| Table B-7.7.7 | Endometriosis associated pain severity score at study entry, Germany | 129 |
| Table B-7.7.8 | Endometriosis associated pain severity score at study entry, Poland | 129 |
| Table B-7.7.9 | Endometriosis associated pain severity score at study entry, Hungary | |
| Table B-7.7.10 | Endometriosis associated pain severity score at study entry, Switzerland | |
| Table B-7.7.11 | Endometriosis associated pain severity score at study entry, Russia | |
| Table B-7.7.12 | Endometriosis associated pain severity score at study entry, Ukraine | |
| Section B-8 Follo | w-up characteristics | |
| Section B-8.1 | Mood symptoms at study entry | 130 |



| Table B-8.1.1 | Mood symptoms at study entry, ITT population, Complete cohort | 130 |
|---|---|---|
| Table B-8.1.2 | Mood symptoms at study entry, AT population, Complete cohort | 131 |
| Table B-8.1.3 | Mood symptoms at study entry, AT population, Starter | 131 |
| Table B-8.1.4 | Mood symptoms at study entry, AT population, Switcher | 131 |
| Table B-8.1.5 | Mood symptoms at study entry, AT population, Restarter | 131 |
| Table B-8.1.6 | Mood symptoms at study entry, AT population, Diagnosis confirmed by surgery | 131 |
| Table B-8.1.7 | Mood symptoms at study entry, AT population, Diagnosis based on clinical symptoms | 131 |
| Table B-8.1.8 | Mood symptoms at study entry, AT population, Germany | 131 |
| Table B-8.1.9 | Mood symptoms at study entry, AT population, Poland | 131 |
| Table B-8.1.10 | Mood symptoms at study entry, AT population, Hungary | 131 |
| Table B-8.1.11 | Mood symptoms at study entry, AT population, Switzerland | 131 |
| Table B-8.1.12 | Mood symptoms at study entry, AT population, Russia | 131 |
| Table B-8.1.13 | Mood symptoms at study entry, AT population, Ukraine | 131 |
| Section B-8.2 | Mood symptoms at 6 months after study entry | 132 |
| Table B-8.2.1 | Mood symptoms at 6 months after study entry, ITT population, Complete cohort | 132 |
| Table B-8.2.2 | Mood symptoms at 6 months after study entry, AT population, Complete cohort | 132 |
| Table B-8.2.3 | Mood symptoms at 6 months after study entry, AT population, Starter | 133 |
| Table B-8.2.4 | Mood symptoms at 6 months after study entry, AT population, Switcher | 133 |
| Table B-8.2.5 | Mood symptoms at 6 months after study entry, AT population, Restarter | 133 |
| Table B-8.2.6 | Mood symptoms at 6 months after study entry, AT population, Diagnosis confirmed by surgery | 133 |
| Table B-8.2.7 | Mood symptoms at 6 months after study entry, AT population, Diagnosis based on clinical symptoms | 133 |
| Table B-8.2.8 | Mood symptoms at 6 months after study entry, AT population, Germany | 133 |
| Table B-8.2.9 | Mood symptoms at 6 months after study entry, AT population, Poland | 133 |
| Table B-8.2.10 | Mood symptoms at 6 months after study entry, AT population, Hungary | 133 |
| Table B-8.2.11 | Mood symptoms at 6 months after study entry, AT population, Switzerland | 133 |
| Table B-8.2.12 | Mood symptoms at 6 months after study entry, AT population, Russia | 133 |
| Table B-8.2.13 | Mood symptoms at 6 months after study entry, AT population, Ukraine | 133 |
| Section B-8.3 | Mood symptoms at 12 months after study entry | 134 |
| Table B-8.3.1 | Mood symptoms at 12 months after study entry, ITT population, Complete cohort | 134 |
| Table B-8.3.2 | Mood symptoms at 12 months after study entry, AT population, Complete cohort | 134 |



| Table B-8.3.3 | Mood symptoms at 12 months after study entry, AT population, Starter | 134 |
|---|---|---|
| Table B-8.3.4 | Mood symptoms at 12 months after study entry, AT population, Switcher | 134 |
| Table B-8.3.5 | Mood symptoms at 12 months after study entry, AT population, Restarter | 134 |
| Table B-8.3.6 | Mood symptoms at 12 months after study entry, AT population, Diagnosis confirmed by surgery | 134 |
| Table B-8.3.7 | Mood symptoms at 12 months after study entry, AT population, Diagnosis based on clinical symptoms | 134 |
| Table B-8.3.8 | Mood symptoms at 12 months after study entry, AT population, Germany | 134 |
| Table B-8.3.9 | Mood symptoms at 12 months after study entry, AT population, Poland | 134 |
| Table B-8.3.10 | Mood symptoms at 12 months after study entry, AT population, Hungary | 134 |
| Table B-8.3.11 | Mood symptoms at 12 months after study entry, AT population, Switzerland | 134 |
| Table B-8.3.12 | Mood symptoms at 12 months after study entry, AT population, Russia | 134 |
| Table B-8.3.13 | Mood symptoms at 12 months after study entry, AT population, Ukraine | 134 |
| Section B-8.4 | Mood symptoms at 24 months after study entry | 134 |
| Table B-8.4.1 | Mood symptoms at 24 months after study entry, ITT population, Complete cohort | 134 |
| Table B-8.4.2 | Mood symptoms at 24 months after study entry, AT population, Complete cohort | 134 |
| Table B-8.4.3 | Mood symptoms at 24 months after study entry, AT population, Starter | 134 |
| Table B-8.4.4 | Mood symptoms at 24 months after study entry, AT population, Switcher | 134 |
| Table B-8.4.5 | Mood symptoms at 24 months after study entry, AT population, Restarter | 134 |
| Table B-8.4.6 | Mood symptoms at 24 months after study entry, AT population, Diagnosis confirmed by surgery | 134 |
| Table B-8.4.7 | Mood symptoms at 24 months after study entry, AT population, Diagnosis based on clinical symptoms | 134 |
| Table B-8.4.8 | Mood symptoms at 24 months after study entry, AT population, Germany | 134 |
| Table B-8.4.9 | Mood symptoms at 24 months after study entry, AT population, Poland | 135 |
| Table B-8.4.10 | Mood symptoms at 24 months after study entry, AT population, Hungary | 135 |
| Table B-8.4.11 | Mood symptoms at 24 months after study entry, AT population, Switzerland | 135 |
| Table B-8.4.12 | Mood symptoms at 24 months after study entry, AT population, Russia | 135 |
| Table B-8.4.13 | Mood symptoms at 24 months after study entry, AT population, Ukraine | 135 |
| Section B-8.5 | Mood symptoms at 36 months after study entry | 135 |
| Table B-8.5.1 | Mood symptoms at 36 months after study entry, ITT population, Complete cohort | 135 |
| Table B-8.5.2 | Mood symptoms at 36 months after study entry, AT population, Complete cohort | 135 |
| Table B-8.5.3 | Mood symptoms at 36 months after study entry, AT population, Starter | 135 |
| Table B-8.5.4 | Mood symptoms at 36 months after study entry, AT population, Switcher | 135 |



| Table B-8.5.5 | Mood symptoms at 36 months after study entry, AT population, Restarter | 135 |
|---|---|---|
| Table B-8.5.6 | Mood symptoms at 36 months after study entry, AT population, Diagnosis confirmed by surgery | 135 |
| Table B-8.5.7 | Mood symptoms at 36 months after study entry, AT population, Diagnosis based on clinical symptoms | 135 |
| Table B-8.5.8 | Mood symptoms at 36 months after study entry, AT population, Germany | 135 |
| Table B-8.5.9 | Mood symptoms at 36 months after study entry, AT population, Poland | 135 |
| Table B-8.5.10 | Mood symptoms at 36 months after study entry, AT population, Hungary | 135 |
| Table B-8.5.11 | Mood symptoms at 36 months after study entry, AT population, Switzerland | 135 |
| Table B-8.5.12 | Mood symptoms at 36 months after study entry, AT population, Russia | 135 |
| Table B-8.5.13 | Mood symptoms at 36 months after study entry, AT population, Ukraine | 135 |
| Section B-8.6 | Mood symptoms at 48 months after study entry | 135 |
| Table B-8.6.1 | Mood symptoms at 48 months after study entry, ITT population, Complete cohort | 135 |
| Table B-8.6.2 | Mood symptoms at 48 months after study entry, AT population, Complete cohort | 135 |
| Table B-8.6.3 | Mood symptoms at 48 months after study entry, AT population, Starter | 136 |
| Table B-8.6.4 | Mood symptoms at 48 months after study entry, AT population, Switcher | 136 |
| Table B-8.6.5 | Mood symptoms at 48 months after study entry, AT population, Restarter | 136 |
| Table B-8.6.6 | Mood symptoms at 48 months after study entry, AT population, Diagnosis confirmed by surgery | 136 |
| Table B-8.6.7 | Mood symptoms at 48 months after study entry, AT population, Diagnosis based on clinical symptoms | 136 |
| Table B-8.6.8 | Mood symptoms at 48 months after study entry, AT population, Germany | 136 |
| Table B-8.6.9 | Mood symptoms at 48 months after study entry, AT population, Poland | 136 |
| Table B-8.6.10 | Mood symptoms at 48 months after study entry, AT population, Hungary | |
| Table B-8.6.11 | Mood symptoms at 48 months after study entry, AT population, Switzerland | 136 |
| Table B-8.6.12 | Mood symptoms at 48 months after study entry, AT population, Russia | 136 |
| Table B-8.6.13 | Mood symptoms at 48 months after study entry, AT population, Ukraine | 136 |
| Section B-8.7 | Mood symptoms at 60 months after study entry | 136 |
| Table B-8.7.1 | Mood symptoms at 60 months after study entry, ITT population, Complete cohort | 136 |
| Table B-8.7.2 | Mood symptoms at 60 months after study entry, AT population, Complete cohort | 136 |
| Table B-8.7.3 | Mood symptoms at 60 months after study entry, AT population, Starter | 136 |
| Table B-8.7.4 | Mood symptoms at 60 months after study entry, AT population, Switcher | 136 |
| Table B-8.7.5 | Mood symptoms at 60 months after study entry, AT population, Restarter | 136 |
| Table B-8.7.6 | Mood symptoms at 60 months after study entry, AT population, Diagnosis confirmed by surgery | 136 |



| Table B-8.7.7 | Mood symptoms at 60 months after study entry, AT population, Diagnosis based on clinical symptoms | 136 |
|---|---|---|
| Table B-8.7.8 | Mood symptoms at 60 months after study entry, AT population, Germany | 136 |
| Table B-8.7.9 | Mood symptoms at 60 months after study entry, AT population, Poland | 136 |
| Table B-8.7.10 | Mood symptoms at 60 months after study entry, AT population, Hungary | 136 |
| Table B-8.7.11 | Mood symptoms at 60 months after study entry, AT population, Switzerland | 136 |
| Table B-8.7.12 | Mood symptoms at 60 months after study entry, AT population, Russia | 136 |
| Table B-8.7.13 | Mood symptoms at 60 months after study entry, AT population, Ukraine | 137 |
| Section B-8.8 | Mood symptoms at 72 months after study entry | 137 |
| Table B-8.8.1 | Mood symptoms at 72 months after study entry, ITT population, Complete cohort | 137 |
| Table B-8.8.2 | Mood symptoms at 72 months after study entry, AT population, Complete cohort | 137 |
| Table B-8.8.3 | Mood symptoms at 72 months after study entry, AT population, Starter | 137 |
| Table B-8.8.4 | Mood symptoms at 72 months after study entry, AT population, Switcher | 137 |
| Table B-8.8.5 | Mood symptoms at 72 months after study entry, AT population, Restarter | 137 |
| Table B-8.8.6 | Mood symptoms at 72 months after study entry, AT population, Diagnosis confirmed by surgery | 137 |
| Table B-8.8.7 | Mood symptoms at 72 months after study entry, AT population, Diagnosis based on clinical symptoms | 137 |
| Table B-8.8.8 | Mood symptoms at 72 months after study entry, AT population, Germany | 137 |
| Table B-8.8.9 | Mood symptoms at 72 months after study entry, AT population, Poland | 137 |
| Table B-8.8.10 | Mood symptoms at 72 months after study entry, AT population, Hungary | 137 |
| Table B-8.8.11 | Mood symptoms at 72 months after study entry, AT population, Switzerland | 137 |
| Table B-8.8.12 | Mood symptoms at 72 months after study entry, AT population, Russia | 137 |
| Table B-8.8.13 | Mood symptoms at 72 months after study entry, AT population, Ukraine | 137 |
| Section B-8.9 | Mood symptoms at 84 months after study entry | 137 |
| Table B-8.9.1 | Mood symptoms at 84 months after study entry, ITT population, Complete cohort | 137 |
| Table B-8.9.2 | Mood symptoms at 84 months after study entry, AT population, Complete cohort | 137 |
| Table B-8.9.3 | Mood symptoms at 84 months after study entry, AT population, Starter | 137 |
| Table B-8.9.4 | Mood symptoms at 84 months after study entry, AT population, Switcher | 137 |
| Table B-8.9.5 | Mood symptoms at 84 months after study entry, AT population, Restarter | 137 |
| Table B-8.9.6 | Mood symptoms at 84 months after study entry, AT population, Diagnosis confirmed by surgery | 137 |
| Table B-8.9.7 | Mood symptoms at 84 months after study entry, AT population, Diagnosis based on clinical symptoms | 138 |
| Table B-8.9.8 | Mood symptoms at 84 months after study entry, AT population, Germany | 138 |



| Table B-8.9.9 | Mood symptoms at 84 months after study entry, AT population, Poland | 138 |
|---|---|---|
| Table B-8.9.10 | Mood symptoms at 84 months after study entry, AT population, Hungary | 138 |
| Table B-8.9.11 | Mood symptoms at 84 months after study entry, AT population, Switzerland | 138 |
| Table B-8.9.12 | Mood symptoms at 84 months after study entry, AT population, Russia | 138 |
| Table B-8.9.13 | Mood symptoms at 84 months after study entry, AT population, Ukraine | 138 |
| Section B-8.10 | Change of Mood Score after study entry, constant user only | 139 |
| Table B-8.10.1 | Change of Mood Score after study entry, constant user only*, AT population, Complete cohort | 139 |
| Table B-8.10.2 | Change of Mood Score after study entry, constant user only*, AT population, Starter | 140 |
| Table B-8.10.3 | Change of Mood Score after study entry, constant user only *, AT population, Switcher | 140 |
| Table B-8.10.4 | Change of Mood Score after study entry, constant user only *, AT population, Restarter | 140 |
| Table B-8.10.5 | Change of Mood Score after study entry, constant user only *, AT population, Diagnosis confirmed by surgery | 140 |
| Table B-8.10.6 | Change of Mood Score after study entry, constant user only *, AT population, Diagnosis based on clinical symptoms | 140 |
| Table B-8.10.7 | Change of Mood Score after study entry, constant user only *, AT population, Germany | 140 |
| Table B-8.10.8 | Change of Mood Score after study entry, constant user only *, AT population, Poland | 140 |
| Table B-8.10.9 | Change of Mood Score after study entry, constant user only *, AT population, Hungary | 140 |
| Table B-8.10.10 | Change of Mood Score after study entry, constant user only *, AT population, Switzerland | 140 |
| Table B-8.10.11 | Change of Mood Score after study entry, constant user only *, AT population, Russia | 140 |
| Table B-8.10.12 | Change of Mood Score after study entry, constant user only *, AT population, Ukraine | 140 |
| Section B-8.11 | Change of Mood Score after study entry, switcher only | 141 |
| Table B-8.11.1 | Change of Mood Score after study entry, switcher only *, AT population, Complete cohort | 141 |
| Table B-8.11.2 | Change of Mood Score after study entry, switcher only *, AT population, Starter | 142 |
| Table B-8.11.3 | Change of Mood Score after study entry, switcher only *, AT population, Switcher | 142 |
| Table B-8.11.4 | Change of Mood Score after study entry, switcher only *, AT population, Restarter | 142 |
| Table B-8.11.5 | Change of Mood Score after study entry, switcher only *, AT population, Diagnosis confirmed by surgery | 142 |
| Table B-8.11.6 | Change of Mood Score after study entry, switcher only *, AT population, Diagnosis based on clinical symptoms | 142 |
| Table B-8.11.7 | Change of Mood Score after study entry, switcher only *, AT population, Germany | 142 |
| Table B-8.11.8 | Change of Mood Score after study entry, switcher only *, AT population, Poland | 142 |
| Table B-8.11.9 | Change of Mood Score after study entry, switcher only *, AT population, Hungary | 142 |
| Table B-8.11.10 | Change of Mood Score after study entry, switcher only *, AT population, Switzerland | 142 |
| Table B-8.11.11 | Change of Mood Score after study entry, switcher only *, AT population, Russia | 142 |



| Table B-8.11.12 | Change of Mood Score after study entry, switcher only *, AT population, Ukraine | 142 |
|---|---|---|
| Section B-8.12 | Cohort status/switch of women during follow-up | 143 |
| Table B-8.12.1 | Cohort status/switch of women during follow-up, AT population, Complete cohort | 143 |
| Table B-8.12.2 | Cohort status/switch of women during follow-up, AT population, Starter | 144 |
| Table B-8.12.3 | Cohort status/switch of women during follow-up, AT population, Switcher | 144 |
| Table B-8.12.4 | Cohort status/switch of women during follow-up, AT population, Restarter | 144 |
| Table B-8.12.5 | Cohort status/switch of women during follow-up, AT population, Diagnosis confirmed by surgery | 144 |
| Table B-8.12.6 | Cohort status/switch of women during follow-up, AT population, Diagnosis based on clinical symptoms | 144 |
| Table B-8.12.7 | Cohort status/switch of women during follow-up, AT population, Germany | 144 |
| Table B-8.12.8 | Cohort status/switch of women during follow-up, AT population, Poland | 144 |
| Table B-8.12.9 | Cohort status/switch of women during follow-up, AT population, Hungary | 144 |
| Table B-8.12.10 | Cohort status/switch of women during follow-up, AT population, Switzerland | 144 |
| Table B-8.12.11 | Cohort status/switch of women during follow-up, AT population, Russia | 144 |
| Table B-8.12.12 | Cohort status/switch of women during follow-up, AT population, Ukraine | 144 |
| Section B-9 Summ | nary tables of selected baseline characteristics | 145 |
| Section B-9.1 | Selected baseline characteristics | 145 |
| Table B-9.1.1 | Selected baseline characteristics, ITT population, Complete cohort | 145 |
| Table B-9.1.2 | Selected baseline characteristics, AT population, Complete cohort | 147 |
| Table B-9.1.3 | Selected baseline characteristics, AT population, Starter | 147 |
| Table B-9.1.4 | Selected baseline characteristics, AT population, Switcher | 147 |
| Table B-9.1.5 | Selected baseline characteristics, AT population, Restarter | 147 |
| Table B-9.1.6 | Selected baseline characteristics, AT population, Diagnosis confirmed by surgery | 147 |
| Table B-9.1.7 | Selected baseline characteristics, AT population, Diagnosis based on clinical symptoms | 147 |
| Table B-9.1.8 | Selected baseline characteristics, AT population, Germany | 147 |
| Table B-9.1.9 | Selected baseline characteristics, AT population, Poland | 147 |
| Table B-9.1.10 | Selected baseline characteristics, AT population, Hungary | 147 |
| Table B-9.1.11 | Selected baseline characteristics, AT population, Switzerland | 147 |
| Table B-9.1.12 | Selected baseline characteristics, AT population, Russia | 147 |
| Table B-9.1.13 | Selected baseline characteristics, AT population, Ukraine | 147 |
| Section B-9.2 | Selected baseline characteristics by age categories | 148 |



| Table B-9.2.1 | Selected baseline characteristics, Adolescence, ITT population | 148 |
|---|---|---|
| Table B-9.2.2 | Selected baseline characteristics, Adolescence, AT population | 148 |
| Table B-9.2.3 | Selected baseline characteristics, Women <20 years, ITT population | 148 |
| Table B-9.2.4 | Selected baseline characteristics, Women <20 years, AT population | 148 |
| Table B-9.2.5 | Selected baseline characteristics Women >=20 and < 30 years, ITT population | 148 |
| Table B-9.2.6 | Selected baseline characteristics Women >=20 and < 30 years, AT population | 148 |
| Table B-9.2.7 | Selected baseline characteristics, Women >=30 and < 40 years, ITT population | 148 |
| Table B-9.2.8 | Selected baseline characteristics, Women >=30 and < 40 years, AT population | 148 |
| Table B-9.2.9 | Selected baseline characteristics, Women >=40 years, ITT population | 148 |
| Table B-9.2.10 | Selected baseline characteristics, Women >=40 years, AT population | 148 |
| Table B-9.2.11 | Selected baseline characteristics, age-standardized, ITT population | 148 |
| Table B-9.2.12 | Selected baseline characteristics, age-standardized, AT population | |
| Section B-9.3 | Selected baseline characteristics for women with treatment failure | 149 |
| Table B-9.3.1 | Selected baseline characteristics for women with treatment failure, AT population, Complete cohort | 149 |
| Table B-9.3.2 | Selected baseline characteristics for women with treatment failure, AT population, Starter | 150 |
| Table B-9.3.3 | Selected baseline characteristics for women with treatment failure, AT population, Switcher | 150 |
| Table B-9.3.4 | Selected baseline characteristics for women with treatment failure, AT population, Restarter | 150 |
| Section B-9.4 | Selected baseline characteristics for women who switched | |
| Table B-9.4.1 | Selected baseline characteristics for women who switched, AT population | |
| Table B-9.4.2 | Selected baseline characteristics for women who switched, Starter | |
| Table B-9.4.3 | Selected baseline characteristics for women who switched, Switcher | 152 |
| Table B-9.4.4 | Selected baseline characteristics for women who switched, Restarter | 152 |
| Section C Clinical O | utcome | 153 |
| Section C-1 Prima | ıry outcomes | |
| Section C-1.1 | Incidence rate of clinically relevant anemia | 153 |
| Table C-1.1.1 | Incidence rate of clinically relevant anemia, ITT population, Complete cohort | |
| Table C-1.1.2 | Incidence rate of newly diagnosed or reoccurrence of anemia, AT population, Complete cohort | 154 |
| Table C-1.1.3 | Incidence rate of newly diagnosed or reoccurrence of anemia, AT population, Starter | |
| Table C-1.1.4 | Incidence rate of newly diagnosed or reoccurrence of anemia, AT population, Switcher | 154 |
| Table C-1.1.5 | Incidence rate of newly diagnosed or reoccurrence of anemia, AT population, Restarter | 154 |



| Table C-1.1.6 | Incidence rate of newly diagnosed or reoccurrence of anemia, AT population, Diagnosis confirmed by surgery | 154 |
|---|---|---|
| Table C-1.1.7 | Incidence rate of newly diagnosed or reoccurrence of anemia, AT population, Diagnosis based on clinical symptoms | 154 |
| Table C-1.1.8 | Incidence rate of newly diagnosed or reoccurrence of anemia, AT population, Germany | 154 |
| Table C-1.1.9 | Incidence rate of newly diagnosed or reoccurrence of anemia, AT population, Poland | 154 |
| Table C-1.1.10 | Incidence rate of newly diagnosed or reoccurrence of anemia, AT population, Hungary | 154 |
| Table C-1.1.11 | Incidence rate of newly diagnosed or reoccurrence of anemia, AT population, Switzerland | 154 |
| Table C-1.1.12 | Incidence rate of newly diagnosed or reoccurrence of anemia, AT population, Russia | 154 |
| Table C-1.1.13 | Incidence rate of newly diagnosed or reoccurrence of anemia, AT population, Ukraine | 154 |
| Section C-1.2 | Incidence rate of new depression or worsening of existing depression | 155 |
| Table C-1.2.1 | Incidence rate of new depression or worsening of existing depression, ITT population, Complete cohort | 155 |
| Table C-1.2.2 | Incidence rate of new depression or worsening of existing depression, AT population, Complete cohort | 156 |
| Table C-1.2.3 | Incidence rate of new depression or worsening of existing depression, AT population, Starter | 156 |
| Table C-1.2.4 | Incidence rate of new depression or worsening of existing depression, AT population, Switcher | 156 |
| Table C-1.2.5 | Incidence rate of new depression or worsening of existing depression, AT population, Restarter | 156 |
| Table C-1.2.6 | Incidence rate of new depression or worsening of existing depression, AT population, Diagnosis confirmed by surgery | 156 |
| Table C-1.2.7 | Incidence rate of new depression or worsening of existing depression, AT population, Diagnosis based on clinical symptoms | 156 |
| Table C-1.2.8 | Incidence rate of new depression or worsening of existing depression, AT population, Germany | 156 |
| Table C-1.2.9 | Incidence rate of new depression or worsening of existing depression, AT population, Poland | 156 |
| Table C-1.2.10 | Incidence rate of new depression or worsening of existing depression, AT population, Hungary | 156 |
| Table C-1.2.11 | Incidence rate of new depression or worsening of existing depression, AT population, Switzerland | 156 |
| Table C-1.2.12 | Incidence rate of new depression or worsening of existing depression, AT population, Russia | 156 |
| Table C-1.2.13 | Incidence rate of new depression or worsening of existing depression, AT population, Ukraine | 156 |
| Section C-1.3 | Incidence proportions of treatment discontinuation due to treatment failure and due to other reasons | 157 |
| Table C-1.3.1 | Incidence proportions of treatment discontinuation due to treatment failure and due to other reasons, AT population, Complete | cohort 157 |
| Table C-1.3.2 | Incidence proportions of treatment discontinuation due to treatment failure and due to other reasons, AT population, Starter | 158 |
| Table C-1.3.3 | Incidence proportions of treatment discontinuation due to treatment failure and due to other reasons, AT population, Switcher | 158 |
| Table C-1.3.4 | Incidence proportions of treatment discontinuation due to treatment failure and due to other reasons, AT population, Restarter. | 158 |
| Table C-1.3.5 | Incidence proportions of treatment discontinuation due to treatment failure and due to other reasons, AT population, Diagnosis | confirmed |
| by surgery | 158 | |



| Table C-1.3.6 | Incidence proportions of treatment discontinuation due to treatment failure and due to other reasons, AT population, Diagnosis based | on |
|---|---|---|
| clinical symptoms | 158 | |
| Table C-1.3.7 | Incidence proportions of treatment discontinuation due to treatment failure and due to other reasons, AT population, Germany | 158 |
| Table C-1.3.8 | Incidence proportions of treatment discontinuation due to treatment failure and due to other reasons, AT population, Poland | 158 |
| Table C-1.3.9 | Incidence proportions of treatment discontinuation due to treatment failure and due to other reasons, AT population, Hungary | 158 |
| Table C-1.3.10 | Incidence proportions of treatment discontinuation due to treatment failure and due to other reasons, AT population, Switzerland | 158 |
| Table C-1.3.11 | Incidence proportions of treatment discontinuation due to treatment failure and due to other reasons, AT population, Russia | 158 |
| Table C-1.3.12 | Incidence proportions of treatment discontinuation due to treatment failure and due to other reasons, AT population, Ukraine | 158 |
| Section C-2 Second | dary outcomes | 159 |
| Section C-2.1 | Incidence proportions of treatment discontinuation unrelated to treatment failure | 159 |
| Table C-2.1.1 | Incidence proportions of treatment discontinuation unrelated to treatment failure, AT population, Complete cohort | 159 |
| Table C-2.1.2 | Incidence proportions of treatment discontinuation unrelated to treatment failure, AT population, Starter | 160 |
| Table C-2.1.3 | Incidence proportions of treatment discontinuation unrelated to treatment failure, AT population, Switcher | 160 |
| Table C-2.1.4 | Incidence proportions of treatment discontinuation unrelated to treatment failure, AT population, Restarter | 160 |
| Table C-2.1.5 | Incidence proportions of treatment discontinuation unrelated to treatment failure, AT population, Diagnosis confirmed by surgery | 160 |
| Table C-2.1.6 | Incidence proportions of treatment discontinuation unrelated to treatment failure, AT population, Diagnosis based on clinical sympton | ns . 160 |
| Table C-2.1.7 | Incidence proportions of treatment discontinuation unrelated to treatment failure, AT population, Germany | 160 |
| Table C-2.1.8 | Incidence proportions of treatment discontinuation unrelated to treatment failure, AT population, Poland | 160 |
| Table C-2.1.9 | Incidence proportions of treatment discontinuation unrelated to treatment failure, AT population, Hungary | 160 |
| Table C-2.1.10 | Incidence proportions of treatment discontinuation unrelated to treatment failure, AT population, Switzerland | 160 |
| Table C-2.1.11 | Incidence proportions of treatment discontinuation unrelated to treatment failure, AT population, Russia | 160 |
| Table C-2.1.12 | Incidence proportions of treatment discontinuation unrelated to treatment failure, AT population, Ukraine | 160 |
| Section C-2.2 | Incidence rate of clinically relevant anemia for adolescence | 161 |
| Table C-2.2.1 | Incidence rate of clinically relevant anemia for adolescence*, AT population, Complete cohort | 161 |
| Table C-2.2.2 | Incidence rate of clinically relevant anemia for adolescence*, AT population, Starter | 162 |
| Table C-2.2.3 | Incidence rate of clinically relevant anemia for adolescence*, AT population, Switcher | 162 |
| Table C-2.2.4 | Incidence rate of clinically relevant anemia for adolescence*, AT population, Restarter | 162 |
| Table C-2.2.5 | Incidence rate of clinically relevant anemia for adolescence*, AT population, Diagnosis confirmed by surgery | 162 |
| Table C-2.2.6 | Incidence rate of clinically relevant anemia for adolescence*, AT population, Diagnosis based on clinical symptoms | 162 |
| Table C-2.2.7 | Incidence rate of clinically relevant of anemia for adolescence*, AT population, Germany | 162 |



| Table C-2.2.8 | Incidence rate of clinically relevant of anemia for adolescence*, AT population, Poland | 162 |
|---|---|---|
| Table C-2.2.9 | Incidence rate of clinically relevant anemia for adolescence*, AT population, Hungary | |
| Table C-2.2.10 | Incidence rate of clinically relevant anemia for adolescence*, AT population, Switzerland | |
| Table C-2.2.11 | Incidence rate of clinically relevant anemia for adolescence*, AT population, Russia | |
| Table C-2.2.12 | Incidence rate of clinically relevant anemia for adolescence*, AT population, Ukraine | |
| Section C-2.3 | Incidence rate of new depression or worsening of existing depression for adolescence | |
| Table C-2.3.1 | Incidence rate of new depression or worsening of existing depression for adolescence*, AT population, Complete cohort | |
| Table C-2.3.2 | Incidence rate of new depression or worsening of existing depression for adolescence*, AT population, Starter | |
| Table C-2.3.3 | Incidence rate of new depression or worsening of existing depression for adolescence*, AT population, Switcher | |
| Table C-2.3.4 | Incidence rate of new depression or worsening of existing depression for adolescence*, AT population, Restarter | |
| Table C-2.3.5 | Incidence rate of new depression or worsening of existing depression for adolescence*, AT population, Diagnosis confirmed by sur | |
| Table C-2.3.6 | Incidence rate of new depression or worsening of existing depression for adolescence*, AT population, Diagnosis based on clinical | |
| | 164 | , , |
| Table C-2.3.7 | Incidence rate of new depression or worsening of existing depression for adolescence*, AT population, Germany | 164 |
| Table C-2.3.8 | Incidence rate of new depression or worsening of existing depression for adolescence*, AT population, Poland | |
| Table C-2.3.9 | Incidence rate of new depression or worsening of existing depression for adolescence*, AT population, Hungary | 164 |
| Table C-2.3.10 | Incidence rate of new depression or worsening of existing depression for adolescence*, AT population, Switzerland | |
| Table C-2.3.11 | Incidence rate of new depression or worsening of existing depression for adolescence*, AT population, Russia | |
| Table C-2.3.12 | Incidence rate of new depression or worsening of existing depression for adolescence*, AT population, Ukraine | 164 |
| Section C-2.4 | Incidence proportions of treatment discontinuation for adolescence | 165 |
| Table C-2.4.1 | Incidence proportions of treatment discontinuation for adolescence*, AT population, Complete cohort | |
| Table C-2.4.2 | Incidence proportions of treatment discontinuation for adolescence*, AT population, Starter | 166 |
| Table C-2.4.3 | Incidence proportions of treatment discontinuation for adolescence*, AT population, Switcher | |
| Table C-2.4.4 | Incidence proportions of treatment discontinuation for adolescence*, AT population, Restarter | 166 |
| Table C-2.4.5 | Incidence proportions of treatment discontinuation for adolescence*, AT population, Diagnosis confirmed by surgery | |
| Table C-2.4.6 | Incidence proportions of treatment discontinuation for adolescence*, AT population, Diagnosis based on clinical symptoms | |
| Table C-2.4.7 | Incidence proportions of treatment discontinuation for adolescence*, AT population, Germany | 166 |
| Table C-2.4.8 | Incidence proportions of treatment discontinuation for adolescence*, AT population, Poland | |
| Table C-2.4.9 | Incidence proportions of treatment discontinuation for adolescence*, AT population, HungaryHungary | |
| Table C-2.4.10 | Incidence proportions of treatment discontinuation for adolescence*, AT population, Switzerland | |



| Table C-2.4.11 | Incidence proportions of treatment discontinuation for adolescence*, AT population, Russia | 166 |
|---|---|---|
| Table C-2.4.12 | Incidence proportions of treatment discontinuation for adolescence*, AT population, UkraineUkraine | 166 |
| Section C-2.5 | Incidence rate of clinically relevant anemia for long-term use, AT population, Complete cohort | 167 |
| Table C-2.5.1 | Incidence rate of clinically relevant anemia for long-term use, AT population, Starter | 167 |
| Table C-2.5.2 | Incidence rate of clinically relevant anemia for long-term use, AT population, Switcher | |
| Table C-2.5.3 | Incidence rate of clinically relevant anemia for long-term use, AT population, Restarter | 167 |
| Table C-2.5.4 | Incidence rate of clinically relevant anemia for long-term use, AT population, Diagnosis confirmed by surgery | |
| Table C-2.5.5 | Incidence rate of clinically relevant anemia for long-term use, AT population, Diagnosis based on clinical symptoms | |
| Table C-2.5.6 | Incidence rate of clinically relevant anemia for long-term use, AT population, Germany | 167 |
| Table C-2.5.7 | Incidence rate of clinically relevant anemia for long-term use, AT population, Poland | 167 |
| Table C-2.5.8 | Incidence rate of clinically relevant anemia for long-term use, AT population, Hungary | |
| Table C-2.5.9 | Incidence rate of clinically relevant anemia for long-term use, AT population, Switzerland | |
| Table C-2.5.10 | Incidence rate of clinically relevant anemia for long-term use, AT population, Russia | |
| Table C-2.5.11 | Incidence rate of clinically relevant anemia for long-term use, AT population, Ukraine | 167 |
| Section C-2.6 | Incidence rate of new depression or worsening of existing depression for long-term use | |
| Table C-2.6.1 | Incidence rate of new depression or worsening of existing depression for long-term use, AT population, Complete cohort | 167 |
| Table C-2.6.2 | Incidence rate of new depression or worsening of existing depression for long-term use, AT population, Starter | 167 |
| Table C-2.6.3 | Incidence rate of new depression or worsening of existing depression for long-term use, AT population, Switcher | 167 |
| Table C-2.6.4 | Incidence rate of new depression or worsening of existing depression for long-term use, AT population, Restarter | 167 |
| Table C-2.6.5 | Incidence rate of new depression or worsening of existing depression for long-term use, AT population, Diagnosis confirmed by s | urgery 167 |
| Table C-2.6.6 | Incidence rate of new depression or worsening of existing depression for long-term use, AT population, Diagnosis based on clinical section of the contract of | al symptoms |
| Table C-2.6.7 | Incidence rate of new depression or worsening of existing depression for long-term use, AT population, Germany | 167 |
| Table C-2.6.8 | Incidence rate of new depression or worsening of existing depression for long-term use, AT population, Poland | 167 |
| Table C-2.6.9 | Incidence rate of new depression or worsening of existing depression for long-term use, AT population, Hungary | 167 |
| Table C-2.6.10 | Incidence rate of new depression or worsening of existing depression for long-term use, AT population, Switzerland | 168 |
| Table C-2.6.11 | Incidence rate of new depression or worsening of existing depression for long-term use, AT population, Russia | 168 |
| Table C-2.6.12 | Incidence rate of new depression or worsening of existing depression for long-term use, AT population, Ukraine | 168 |
| Section C-2.7 | Incidence proportions of treatment discontinuation for long-term use | 168 |
| Table C-2.7.1 | Incidence proportions of treatment discontinuation for long-term use, AT population, Complete cohort | 168 |



| Table C-2.7.2 | Incidence proportions of treatment discontinuation for long-term use, AT population, Starter | 168 |
|---|---|---|
| Table C-2.7.3 | Incidence proportions of treatment discontinuation for long-term use, AT population, Switcher | 168 |
| Table C-2.7.4 | Incidence proportions of treatment discontinuation for long-term use, AT population, Restarter | 168 |
| Table C-2.7.5 | Incidence proportions of treatment discontinuation for long-term use, AT population, Diagnosis confirmed by surgery | 168 |
| Table C-2.7.6 | Incidence proportions of treatment discontinuation for long-term use, AT population, Diagnosis based on clinical symptoms | 168 |
| Table C-2.7.7 | Incidence proportions of treatment discontinuation for long-term use, AT population, Germany | 168 |
| Table C-2.7.8 | Incidence proportions of treatment discontinuation for long-term use, AT population, Poland | 168 |
| Table C-2.7.9 | Incidence proportions of treatment discontinuation for long-term use, AT population, Hungary | 168 |
| Table C-2.7.10 | Incidence proportions of treatment discontinuation for long-term use, AT population, Switzerland | 168 |
| Table C-2.7.11 | Incidence proportions of treatment discontinuation for long-term use, AT population, Russia | 168 |
| Table C-2.7.12 | Incidence proportions of treatment discontinuation for long-term use, AT population, Ukraine | 168 |
| Section C-3 Other s | afety outcomes | 169 |
| Section C-3.1 | Incidence rate of confirmed thromboembolic events | 169 |
| Table C-3.1.1 | Incidence rate of confirmed thromboembolic events, AT population, Complete cohort | 169 |
| Table C-3.1.2 | Incidence rate of confirmed thromboembolic events, AT population, Starter | 170 |
| Table C-3.1.3 | Incidence rate of confirmed thromboembolic events, AT population, Switcher | 170 |
| Table C-3.1.4 | Incidence rate of confirmed thromboembolic events, AT population, Restarter | 170 |
| Table C-3.1.5 | Incidence rate of confirmed thromboembolic events, AT population, Diagnosis confirmed by surgery | 170 |
| Table C-3.1.6 | Incidence rate of confirmed thromboembolic events, AT population, Diagnosis based on clinical symptoms | 170 |
| Table C-3.1.7 | Incidence rate of confirmed thromboembolic events, AT population, Germany | 170 |
| Table C-3.1.8 | Incidence rate of confirmed thromboembolic events, AT population, Poland | 170 |
| Table C-3.1.9 | Incidence rate of confirmed thromboembolic events, AT population, Hungary | 170 |
| Table C-3.1.10 | Incidence rate of confirmed thromboembolic events, AT population, Switzerland | 170 |
| Table C-3.1.11 | Incidence rate of confirmed thromboembolic events, AT population, Russia | 170 |
| Table C-3.1.12 | Incidence rate of confirmed thromboembolic events, AT population, Ukraine | 170 |
| Section C-3.2 | Incidence rate of fatal cases (all deaths) | 171 |
| Table C-3.2.1 | Incidence rate of fatal cases (all deaths), AT population, Complete cohort | |
| Table C-3.2.2 | Incidence rate of fatal cases (all deaths), AT population, Starter | 172 |
| Table C-3.2.3 | Incidence rate of fatal cases (all deaths), AT population, Switcher | 172 |
| Table C-3.2.4 | Incidence rate of fatal cases (all deaths), AT population, Restarter | 172 |



| Table C-3.2.5 | Incidence rate of fatal cases (all deaths), AT population, Diagnosis confirmed by surgery | 172 |
|---|---|---|
| Table C-3.2.6 | Incidence rate of fatal cases (all deaths), AT population, Diagnosis based on clinical symptoms | 172 |
| Table C-3.2.7 | Incidence rate of fatal cases (all deaths), AT population, Germany | 172 |
| Table C-3.2.8 | Incidence rate of fatal cases (all deaths), AT population, Poland | 172 |
| Table C-3.2.9 | Incidence rate of fatal cases (all deaths), AT population, Hungary | 172 |
| Table C-3.2.10 | Incidence rate of fatal cases (all deaths), AT population, Switzerland | 172 |
| Table C-3.2.11 | Incidence rate of fatal cases (all deaths), AT population, Russia | 172 |
| Table C-3.2.12 | Incidence rate of fatal cases (all deaths), AT population, Ukraine | 172 |
| Section C-3.3 | Incidence rate of serious adverse events by organ system | 173 |
| Table C-3.3.1 | Incidence rate of serious adverse events by organ system, AT population, Complete cohort | 173 |
| Table C-3.3.2 | Incidence rate of serious adverse events by organ system, AT population, Starter | 175 |
| Table C-3.3.3 | Incidence rate of serious adverse events by organ system, AT population, Switcher | |
| Table C-3.3.4 | Incidence rate of serious adverse events by organ system, AT population, Restarter | 175 |
| Table C-3.3.5 | Incidence rate of serious adverse events by organ system, AT population, Diagnosis confirmed by surgery | 175 |
| Table C-3.3.6 | Incidence rate of serious adverse events by organ system, AT population, Diagnosis based on clinical symptoms | 175 |
| Table C-3.3.7 | Incidence rate of serious adverse events by organ system, AT population, Germany | 175 |
| Table C-3.3.8 | Incidence rate of serious adverse events by organ system, AT population, Poland | 175 |
| Table C-3.3.9 | Incidence rate of serious adverse events by organ system, AT population, Hungary | 175 |
| Table C-3.3.10 | Incidence rate of serious adverse events by organ system, AT population, Switzerland | 175 |
| Table C-3.3.11 | Incidence rate of serious adverse events by organ system, AT population, Russia | 175 |
| Table C-3.3.12 | Incidence rate of serious adverse events by organ system, AT population, Ukraine | 175 |
| Section C-3.4 | Incidence rate of serious adverse events by organ system for long-term use | 176 |
| Table C-3.4.1 | Incidence rate of serious adverse events by organ system for long-term use, AT population, Complete cohort | 176 |
| Table C-3.4.2 | Incidence rate of serious adverse events by organ system for long-term use, AT population, Starter | 177 |
| Table C-3.4.3 | Incidence rate of serious adverse events by organ system for long-term use, AT population, Switcher | 177 |
| Table C-3.4.4 | Incidence rate of serious adverse events by organ system for long-term use, AT population, Restarter | 177 |
| Table C-3.4.5 | Incidence rate of serious adverse events by organ system for long-term use, AT population, Diagnosis confirmed by surgery | 177 |
| Table C-3.4.6 | Incidence rate of serious adverse events by organ system for long-term use, AT population, Diagnosis based on clinical symptoms | 177 |
| Table C-3.4.7 | Incidence rate of serious adverse events by organ system for long-term use, AT population, Germany | 177 |
| Table C-3.4.8 | Incidence rate of serious adverse events by organ system for long-term use, AT population, Poland | 177 |



| Table C-3.4.10 Incidence rate of serious adverse events by organ system for long-term use, AT population, Switzerland | Table C-3.4.9 | Incidence rate of serious adverse events by organ system for long-term use, AT population, Hungary | 177 |
|---|---|---|---|
| Table C-3.4.12 Incidence rate of serious adverse events by organ system for long-term use, AT population, Ukraine | Table C-3.4.10 | Incidence rate of serious adverse events by organ system for long-term use, AT population, Switzerland | 178 |
| Incidence rate of malignant neoplasms by organ system, AT population, Complete cohort | Table C-3.4.11 | Incidence rate of serious adverse events by organ system for long-term use, AT population, Russia | 178 |
| Table C-3.5.1 Incidence rate of malignant neoplasms by organ system, AT population, Complete cohort | Table C-3.4.12 | Incidence rate of serious adverse events by organ system for long-term use, AT population, Ukraine | 178 |
| Table C-3.5.2Incidence rate of malignant neoplasms by organ system, AT population, Switcher18Table C-3.5.3Incidence rate of malignant neoplasms by organ system, AT population, Switcher18Table C-3.5.4Incidence rate of malignant neoplasms by organ system, AT population, Restarter18Table C-3.5.5Incidence rate of malignant neoplasms by organ system, AT population, Diagnosis confirmed by surgery18Table C-3.5.6Incidence rate of malignant neoplasms by organ system, AT population, Diagnosis based on clinical symptoms18Table C-3.5.7Incidence rate of malignant neoplasms by organ system, AT population, Germany18Table C-3.5.8Incidence rate of malignant neoplasms by organ system, AT population, Poland18Table C-3.5.9Incidence rate of malignant neoplasms by organ system, AT population, Hungary18Table C-3.5.10Incidence rate of malignant neoplasms by organ system, AT population, Switzerland18Table C-3.5.11Incidence rate of malignant neoplasms by organ system, AT population, Russia18Table C-3.5.12Incidence rate of malignant neoplasms by organ system, AT population, Russia18Table C-3.5.13Incidence proportion of malformations18Table C-3.6.1Incidence proportion of malformations, AT population, Complete cohort18Table C-3.6.2Incidence proportion of malformations, AT population, Switcher18Table C-3.6.3Incidence proportion of malformations, AT population, Diagnosis confirmed by surgery18Table C-3.6.5Incidence proportion of malformations, AT population, Diagnosis based on clinical s | Section C-3.5 | Incidence rate of malignant neoplasms by organ system | 179 |
| Table C-3.5.3Incidence rate of malignant neoplasms by organ system, AT population, Switcher18Table C-3.5.4Incidence rate of malignant neoplasms by organ system, AT population, Restarter.18Table C-3.5.5Incidence rate of malignant neoplasms by organ system, AT population, Diagnosis confirmed by surgery18Table C-3.5.6Incidence rate of malignant neoplasms by organ system, AT population, Diagnosis based on clinical symptoms18Table C-3.5.7Incidence rate of malignant neoplasms by organ system, AT population, Germany.18Table C-3.5.8Incidence rate of malignant neoplasms by organ system, AT population, Poland18Table C-3.5.9Incidence rate of malignant neoplasms by organ system, AT population, Hungary.18Table C-3.5.10Incidence rate of malignant neoplasms by organ system, AT population, Switzerland18Table C-3.5.11Incidence rate of malignant neoplasms by organ system, AT population, Switzerland18Table C-3.5.12Incidence rate of malignant neoplasms by organ system, AT population, Switzerland18Table C-3.6.1Incidence proportion of malformations18Table C-3.6.2Incidence proportion of malformations, AT population, Complete cohort18Table C-3.6.3Incidence proportion of malformations, AT population, Switcher18Table C-3.6.4Incidence proportion of malformations, AT population, Diagnosis confirmed by surgery18Table C-3.6.5Incidence proportion of malformations, AT population, Diagnosis based on clinical symptoms18Table C-3.6.6Incidence proportion of malformations, AT population, Diagn | Table C-3.5.1 | Incidence rate of malignant neoplasms by organ system, AT population, Complete cohort | 179 |
| Table C-3.5.4Incidence rate of malignant neoplasms by organ system, AT population, Restarter.18Table C-3.5.5Incidence rate of malignant neoplasms by organ system, AT population, Diagnosis confirmed by surgery.18Table C-3.5.6Incidence rate of malignant neoplasms by organ system, AT population, Diagnosis based on clinical symptoms18Table C-3.5.7Incidence rate of malignant neoplasms by organ system, AT population, Germany.18Table C-3.5.8Incidence rate of malignant neoplasms by organ system, AT population, Poland18Table C-3.5.9Incidence rate of malignant neoplasms by organ system, AT population, Hungary.18Table C-3.5.10Incidence rate of malignant neoplasms by organ system, AT population, Switzerland.18Table C-3.5.11Incidence rate of malignant neoplasms by organ system, AT population, Russia18Table C-3.5.12Incidence rate of malignant neoplasms by organ system, AT population, Ukraine.18Section C-3.6Incidence proportion of malformations.18Table C-3.6.1Incidence proportion of malformations, AT population, Complete cohort18Table C-3.6.2Incidence proportion of malformations, AT population, Switcher18Table C-3.6.3Incidence proportion of malformations, AT population, Switcher18Table C-3.6.5Incidence proportion of malformations, AT population, Diagnosis based on clinical symptoms18Table C-3.6.6Incidence proportion of malformations, AT population, Diagnosis based on clinical symptoms18Table C-3.6.7Incidence proportion of malformations, AT population, Poland18 <td>Table C-3.5.2</td> <td>Incidence rate of malignant neoplasms by organ system, AT population, Starter</td> <td> 182</td> | Table C-3.5.2 | Incidence rate of malignant neoplasms by organ system, AT population, Starter | 182 |
| Table C-3.5.5Incidence rate of malignant neoplasms by organ system, AT population, Diagnosis confirmed by surgery18Table C-3.5.6Incidence rate of malignant neoplasms by organ system, AT population, Diagnosis based on clinical symptoms18Table C-3.5.7Incidence rate of malignant neoplasms by organ system, AT population, Germany18Table C-3.5.8Incidence rate of malignant neoplasms by organ system, AT population, Poland18Table C-3.5.9Incidence rate of malignant neoplasms by organ system, AT population, Hungary18Table C-3.5.10Incidence rate of malignant neoplasms by organ system, AT population, Switzerland18Table C-3.5.11Incidence rate of malignant neoplasms by organ system, AT population, Russia18Table C-3.5.12Incidence rate of malignant neoplasms by organ system, AT population, Ukraine18Table C-3.6.1Incidence proportion of malformations18Table C-3.6.2Incidence proportion of malformations, AT population, Complete cohort18Table C-3.6.3Incidence proportion of malformations, AT population, Switcher18Table C-3.6.4Incidence proportion of malformations, AT population, Switcher18Table C-3.6.5Incidence proportion of malformations, AT population, Diagnosis confirmed by surgery18Table C-3.6.6Incidence proportion of malformations, AT population, Diagnosis based on clinical symptoms18Table C-3.6.8Incidence proportion of malformations, AT population, Poland18Table C-3.6.9Incidence proportion of malformations, AT population, Poland18Table C-3.6.10 <td>Table C-3.5.3</td> <td></td> <td></td> | Table C-3.5.3 | | |
| Table C-3.5.6 Incidence rate of malignant neoplasms by organ system, AT population, Diagnosis based on clinical symptoms | Table C-3.5.4 | Incidence rate of malignant neoplasms by organ system, AT population, Restarter | 182 |
| Table C-3.5.7Incidence rate of malignant neoplasms by organ system, AT population, Germany.18Table C-3.5.8Incidence rate of malignant neoplasms by organ system, AT population, Poland.18Table C-3.5.9Incidence rate of malignant neoplasms by organ system, AT population, Hungary.18Table C-3.5.10Incidence rate of malignant neoplasms by organ system, AT population, Switzerland.18Table C-3.5.11Incidence rate of malignant neoplasms by organ system, AT population, Russia.18Table C-3.5.12Incidence rate of malignant neoplasms by organ system, AT population, Ukraine.18Section C-3.6Incidence proportion of malformations.18Table C-3.6.1Incidence proportion of malformations, AT population, Complete cohort.18Table C-3.6.2Incidence proportion of malformations, AT population, Starter.18Table C-3.6.3Incidence proportion of malformations, AT population, Switcher.18Table C-3.6.4Incidence proportion of malformations, AT population, Restarter.18Table C-3.6.5Incidence proportion of malformations, AT population, Diagnosis confirmed by surgery.18Table C-3.6.7Incidence proportion of malformations, AT population, Diagnosis based on clinical symptoms18Table C-3.6.8Incidence proportion of malformations, AT population, Poland18Table C-3.6.9Incidence proportion of malformations, AT population, Hungary18Table C-3.6.10Incidence proportion of malformations, AT population, Switzerland18Table C-3.6.11Incidence proportion of malformations, AT population, Switz | Table C-3.5.5 | Incidence rate of malignant neoplasms by organ system, AT population, Diagnosis confirmed by surgery | 182 |
| Table C-3.5.8Incidence rate of malignant neoplasms by organ system, AT population, Poland18Table C-3.5.9Incidence rate of malignant neoplasms by organ system, AT population, Hungary18Table C-3.5.10Incidence rate of malignant neoplasms by organ system, AT population, Switzerland18Table C-3.5.11Incidence rate of malignant neoplasms by organ system, AT population, Russia18Table C-3.5.12Incidence rate of malignant neoplasms by organ system, AT population, Ukraine18Section C-3.6Incidence proportion of malformations18Table C-3.6.1Incidence proportion of malformations, AT population, Complete cohort18Table C-3.6.2Incidence proportion of malformations, AT population, Switcher18Table C-3.6.3Incidence proportion of malformations, AT population, Switcher18Table C-3.6.4Incidence proportion of malformations, AT population, Restarter18Table C-3.6.5Incidence proportion of malformations, AT population, Diagnosis confirmed by surgery18Table C-3.6.6Incidence proportion of malformations, AT population, Diagnosis based on clinical symptoms18Table C-3.6.7Incidence proportion of malformations, AT population, Germany18Table C-3.6.8Incidence proportion of malformations, AT population, Poland18Table C-3.6.9Incidence proportion of malformations, AT population, Hungary18Table C-3.6.10Incidence proportion of malformations, AT population, Switzerland18Table C-3.6.11Incidence proportion of malformations, AT population, Switzerland18 | Table C-3.5.6 | Incidence rate of malignant neoplasms by organ system, AT population, Diagnosis based on clinical symptoms | 182 |
| Table C-3.5.9Incidence rate of malignant neoplasms by organ system, AT population, Hungary18Table C-3.5.10Incidence rate of malignant neoplasms by organ system, AT population, Switzerland18Table C-3.5.11Incidence rate of malignant neoplasms by organ system, AT population, Russia18Table C-3.5.12Incidence rate of malignant neoplasms by organ system, AT population, Ukraine18Section C-3.6Incidence proportion of malformations18Table C-3.6.1Incidence proportion of malformations, AT population, Complete cohort18Table C-3.6.2Incidence proportion of malformations, AT population, Starter18Table C-3.6.3Incidence proportion of malformations, AT population, Switcher18Table C-3.6.4Incidence proportion of malformations, AT population, Switcher18Table C-3.6.5Incidence proportion of malformations, AT population, Diagnosis confirmed by surgery18Table C-3.6.6Incidence proportion of malformations, AT population, Diagnosis based on clinical symptoms18Table C-3.6.7Incidence proportion of malformations, AT population, Germany18Table C-3.6.8Incidence proportion of malformations, AT population, Poland18Table C-3.6.9Incidence proportion of malformations, AT population, Hungary18Table C-3.6.10Incidence proportion of malformations, AT population, Switzerland18Table C-3.6.11Incidence proportion of malformations, AT population, Switzerland18 | Table C-3.5.7 | Incidence rate of malignant neoplasms by organ system, AT population, Germany | 182 |
| Table C-3.5.10Incidence rate of malignant neoplasms by organ system, AT population, Switzerland.18Table C-3.5.11Incidence rate of malignant neoplasms by organ system, AT population, Russia18Table C-3.5.12Incidence rate of malignant neoplasms by organ system, AT population, Ukraine18Section C-3.6Incidence proportion of malformations18Table C-3.6.1Incidence proportion of malformations, AT population, Complete cohort18Table C-3.6.2Incidence proportion of malformations, AT population, Starter18Table C-3.6.3Incidence proportion of malformations, AT population, Switcher18Table C-3.6.4Incidence proportion of malformations, AT population, Restarter18Table C-3.6.5Incidence proportion of malformations, AT population, Diagnosis confirmed by surgery18Table C-3.6.6Incidence proportion of malformations, AT population, Diagnosis based on clinical symptoms18Table C-3.6.7Incidence proportion of malformations, AT population, Germany18Table C-3.6.8Incidence proportion of malformations, AT population, Poland18Table C-3.6.9Incidence proportion of malformations, AT population, Hungary18Table C-3.6.10Incidence proportion of malformations, AT population, Switzerland18Table C-3.6.11Incidence proportion of malformations, AT population, Russia18 | Table C-3.5.8 | Incidence rate of malignant neoplasms by organ system, AT population, Poland | 182 |
| Table C-3.5.11Incidence rate of malignant neoplasms by organ system, AT population, Russia18Table C-3.5.12Incidence rate of malignant neoplasms by organ system, AT population, Ukraine18Section C-3.6Incidence proportion of malformations18Table C-3.6.1Incidence proportion of malformations, AT population, Complete cohort18Table C-3.6.2Incidence proportion of malformations, AT population, Starter18Table C-3.6.3Incidence proportion of malformations, AT population, Switcher18Table C-3.6.4Incidence proportion of malformations, AT population, Restarter18Table C-3.6.5Incidence proportion of malformations, AT population, Diagnosis confirmed by surgery18Table C-3.6.6Incidence proportion of malformations, AT population, Diagnosis based on clinical symptoms18Table C-3.6.7Incidence proportion of malformations, AT population, Germany18Table C-3.6.8Incidence proportion of malformations, AT population, Poland18Table C-3.6.9Incidence proportion of malformations, AT population, Hungary18Table C-3.6.10Incidence proportion of malformations, AT population, Switzerland18Table C-3.6.11Incidence proportion of malformations, AT population, Russia18 | Table C-3.5.9 | Incidence rate of malignant neoplasms by organ system, AT population, Hungary | 182 |
| Table C-3.5.12Incidence rate of malignant neoplasms by organ system, AT population, Ukraine18Section C-3.6Incidence proportion of malformations18Table C-3.6.1Incidence proportion of malformations, AT population, Complete cohort18Table C-3.6.2Incidence proportion of malformations, AT population, Starter18Table C-3.6.3Incidence proportion of malformations, AT population, Switcher18Table C-3.6.4Incidence proportion of malformations, AT population, Restarter18Table C-3.6.5Incidence proportion of malformations, AT population, Diagnosis confirmed by surgery18Table C-3.6.6Incidence proportion of malformations, AT population, Diagnosis based on clinical symptoms18Table C-3.6.7Incidence proportion of malformations, AT population, Germany18Table C-3.6.8Incidence proportion of malformations, AT population, Poland18Table C-3.6.9Incidence proportion of malformations, AT population, Hungary18Table C-3.6.10Incidence proportion of malformations, AT population, Switzerland18Table C-3.6.11Incidence proportion of malformations, AT population, Russia18 | Table C-3.5.10 | Incidence rate of malignant neoplasms by organ system, AT population, Switzerland | 182 |
| Incidence proportion of malformations | Table C-3.5.11 | Incidence rate of malignant neoplasms by organ system, AT population, Russia | 182 |
| Table C-3.6.1Incidence proportion of malformations, AT population, Complete cohort18Table C-3.6.2Incidence proportion of malformations, AT population, Starter18Table C-3.6.3Incidence proportion of malformations, AT population, Switcher18Table C-3.6.4Incidence proportion of malformations, AT population, Restarter18Table C-3.6.5Incidence proportion of malformations, AT population, Diagnosis confirmed by surgery18Table C-3.6.6Incidence proportion of malformations, AT population, Diagnosis based on clinical symptoms18Table C-3.6.7Incidence proportion of malformations, AT population, Germany18Table C-3.6.8Incidence proportion of malformations, AT population, Poland18Table C-3.6.9Incidence proportion of malformations, AT population, Hungary18Table C-3.6.10Incidence proportion of malformations, AT population, Switzerland18Table C-3.6.11Incidence proportion of malformations, AT population, Russia18 | Table C-3.5.12 | Incidence rate of malignant neoplasms by organ system, AT population, Ukraine | 182 |
| Table C-3.6.2Incidence proportion of malformations, AT population, Starter18Table C-3.6.3Incidence proportion of malformations, AT population, Switcher18Table C-3.6.4Incidence proportion of malformations, AT population, Restarter18Table C-3.6.5Incidence proportion of malformations, AT population, Diagnosis confirmed by surgery18Table C-3.6.6Incidence proportion of malformations, AT population, Diagnosis based on clinical symptoms18Table C-3.6.7Incidence proportion of malformations, AT population, Germany18Table C-3.6.8Incidence proportion of malformations, AT population, Poland18Table C-3.6.9Incidence proportion of malformations, AT population, Hungary18Table C-3.6.10Incidence proportion of malformations, AT population, Switzerland18Table C-3.6.11Incidence proportion of malformations, AT population, Russia18 | Section C-3.6 | Incidence proportion of malformations | 183 |
| Table C-3.6.3Incidence proportion of malformations, AT population, Switcher18Table C-3.6.4Incidence proportion of malformations, AT population, Restarter18Table C-3.6.5Incidence proportion of malformations, AT population, Diagnosis confirmed by surgery18Table C-3.6.6Incidence proportion of malformations, AT population, Diagnosis based on clinical symptoms18Table C-3.6.7Incidence proportion of malformations, AT population, Germany18Table C-3.6.8Incidence proportion of malformations, AT population, Poland18Table C-3.6.9Incidence proportion of malformations, AT population, Hungary18Table C-3.6.10Incidence proportion of malformations, AT population, Switzerland18Table C-3.6.11Incidence proportion of malformations, AT population, Russia18 | Table C-3.6.1 | Incidence proportion of malformations, AT population, Complete cohort | 183 |
| Table C-3.6.4Incidence proportion of malformations, AT population, Restarter18-Table C-3.6.5Incidence proportion of malformations, AT population, Diagnosis confirmed by surgery18-Table C-3.6.6Incidence proportion of malformations, AT population, Diagnosis based on clinical symptoms18-Table C-3.6.7Incidence proportion of malformations, AT population, Germany18-Table C-3.6.8Incidence proportion of malformations, AT population, Poland18-Table C-3.6.9Incidence proportion of malformations, AT population, Hungary18-Table C-3.6.10Incidence proportion of malformations, AT population, Switzerland18-Table C-3.6.11Incidence proportion of malformations, AT population, Russia18- | Table C-3.6.2 | Incidence proportion of malformations, AT population, Starter | 184 |
| Incidence proportion of malformations, AT population, Diagnosis confirmed by surgery | Table C-3.6.3 | Incidence proportion of malformations, AT population, Switcher | 184 |
| Incidence proportion of malformations, AT population, Diagnosis based on clinical symptoms | Table C-3.6.4 | Incidence proportion of malformations, AT population, Restarter | 184 |
| Table C-3.6.7 Incidence proportion of malformations, AT population, Germany | Table C-3.6.5 | Incidence proportion of malformations, AT population, Diagnosis confirmed by surgery | 184 |
| Table C-3.6.8 Incidence proportion of malformations, AT population, Poland | Table C-3.6.6 | Incidence proportion of malformations, AT population, Diagnosis based on clinical symptoms | 184 |
| Table C-3.6.9 Incidence proportion of malformations, AT population, Hungary | Table C-3.6.7 | Incidence proportion of malformations, AT population, Germany | 184 |
| Table C-3.6.10 Incidence proportion of malformations, AT population, Switzerland | Table C-3.6.8 | Incidence proportion of malformations, AT population, Poland | 184 |
| Table C-3.6.11 Incidence proportion of malformations, AT population, Russia | Table C-3.6.9 | Incidence proportion of malformations, AT population, Hungary | 184 |
| | Table C-3.6.10 | Incidence proportion of malformations, AT population, Switzerland | |
| Table C-3.6.12 Incidence proportion of malformations, AT population, Ukraine | Table C-3.6.11 | Incidence proportion of malformations, AT population, Russia | |
| | Table C-3.6.12 | Incidence proportion of malformations, AT population, Ukraine | 184 |



| Section C-4 | Other outcomes of interest | 185 |
|---|---|---|
| Section C-4.1 | Incidence rate of surgery / laparoscopy because of endometriosis | 185 |
| Section C-4.1 | Incidence rate of surgery / laparoscopy because of endometriosis, ITT population, Complete cohort | 185 |
| Table C-4.1.2 | Incidence rate of surgery / laparoscopy because of endometriosis, AT population, Starter | 187 |
| Table C-4.1.3 | Incidence rate of surgery / laparoscopy because of endometriosis, AT population, Switcher | 187 |
| Table C-4.1.4 | Incidence rate of surgery / laparoscopy because of endometriosis, AT population, Restarter | 187 |
| Table C-4.1.5 | Incidence rate of surgery / laparoscopy because of endometriosis, AT population, Diagnosis confirmed by surgery | 187 |
| Table C-4.1.6 | Incidence rate of surgery / laparoscopy because of endometriosis, AT population, Diagnosis based on clinical symptoms | 187 |
| Table C-4.1.7 | Incidence rate of surgery / laparoscopy because of endometriosis, AT population, Germany | 187 |
| Table C-4.1.8 | Incidence rate of surgery / laparoscopy because of endometriosis, AT population, Poland | 187 |
| Table C-4.1.9 | Incidence rate of surgery / laparoscopy because of endometriosis, AT population, Hungary | 187 |
| Table C-4.1.1 | O Incidence rate of surgery / laparoscopy because of endometriosis, AT population, Switzerland | 187 |
| Table C-4.1.1 | 1 Incidence rate of surgery / laparoscopy because of endometriosis, AT population, Russia | 187 |
| Table C-4.1.1 | 2 Incidence rate of surgery / laparoscopy because of endometriosis, AT population, Ukraine | 187 |
| Section C-4.2 | Incidence rate of self-reported anemia | 188 |
| Table C-4.2.1 | Incidence rate of self-reported anemia, AT population, Complete cohort | 188 |
| Table C-4.2.2 | Incidence rate of self-reported anemia, AT population, Starter | 189 |
| Table C-4.2.3 | Incidence rate of self-reported anemia, AT population, Switcher | 189 |
| Table C-4.2.4 | Incidence rate of self-reported anemia, AT population, Restarter | 189 |
| Table C-4.2.5 | Incidence rate of self-reported anemia, AT population, Diagnosis confirmed by surgery | 189 |
| Table C-4.2.6 | Incidence rate of self-reported anemia, AT population, Diagnosis based on clinical symptoms | 189 |
| Table C-4.2.7 | Incidence rate of self-reported anemia, AT population, Germany | 189 |
| Table C-4.2.8 | Incidence rate of self-reported anemia, AT population, Poland | 189 |
| Table C-4.2.9 | Incidence rate of self-reported anemia, AT population, Hungary | 189 |
| Table C-4.2.1 | 0 Incidence rate of self-reported anemia, AT population, Switzerland | 189 |
| Table C-4.2.1 | 1 Incidence rate of self-reported anemia, AT population, Russia | 189 |
| Table C-4.2.1 | 2 Incidence rate of self-reported anemia, AT population, Ukraine | 189 |
| Section C-4.3 | Incidence rate of self-reported depression | 190 |
| Table C-4.3.1 | Incidence rate of self-reported depression, AT population, Compete cohort | 190 |
| Table C-4.3.2 | Incidence rate of self-reported depression, AT population, Starter | 191 |



| Table C-4.3.3 | Incidence rate of self-reported depression, AT population, Switcher | 191 |
|---|---|---|
| Table C-4.3.4 | Incidence rate of self-reported depression, AT population, Restarter | 191 |
| Table C-4.3.5 | Incidence rate of self-reported depression, AT population, Diagnosis confirmed by surgery | |
| Table C-4.3.6 | Incidence rate of self-reported depression, AT population, Diagnosis based on clinical symptoms | 191 |
| Table C-4.3.7 | Incidence rate of self-reported depression, AT population, Germany | 191 |
| Table C-4.3.8 | Incidence rate of self-reported depression, AT population, Poland | 191 |
| Table C-4.3.9 | Incidence rate of self-reported depression, AT population, Hungary | 191 |
| Table C-4.3.10 | Incidence rate of self-reported depression, AT population, Switzerland | 191 |
| Table C-4.3.11 | Incidence rate of self-reported depression, AT population, Russia | 191 |
| Table C-4.3.12 | Incidence rate of self-reported depression, AT population, Ukraine | 191 |
| Section D <b>Comparisons</b> a | and Inferential Statistics of Primary Outcomes | 192 |
| Section D-1 New anem | nia and reoccurrence of anemia | 192 |
| Table D-1.1.1 | Incidence rate ratio of new anemia and reoccurrence of anemia between EMT user cohorts, AT population | 192 |
| Table D-1.1.2 | Risk of new anemia and reoccurrence of anemia obtained from Cox model (HR), AT population | 193 |
| Section D-2 New depre | ession or deterioration of existing depression | 194 |
| Section D-2.1 | Incidence rate ratio of new depression or deterioration of existing depression between EMT user cohorts, AT population | 194 |
| Section D-2.2 | Risk of new depression or deterioration of existing depression obtained from the Cox model (HR), AT population | 194 |
| Section D-3 Treatment | failure | 194 |
| Section D-3.1 | Incidence rate ratio of treatment failure between EMT user cohorts, AT population | 194 |
| Section D-3.2 | Risk of treatment failure obtained from the Cox model (HR), AT population | 194 |



Supporting document SOP BMT 01.09 – Doc 5002.02 – Effective date 21.03.2017

#### Section A Population Distribution

Section A-1 Eligibility status

Section A-1.1 Eligibility Status (all recruited women)

Table A-1.1.1 Eligibility Status (all recruited women)

| | Total |
|------------------------------------------|-------------|
| Number (%) of recruited women | xx ( 100%) |
| Thereof | |
| Enrolled women | xx ( xx.x%) |
| Not enrolled women | xx ( xx.x%) |
| Number (%) of women not enrolled Reason | xx ( 100%) |
| Duplicate | xx ( xx.x%) |
| No complete informed consent available | xx ( xx.x%) |
| Language problems | xx ( xx.x%) |
| < <category>&gt;</category> | xx ( xx.x%) |

Supporting document SOP BMT 01.09 – Doc 5002.02 – Effective date 21.03.2017

#### Section A-1.2 Study status of women at follow-up

Table A-1.2.1 Study status of women at follow-up, ITT population, Complete cohort

| | DNG | OAED | | | | NAED | Allocation<br>unknown | Total | |
|---|---|---|---|---|---|---|---|---|---|
| | | GnRH-a | Danazol | All OAED | CC | Other progestin | All NAED | | |
| Number (%) of women | xx (100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) |
| At study entry Thereof | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Drop out | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Loss to follow-up | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| At < 6 months Thereof Drop out Loss to follow-up | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| <br>At 72 months or later<br> | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

Note: \*Presented at the end of follow-up only.

Table A-1.2.2 Study status of women at follow-up, AT population, Complete cohort



Supporting document SOP BMT 01.09 – Doc 5002.02 – Effective date 21.03.2017

#### Section A-2 Distribution of women

#### Section A-2.1 Regional distribution

Table A-2.1.1 Study status of women at follow-up, ITT population, Complete cohort

| | DNG | | OAED | | | NAED | Allocation<br>unknown | Total | |
|---|---|---|---|---|---|---|---|---|---|
| | | GnRH-a | Danazol | All OAED | СС | Other progestin | All NAED | | |
| Number (%) of women | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( 100%) |
| Germany | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( 100%) |
| Poland | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( 100%) |
| Russia | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( 100%) |
| Hungary | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( 100%) |
| Switzerland | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( 100%) |
| Ukraine | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( 100%) |



Supporting document SOP BMT 01.09 – Doc 5002.02 – Effective date 21.03.2017

#### Section A-2.2 EMT user type at study entry

Table A-2.2.1 EMT user type at study entry, ITT population, Complete cohort

| | DNG | | OAED | | | NAED | Allocation<br>unknown | Total | |
|---|---|---|---|---|---|---|---|---|---|
| | | GnRH-a | Danazol | All OAED | CC | Other progestin | All NAED | | |
| Number (%) of women | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) |
| Starters | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Switchers | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Restarters | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

Date of analysis:

Table A-2.2.2 EMT user type at study entry, ITT population, Germany

Table A-2.2.3 EMT user type at study entry, ITT population, Poland

Table A-2.2.4 EMT user type at study entry, ITT population, Hungary

Table A-2.2.5 EMT user type at study entry, ITT population, Switzerland

Table A-2.2.6 EMT user type at study entry, ITT population, Russia

Table A-2.2.7 EMT user type at study entry, ITT population, Ukraine



Supporting document SOP BMT 01.09 - Doc 5002.02 - Effective date 21.03.2017

#### Section A-2.3 Classification of endometriosis diagnosis at study entry

Table A-2.3.1 Classification of endometriosis diagnosis at study entry, ITT population, Complete cohort

| | DNG | OAED | | | NAED | Allocation<br>unknown | Total | | |
|---|---|---|---|---|---|---|---|---|---|
| | | GnRH-a | Danazol | All OAED | CC | Other progestin | All NAED | | |
| Number (%) of women | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) |
| Surgically confirmed diagnosis | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Clinically confirmed diagnosis | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

Date of analysis:

| Table A-2.3.2 | Classification of endometriosis | s diagnosis at study entry, | ITT population, Starter |
|---|---|---|---|
|---|---|---|---|

Table A-2.3.3 Classification of endometriosis diagnosis at study entry, ITT population, ITT, Switcher

Table A-2.3.4 Classification of endometriosis diagnosis at study entry, ITT population, Restarter

Table A-2.3.5 Classification of endometriosis diagnosis at study entry, ITT population, Germany

Table A-2.3.6 Classification of endometriosis diagnosis at study entry, ITT population, Poland

Table A-2.3.7 Classification of endometriosis diagnosis at study entry, ITT population, Hungary

Table A-2.3.8 Classification of endometriosis diagnosis at study entry, ITT population, Switzerland

Table A-2.3.9 Classification of endometriosis diagnosis at study entry, ITT population, Russia

Table A-2.3.10 Classification of endometriosis diagnosis at study entry, ITT population, Ukraine



Supporting document SOP BMT 01.09 - Doc 5002.02 - Effective date 21.03.2017

#### Section B **Population Characteristics**

Section B-1 Age and body measurements

Section B-1.1 Age at study entry

Table B-1.1.1 Age (years) at study entry, ITT population, Complete cohort

| | DNG | | OAED | | | NAED | | Allocation unknown | Total |
|---|---|---|---|---|---|---|---|---|---|
| | | GnRH-a | Danazol | All OAED | CC | Other progestin | All NAED | | |
| Number (%) of women | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) |
| Age (years) | | | | | | | | | |
| n | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Missing | 0 ( 0.00%) | 0 ( 0.00%) | 0 ( 0.00%) | 0 ( 0.00%) | 0 ( 0.00%) | 0 ( 0.00%) | 0 ( 0.00%) | 0 ( 0.00%) | 0 ( 0.00%) |
| Mean | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | XX.X |
| SD | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx | XX.XX | XX.XX | xx.xx |
| Min | XX | XX | xx | XX | xx | XX | xx | XX | xx |
| Q1 | XX.X | XX.X | xx.x | XX.X | xx.x | XX.X | xx.x | XX.X | xx.x |
| Median | XX.X | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | XX.X | xx.x |
| Q3 | XX.X | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | XX.X | xx.x |
| Max | xx | XX | XX | XX | XX | XX | XX | XX | XX |
| Adolescents <18 years | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Age category | | | | | | | | | |
| <20 years | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 20 to <30 years | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 30 to <40 years | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| ≥40 years | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Missing | 0 ( 0.00%) | 0 ( 0.00%) | 0 ( 0.00%) | 0 ( 0.00%) | 0 ( 0.00%) | 0 ( 0.00%) | 0 ( 0.00%) | 0 ( 0.00%) | 0 ( 0.00%) |



| Table B-1.1.2 | Age (years) at study entry, AT population, Complete cohort |
|---|---|
| Table B-1.1.3 | Age (years) at study entry, AT population, Starter |
| Table B-1.1.4 | Age (years) at study entry, AT population, Switcher |
| Table B-1.1.5 | Age (years) at study entry, AT population, Restarter |
| Table B-1.1.6 | Age (years) at study entry, AT population, Diagnosis confirmed by surgery |
| Table B-1.1.7 | Age (years) at study entry, AT population, Diagnosis based on clinical symptoms |
| Table B-1.1.8 | Age (years) at study entry, AT population, Germany |
| Table B-1.1.9 | Age (years) at study entry, AT population, Poland |
| Table B-1.1.10 | Age (years) at study entry, AT population, Hungary |
| Table B-1.1.11 | Age (years) at study entry, AT population, Switzerland |
| Table B-1.1.12 | Age (years) at study entry, AT population, Russia |
| Table B-1.1.13 | Age (years) at study entry, AT population, Ukraine |



Supporting document SOP BMT 01.09 – Doc 5002.02 – Effective date 21.03.2017

Section B-1.2 Height (cm) and Weight (kg) at study entry

Table B-1.2.1 Height (cm) and Weight (kg) at study entry, ITT population, Complete cohort

| | DNG | OAED | | | NAED | | | Allocation unknown | Total |
|---|---|---|---|---|---|---|---|---|---|
| | | GnRH-a | Danazol | All OAED | CC | Other progestin | All NAED | | |
| Number (%) of women | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) |
| Height (cm) | | | | | | | | | |
| n | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Missing | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Mean | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |
| SD | xx.xx | xx.xx | XX.XX | XX.XX | XX.XX | XX.XX | xx.xx | XX.XX | XX.XX |
| Min | XX | XX | xx | XX | xx | xx | xx | XX | XX |
| Q1 | XX.X | XX.X | xx.x | xx.x | XX.X | xx.x | xx.x | XX.X | XX.X |
| Median | XX.X | XX.X | xx.x | xx.x | XX.X | xx.x | xx.x | XX.X | XX.X |
| Q3 | XX.X | XX.X | xx.x | XX.X | xx.x | xx.x | xx.x | XX.X | xx.x |
| Max | XX | XX | XX | XX | XX | XX | XX | xx | XX |
| Weight (kg) | | | | | | | | | |
| n | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Missing | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Mean | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |
| SD | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx |
| Min | XX | XX | XX | xx | XX | xx | xx | XX | xx |
| Q1 | XX.X | xx.x | xx.x | xx.x | xx.x | XX.X | XX.X | XX.X | xx.x |
| Median | XX.X | xx.x | xx.x | xx.x | xx.x | XX.X | XX.X | XX.X | xx.x |
| Q3 | XX.X | xx.x | xx.x | xx.x | xx.x | XX.X | XX.X | XX.X | xx.x |
| Max | XX | XX | xx | xx | xx | xx | xx | XX | xx |


| Table B-1.2.2 | Height (cm) and Weight (kg) at study entry, AT population, Complete cohort |
|---|---|
| Table B-1.2.3 | Height (cm) and Weight (kg) at study entry, AT population, Starter |
| Table B-1.2.4 | Height (cm) and Weight (kg) at study entry, AT population, Switcher |
| Table B-1.2.5 | Height (cm) and Weight (kg) at study entry, AT population, Restarter |
| Table B-1.2.6 | Height (cm) and Weight (kg) at study entry, AT population, Diagnosis confirmed by surgery |
| Table B-1.2.7 | Height (cm) and Weight (kg) at study entry, AT population, Diagnosis based on clinical symptoms |
| Table B-1.2.8 | Height (cm) and Weight (kg) at study entry, AT population, Germany |
| Table B-1.2.9 | Height (cm) and Weight (kg) at study entry, AT population, Poland |
| Table B-1.2.10 | Height (cm) and Weight (kg) at study entry, AT population, Hungary |
| Table B-1.2.11 | Height (cm) and Weight (kg) at study entry, AT population, Switzerland |
| Table B-1.2.12 | Height (cm) and Weight (kg) at study entry, AT population, Russia |
| Table B-1.2.13 | Height (cm) and Weight (kg) at study entry, AT population, Ukraine |



Supporting document SOP BMT 01.09 – Doc 5002.02 – Effective date 21.03.2017

Section B-1.3 Body Mass Index (BMI) at study entry

Table B-1.3.1 Body Mass Index (BMI) at study entry, ITT population, Complete Cohort

| | DNG | | | | | NAED | | Allocation unknown | Total |
|---|---|---|---|---|---|---|---|---|---|
| | | GnRH-a | Danazol | All OAED | СС | Other progestin | All NAED | •• | |
| Number (%) of women | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100% |
| BMI (kg/m²) | | | | | | | | | |
| n | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x% |
| Missing | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x% |
| Mean | XX.X | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | XX.) |
| SD | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx | XX.XX | xx.xx | xx.xx |
| Min | xx | xx | xx | xx | xx | XX | xx | XX | x |
| Q1 | xx.x | xx.x | xx.x | XX.X | xx.x | XX.X | XX.X | XX.X | XX.) |
| Median | XX.X | XX.X | xx.x | XX.X | XX.X | XX.X | xx.x | XX.X | XX.) |
| Q3 | XX.X | xx.x | xx.x | XX.X | xx.x | XX.X | xx.x | XX.X | XX.) |
| Max | XX | XX | XX | XX | xx | XX | XX | xx | XX |
| BMI category | | | | | | | | | |
| <20 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x% |
| 20 to <25 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x% |
| 25 to <30 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x% |
| 30 to <35 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x% |
| ≥35 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x% |
| Missing | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x% |



| Table B-1.3.2 | Body Mass Index (BMI) at study entry, AT population, Complete cohort |
|---|---|
| Table B-1.3.3 | Body Mass Index (BMI) at study entry, AT population, Starter |
| Table B-1.3.4 | Body Mass Index (BMI) at study entry, AT population, Switcher |
| Table B-1.3.5 | Body Mass Index (BMI) at study entry, AT population, Restarter |
| Table B-1.3.6 | Body Mass Index (BMI) at study entry, AT population, Diagnosis confirmed by surgery |
| Table B-1.3.7 | Body Mass Index (BMI) at study entry, AT population, Diagnosis based on clinical symptoms |
| Table B-1.3.8 | Body Mass Index (BMI) at study entry, AT population, Germany |
| Table B-1.3.9 | Body Mass Index (BMI) at study entry, AT population, Poland |
| Table B-1.3.10 | Body Mass Index (BMI) at study entry, AT population, Hungary |
| Table B-1.3.11 | Body Mass Index (BMI) at study entry, AT population, Switzerland |
| Table B-1.3.12 | Body Mass Index (BMI) at study entry, AT population, Russia |
| Table B-1.3.13 | Body Mass Index (BMI) at study entry, AT population, Ukraine |



Supporting document SOP BMT 01.09 – Doc 5002.02 – Effective date 21.03.2017

#### Section B-2 Socio-economic characteristics and lifestyle factors

#### Section B-2.1 Status of cigarette smoking at study entry

Table B-2.1.1 Status of cigarette smoking at study entry, ITT population, Complete cohort

| | DNG | OAED | | | | NAED | Allocation<br>unknown | Total | |
|---|---|---|---|---|---|---|---|---|---|
| | | GnRH-a | Danazol | All OAED | CC | Other progestin | All NAED | | |
| Number (%) of women | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) |
| Status of smoking | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Never | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Current | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Thereof | | | | | | | | | |
| Heavy smoker | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| (>15 cigarettes/day) | | | | | | | | | |
| Ex-Smoker | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Missing | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |



| Table B-2.1.2 | Status of cigarette smoking at study entry, AT population, Complete cohort |
|---|---|
| Table B-2.1.3 | Status of cigarette smoking at study entry, AT population, Starter |
| Table B-2.1.4 | Status of cigarette smoking at study entry, AT population, Switcher |
| Table B-2.1.5 | Status of cigarette smoking at study entry, AT population, Restarter |
| Table B-2.1.6 | Status of cigarette smoking at study entry, AT population, Diagnosis confirmed by surgery |
| Table B-2.1.7 | Status of cigarette smoking at study entry, AT population, Diagnosis based on clinical symptoms |
| Table B-2.1.8 | Status of cigarette smoking at study entry, AT population, Germany |
| Table B-2.1.9 | Status of cigarette smoking at study entry, AT population, Poland |
| Table B-2.1.10 | Status of cigarette smoking at study entry, AT population, Hungary |
| Table B-2.1.11 | Status of cigarette smoking at study entry, AT population, Switzerland |
| Table B-2.1.12 | Status of cigarette smoking at study entry, AT population, Russia |
| Table B-2.1.13 | Status of cigarette smoking at study entry, AT population, Ukraine |



Supporting document SOP BMT 01.09 – Doc 5002.02 – Effective date 21.03.2017

#### Section B-2.2 Educational level at study entry

Table B-2.2.1 Educational level at study entry, ITT population, Complete cohort

| | DNG | | OAED | | | NAED | Allocation<br>unknown | Total | |
|---|---|---|---|---|---|---|---|---|---|
| | | GnRH-a | Danazol | All OAED | CC C | Other progestin | All NAED | | _ |
| Number (%) of women | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) |
| Education level | | | | | | | | | |
| Less than university entrance level | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| University entrance level | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Higher than university entrance level | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Missing | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |



| Table B-2.2.2 | Educational level at study entry, AT population, Complete cohort |
|---|---|
| Table B-2.2.3 | Educational level at study entry, AT population, Starter |
| Table B-2.2.4 | Educational level at study entry, AT population, Switcher |
| Table B-2.2.5 | Educational level at study entry, AT population, Restarter |
| Table B-2.2.6 | Educational level at study entry, AT population, Diagnosis confirmed by surgery |
| Table B-2.2.7 | Educational level at study entry, AT population, Diagnosis based on clinical symptoms |
| Table B-2.2.8 | Educational level at study entry, AT population, Germany |
| Table B-2.2.9 | Educational level at study entry, AT population, Poland |
| Table B-2.2.10 | Educational level at study entry, AT population, Hungary |
| Table B-2.2.11 | Educational level at study entry, AT population, Switzerland |
| Table B-2.2.12 | Educational level at study entry, AT population, Russia |
| Table B-2.2.13 | Educational level at study entry, AT population, Ukraine |



Supporting document SOP BMT 01.09 – Doc 5002.02 – Effective date 21.03.2017

#### Section B-3 Gynecological history

Section B-3.1 Age (years) at menarche at study entry

Table B-3.1.1 Age (years) at menarche at study entry, ITT population, Complete cohort

| | DNG | NG OAED | | | | NAED | Allocation unknown | Total | |
|---|---|---|---|---|---|---|---|---|---|
| | | GnRH-a | Danazol | All OAED | СС | Other progestin | All NAED | | |
| Number (%) of women | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100% |
| Age at menarche (years) | | | | | | | | | |
| n | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x% |
| Missing | 0 ( 0.00%) | 0 ( 0.00%) | 0 ( 0.00%) | 0 ( 0.00%) | 0 ( 0.00%) | 0 ( 0.00%) | 0 ( 0.00%) | 0 ( 0.00%) | 0 ( 0.00% |
| Mean | XX.X | xx.x | xx.x | xx.x | xx.x | XX.X | XX.X | xx.x | xx. |
| SD | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx | XX.XX | xx.x |
| Min | xx | xx | xx | xx | xx | xx | xx | XX | x |
| Q1 | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | XX.X | XX. |
| Median | xx.x | XX.X | xx.x | xx.x | xx.x | xx.x | xx.x | XX.X | xx.: |
| Q3 | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | XX.X | xx.: |
| Max | XX | xx | XX | XX | xx | XX | XX | XX | x |



| Table B-3.1.2 | Age (years) at menarche at study entry, AT population, Complete cohort |
|---|---|
| Table B-3.1.3 | Age (years) at menarche at study entry, AT population, Starter |
| Table B-3.1.4 | Age (years) at menarche at study entry, AT population, Switcher |
| Table B-3.1.5 | Age (years) at menarche at study entry, AT population, Restarter |
| Table B-3.1.6 | Age (years) at menarche at study entry, AT population, Diagnosis confirmed by surgery |
| Table B-3.1.7 | Age (years) at menarche at study entry, AT population, Diagnosis based on clinical symptoms |
| Table B-3.1.8 | Age (years) at menarche at study entry, AT population, Germany |
| Table B-3.1.9 | Age (years) at menarche at study entry, AT population, Poland |
| Table B-3.1.10 | Age (years) at menarche at study entry, AT population, Hungary |
| Table B-3.1.11 | Age (years) at menarche at study entry, AT population, Switzerland |
| Table B-3.1.12 | Age (years) at menarche at study entry, AT population, Russia |
| Table B-3.1.13 | Age (years) at menarche at study entry, AT population, Ukraine |



Supporting document SOP BMT 01.09 – Doc 5002.02 – Effective date 21.03.2017

#### Section B-3.2 Pregnancy status at study entry

Table B-3.2.1 Pregnancy status at study entry, ITT population, Complete cohort

| | DNG | OAED | | | | NAED | | Allocation unknown | Total |
|---|---|---|---|---|---|---|---|---|---|
| | | GnRH-a | Danazol | All OAED | CC | Other progestin | All NAED | ** | |
| Number (%) of women | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) |
| Ever been pregnant | | | | | | | | | |
| Yes | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| No | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Missing | 0 ( 0.00%) | 0 ( 0.00%) | 0 ( 0.00%) | 0 ( 0.00%) | 0 ( 0.00%) | 0 ( 0.00%) | 0 ( 0.00%) | 0 ( 0.00%) | 0 ( 0.00%) |



| Table B-3.2.2 | Pregnancy status at study entry, AT population, Complete cohort |
|---|---|
| Table B-3.2.3 | Pregnancy status at study entry, AT population, Starter |
| Table B-3.2.4 | Pregnancy status at study entry, AT population, Switcher |
| Table B-3.2.5 | Pregnancy status at study entry, AT population, Restarter |
| Table B-3.2.6 | Pregnancy status at study entry, AT population, Diagnosis confirmed by surgery |
| Table B-3.2.7 | Pregnancy status at study entry, AT population, Diagnosis based on clinical symptoms |
| Table B-3.2.8 | Pregnancy status at study entry, AT population, Germany |
| Table B-3.2.9 | Pregnancy status at study entry, AT population, Poland |
| Table B-3.2.10 | Pregnancy status at study entry, AT population, Hungary |
| Table B-3.2.11 | Pregnancy status at study entry, AT population, Switzerland |
| Table B-3.2.12 | Pregnancy status at study entry, AT population, Russia |
| Table B-3.2.13 | Pregnancy status at study entry, AT population, Ukraine |



Section B-3.3 Number of live births, abortions, miscarriages and/or still births at study entry

Table B-3.3.1 Number of live births, abortions, miscarriages and/or still births at study entry, ITT population, Complete cohort

| | DNG | | OAED | | | NAED | | Allocation unknown | Total |
|---|---|---|---|---|---|---|---|---|---|
| | | GnRH-a | Danazol | All OAED | СС | Other progestin | All NAED | | |
| Number (%) of women ever been pregnant | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100% |
| Number of live births | | | | | | | | | |
| n | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x% |
| Missing | 0 ( 0.00%) | 0 ( 0.00%) | 0 ( 0.00%) | 0 ( 0.00%) | 0 ( 0.00%) | 0 ( 0.00%) | 0 ( 0.00%) | 0 ( 0.00%) | 0 ( 0.00% |
| Mean | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | XX.) |
| SD | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx | XX.XX | XX.XX | XX.XX |
| Min | xx | xx | xx | xx | xx | XX | XX | XX | XX |
| Q1 | xx.x | XX.X | XX.X | xx.x | XX.X | XX.X | XX.X | XX.X | XX. |
| Median | xx.x | XX.X | xx.x | xx.x | xx.x | xx.x | XX.X | XX.X | XX. |
| Q3 | xx.x | XX.X | xx.x | xx.x | xx.x | xx.x | XX.X | XX.X | XX. |
| Max | xx | XX | XX | XX | XX | XX | xx | xx | XX |
| Number of abortions/<br>miscariages/still births | | | | | | | | | |
| n | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x% |
| Missing | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x% |
| Mean | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | XX.) |
| SD | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx | XX.XX | XX.XX | xx.x |
| Min | xx | xx | XX | xx | xx | XX | XX | XX | x |
| Q1 | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | XX.X | XX.X | XX. |
| Median | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | XX.X | XX.X | XX. |
| Q3 | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | XX.X | XX.X | XX. |
| Max | XX | XX | XX | XX | XX | XX | xx | XX | x |



Supporting document SOP BMT 01.09 – Doc 5002.02 – Effective date 21.03.2017

| Table B-3.3.2 | Number of live births, miscarriages, abortions and/or still births at study entry, AT population, Complete cohort |
|---|---|
| Table B-3.3.3 | Number of live births, miscarriages, abortions and/or still births at study entry, AT population, Starter |
| Table B-3.3.4 | Number of live births, miscarriages, abortions and/or still births at study entry, AT population, Switcher |
| Table B-3.3.5 | Number of live births, miscarriages, abortions and/or still births at study entry, AT population, Restarter |
| Table B-3.3.6 | Number of live births, miscarriages, abortions and/or still births at study entry, AT population, Diagnosis confirmed by surgery |
| Table B-3.3.7 | Number of live births, miscarriages, abortions and/or still births at study entry, AT population, Diagnosis based on clinical symptoms |
| Table B-3.3.8 | Number of live births, miscarriages, abortions and/or still births at study entry, AT population, Germany |
| Table B-3.3.9 | Number of live births, miscarriages, abortions and/or still births at study entry, AT population, Poland |
| Table B-3.3.10 | Number of live births, miscarriages, abortions and/or still births at study entry, AT population, Hungary |
| Table B-3.3.11 | Number of live births, miscarriages, abortions and/or still births at study entry, AT population, Switzerland |
| Table B-3.3.12 | Number of live births, miscarriages, abortions and/or still births at study entry, AT population, Russia |
| Table B-3.3.13 | Number of live births, miscarriages, abortions and/or still births at study entry, AT population, Ukraine |



Supporting document SOP BMT 01.09 – Doc 5002.02 – Effective date 21.03.2017

#### Section B-4 Endometriosis characteristics

#### Section B-4.1 Time since first endometriosis symptoms at study entry

Table B-4.1.1 Time since first endometriosis symptoms at study entry, ITT population, Complete cohort

| | DNG | OAED | | | NAED | | | Allocation<br>unknown | Total |
|---|---|---|---|---|---|---|---|---|---|
| | | GnRH-a | Danazol | All OAED | CC | Other progestin | All NAED | | |
| Number (%) of women | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) |
| Time since first endometriosis | | | | | | | | | |
| symptoms | | | | | | | | | |
| < 6 months | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 6 months to <1 year | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 to <2 years | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 to <5 years | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 5 to <10 years | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| >=10 years | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Missing | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |



| Table B-4.1.2 | Time since first endometriosis symptoms at study entry, ITT population, Complete cohort |
|---|---|
| Table B-4.1.3 | Time since first endometriosis symptoms at study entry, AT population, Starter |
| Table B-4.1.4 | Time since first endometriosis symptoms at study entry, AT population, Switcher |
| Table B-4.1.5 | Time since first endometriosis symptoms at study entry, AT population, Restarter |
| Table B-4.1.6 | Time since first endometriosis symptoms at study entry, AT population, Diagnosis confirmed by surgery |
| Table B-4.1.7 | Time since first endometriosis symptoms at study entry, AT population, Diagnosis based on clinical symptoms |
| Table B-4.1.8 | Time since first endometriosis symptoms at study entry, AT population, Germany |
| Table B-4.1.9 | Time since first endometriosis symptoms at study entry, AT population, Poland |
| Table B-4.1.1 | Time since first endometriosis symptoms at study entry, AT population, Hungary |
| Table B-4.1.1 | 1 Time since first endometriosis symptoms at study entry, AT population, Switzerland |
| Table B-4.1.1 | 2 Time since first endometriosis symptoms at study entry, AT population, Russia |
| Table B-4.1.1 | 3 Time since first endometriosis symptoms at study entry, AT population, Ukraine |



Supporting document SOP BMT 01.09 – Doc 5002.02 – Effective date 21.03.2017

#### Section B-4.2 Time since first diagnosis of endometriosis at study entry

Table B-4.2.1 Time since first diagnosis of endometriosis at study entry, ITT population, Complete cohort

| | DNG | OAED | | | NAED | | | Allocation<br>unknown | Total |
|---|---|---|---|---|---|---|---|---|---|
| | | GnRH-a | Danazol | All OAED | CC | Other progestin | All NAED | | |
| Number (%) of women | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) |
| Time since first diagnosis of | | | | | | | | | |
| endometriosis | | | | | | | | | |
| < 6 months | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 6 months to <1 year | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 to <2 years | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 to <5 years | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 5 to <10 years | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| >=10 years | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Missing | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |



| Table B-4.2.2 | Time since first diagnosis of endometriosis at study entry, AT population, Complete cohort |
|---|---|
| Table B-4.2.3 | Time since first diagnosis of endometriosis at study entry, AT population, Starter |
| Table B-4.2.4 | Time since first diagnosis of endometriosis at study entry, AT population, Switcher |
| Table B-4.2.5 | Time since first diagnosis of endometriosis at study entry, AT population, Restarter |
| Table B-4.2.6 | Time since first diagnosis of endometriosis at study entry, AT population, Diagnosis confirmed by surgery |
| Table B-4.2.7 | Time since first diagnosis of endometriosis at study entry, AT population, Diagnosis based on clinical symptoms |
| Table B-4.2.8 | Time since first diagnosis of endometriosis at study entry, AT population, Germany |
| Table B-4.2.9 | Time since first diagnosis of endometriosis at study entry, AT population, Poland |
| Table B-4.2.10 | Time since first diagnosis of endometriosis at study entry, AT population, Hungary |
| Table B-4.2.11 | Time since first diagnosis of endometriosis at study entry, AT population, Switzerland |
| Table B-4.2.12 | Time since first diagnosis of endometriosis at study entry, AT population, Russia |
| Table B-4.2.13 | Time since first diagnosis of endometriosis at study entry, AT population, Ukraine |



Supporting document SOP BMT 01.09 – Doc 5002.02 – Effective date 21.03.2017

#### Section B-4.3 Time span between occurrence of endometriosis symptoms and diagnosis

Table B-4.3.1 Time span between occurrence of endometriosis symptoms and diagnosis, ITT population, Complete cohort

| | DNG | OAED | | | NAED | | | Allocation<br>unknown | Total |
|---|---|---|---|---|---|---|---|---|---|
| | | GnRH-a | Danazol | All OAED | CC | Other progestin | All NAED | | |
| Number (%) of women | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) |
| Time span between first | | | | | | | | | |
| endometriosis symptoms and | | | | | | | | | |
| diagnosis | | | | | | | | | |
| < 6 months | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 6 months to <1 year | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 to <2 years | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 to <5 years | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 5 to <10 years | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| >=10 years | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Missing | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |



| Table B-4.3.2 | Time span between occurrence of endometriosis symptoms and diagnosis, AT population, Complete cohort |
|---|---|
| Table B-4.3.3 | Time span between occurrence of endometriosis symptoms and diagnosis, AT population, Starter |
| Table B-4.3.4 | Time span between occurrence of endometriosis symptoms and diagnosis, AT population, Switcher |
| Table B-4.3.5 | Time span between occurrence of endometriosis symptoms and diagnosis, AT population, Restarter |
| Table B-4.3.6 | Time span between occurrence of endometriosis symptoms and diagnosis, AT population, Diagnosis confirmed by surgery |
| Table B-4.3.7 | Time span between occurrence of endometriosis symptoms and diagnosis, AT population, Diagnosis based on clinical symptoms |
| Table B-4.3.8 | Time span between occurrence of endometriosis symptoms and diagnosis, AT population, Germany |
| Table B-4.3.9 | Time span between occurrence of endometriosis symptoms and diagnosis, AT population, Poland |
| Table B-4.3.10 | Time span between occurrence of endometriosis symptoms and diagnosis, AT population, Hungary |
| Table B-4.3.11 | Time span between occurrence of endometriosis symptoms and diagnosis, AT population, Switzerland |
| Table B-4.3.12 | Time span between occurrence of endometriosis symptoms and diagnosis, AT population, Russia |
| Table B-4.3.13 | Time span between occurrence of endometriosis symptoms and diagnosis, AT population, Ukraine |



Supporting document SOP BMT 01.09 - Doc 5002.02 - Effective date 21.03.2017

Section B-4.4 Surgical procedures for the management of endometriosis during the past two years

Table B-4.4.1 Surgical procedures for the management of endometriosis during the past two years, ITT population, Complete cohort

| | DNG | OAED | | NAED | | | Allocation<br>unknown | Total | |
|---|---|---|---|---|---|---|---|---|---|
| | | GnRH-a | Danazol | All OAED | CC | Other progestin | All NAED | | |
| Number (%) of women | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) |
| Number of surgical procedures | | | | | | | | | |
| None | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3-4 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| >= 5 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Missing | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |



| Table B-4.4.2 | Surgical procedures for the management of endometriosis during the past two years, AT population, Complete cohort |
|---|---|
| Table B-4.4.3 | Surgical procedures for the management of endometriosis during the past two years, AT population, Starter |
| Table B-4.4.4 | Surgical procedures for the management of endometriosis during the past two years, AT population, Switcher |
| Table B-4.4.5 | Surgical procedures for the management of endometriosis during the past two years, AT population, Restarter |
| Table B-4.4.6 | Surgical procedures for the management of endometriosis during the past two years, AT population, Diagnosis confirmed by surgery |
| Table B-4.4.7 | Surgical procedures for the management of endometriosis during the past two years, AT population, Diagnosis based on clinical symptoms |
| Table B-4.4.8 | Surgical procedures for the management of endometriosis during the past two years, AT population, Germany |
| Table B-4.4.9 | Surgical procedures for the management of endometriosis during the past two years, AT population, Poland |
| Table B-4.4.10 | Surgical procedures for the management of endometriosis during the past two years, AT population, Hungary |
| Table B-4.4.11 | Surgical procedures for the management of endometriosis during the past two years, AT population, Switzerland |
| Table B-4.4.12 | Surgical procedures for the management of endometriosis during the past two years, AT population, Russia |
| Table B-4.4.13 | Surgical procedures for the management of endometriosis during the past two years, AT population, Ukraine |



Section B-4.5 Self-reported surgical procedures related to endometriosis at study entry,

Table B-4.5.1 Self-reported surgical procedures related to endometriosis at study entry, ITT population, Complete cohort

| | DNG | OAED | | | NAED | | | Allocation<br>unknown | Total |
|---|---|---|---|---|---|---|---|---|---|
| | | GnRH-a | Danazol | All OAED | CC | Other progestin | All NAED | | |
| Number (%) of women | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100% |
| Diagnostic surgical | | | | | | | | | |
| intervention | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x% |
| Therapeutic surgery | | | | | | | | | |
| (laparoscopic)* | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x% |
| Thereof | | | | | | | | | |
| Excisions of lesions / | | , | | , | , -0 | | | | , |
| adhesions | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | , , | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x% |
| Removal of ovarian cysts | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x% |
| Removal of ovary / fallopian | , -, | , | | | , -0 | | | | , . |
| tubes | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x% |
| Hysterectomy | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | • | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x% |
| Other | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x% |
| Therapeutic surgery (open | | | | | | | | | |
| abdominal) * | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x% |
| Thereof | | | | | | | | | |
| Excisions of lesions / | | | | | | | | | |
| adhesions | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x% |
| Removal of ovarian cysts | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x% |
| Removal of ovary / fallopian | | | | | | | | | |
| tubes | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x% |
| Hysterectomy | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x% |
| Other | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x% |



Supporting document SOP BMT 01.09 – Doc 5002.02 – Effective date 21.03.2017

| Therapeutic surgery (other, incl. type unknown)* | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
|---|---|---|---|---|---|---|---|---|---|
| Thereof | | | | | | | | | |
| Excisions of lesions / | | | | | | | | | |
| adhesions | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Removal of ovarian cysts | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Removal of ovary / fallopian | | | | | | | | | |
| tubes | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Hysterectomy | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Other | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

Note: \* Multiple answers possible.



| Table B-4.5.2 | Self-reported surgical procedures related to endometriosis at study entry, AT population, Complete cohort |
|---|---|
| Table B-4.5.3 | Self-reported surgical procedures related to endometriosis at study entry, AT population, Starter |
| Table B-4.5.4 | Self-reported surgical procedures related to endometriosis at study entry, AT population, Switcher |
| Table B-4.5.5 | Self-reported surgical procedures related to endometriosis at study entry, AT population, Restarter |
| Table B-4.5.6 | Self-reported surgical procedures related to endometriosis at study entry, AT population, Diagnosis confirmed by surgery |
| Table B-4.5.7 | Self-reported surgical procedures related to endometriosis at study entry, AT population, Diagnosis based on clinical symptoms |
| Table B-4.5.8 | Self-reported surgical procedures related to endometriosis at study entry, AT population, Germany |
| Table B-4.5.9 | Self-reported surgical procedures related to endometriosis at study entry, AT population, Poland |
| Table B-4.5.10 | Self-reported surgical procedures related to endometriosis at study entry, AT population, Hungary |
| Table B-4.5.11 | Self-reported surgical procedures related to endometriosis at study entry, AT population, Switzerland |
| Table B-4.5.12 | Self-reported surgical procedures related to endometriosis at study entry, AT population, Russia |
| Table B-4.5.13 | Self-reported surgical procedures related to endometriosis at study entry, AT population, Ukraine |

Supporting document SOP BMT 01.09 – Doc 5002.02 – Effective date 21.03.2017

Section B-4.6 Endometriosis associated symptoms at study entry

Table B-4.6.1 Endometriosis associated symptoms at study entry, ITT population, Complete cohort

| | DNG | OAED | | | NAED | | | Allocation<br>unknown | Total |
|---|---|---|---|---|---|---|---|---|---|
| | | GnRH-a | Danazol | All OAED | CC | Other progestin | All NAED | | |
| Number (%) of women | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) |
| Endometriosis associated | | | | | | | | | |
| symptoms* | | | | | | | | | |
| Pelvic pain | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Pain during or after sexual intercourse | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Difficulty conceiving / infertility | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Painful periods | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Heavy or irregular bleeding | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Pain when passing urine | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Pain during bowel movement | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Constipation or diarrhea | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Tiredness / weakness | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Other | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Missing | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Three selected pain symptoms* | | | | | | | | | |
| At least one | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| All three | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

Note: \* Multiple answers possible.

Note: \*\* Apply to pelvic pain, pain during or after sexual intercourse and painful periods



| Table B-4.6.2 | Endometriosis associated symptoms at study entry, AT population, Complete cohort |
|---|---|
| Table B-4.6.3 | Endometriosis associated symptoms at study entry, AT population, Starter |
| Table B-4.6.4 | Endometriosis associated symptoms at study entry, AT population, Switcher |
| Table B-4.6.5 | Endometriosis associated symptoms at study entry, AT population, Restarter |
| Table B-4.6.6 | Endometriosis associated symptoms at study entry, AT population, Diagnosis confirmed by surgery |
| Table B-4.6.7 | Endometriosis associated symptoms at study entry, AT population, Diagnosis based on clinical symptoms |
| Table B-4.6.8 | Endometriosis associated symptoms at study entry, AT population, Germany |
| Table B-4.6.9 | Endometriosis associated symptoms at study entry, AT population, Poland |
| Table B-4.6.10 | Endometriosis associated symptoms at study entry, AT population, Hungary |
| Table B-4.6.11 | Endometriosis associated symptoms at study entry, AT population, Switzerland |
| Table B-4.6.12 | Endometriosis associated symptoms at study entry, AT population, Russia |
| Table B-4.6.13 | Endometriosis associated symptoms at study entry, AT population, Ukraine |



Supporting document SOP BMT 01.09 – Doc 5002.02 – Effective date 21.03.2017

#### Section B-4.7 Disabling endometriosis associated pain preventing the woman from working or attending social events at study entry

Table B-4.7.1 Disabling endometriosis associated pain preventing the woman from working or attending social events at study entry, ITT population, Complete cohort

| | DNG | OAED | | | NAED | | | Allocation<br>unknown | Total |
|---|---|---|---|---|---|---|---|---|---|
| | | GnRH-a | Danazol | All OAED | CC | Other progestin | All NAED | | |
| Number (%) of women | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) |
| Disabling endometriosis associated pain* | | | | | | | | | |
| Yes | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| No | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Missing | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

Note:\* On at least two days in the last four weeks before study entry



| Table B-4.7.2 | Disabling endometriosis associated pain preventing the woman from working or attending social events at study entry, AT population, Complete cohort |
|---|---|
| Table B-4.7.3 | Disabling endometriosis associated pain preventing the woman from working or attending social events at study entry, AT population, Starter |
| Table B-4.7.4 | Disabling endometriosis associated pain preventing the woman from working or attending social events at study entry, AT population, Switcher |
| Table B-4.7.5 | Disabling endometriosis associated pain preventing the woman from working or attending social events at study entry, AT population, Restarter |
| Table B-4.7.6<br>by surge | Disabling endometriosis associated pain preventing the woman from working or attending social events at study entry, AT population, Diagnosis confirmed ry |
| Table B-4.7.7<br>clinical sy | Disabling endometriosis associated pain preventing the woman from working or attending social events at study entry, AT population, Diagnosis based on mptoms |
| Table B-4.7.8 | Disabling endometriosis associated pain preventing the woman from working or attending social events at study entry, AT population, Germany |
| Table B-4.7.9 | Disabling endometriosis associated pain preventing the woman from working or attending social events at study entry, AT population, Poland |
| Table B-4.7.10 | Disabling endometriosis associated pain preventing the woman from working or attending social events at study entry, AT population, Hungary |
| Table B-4.7.11 | Disabling endometriosis associated pain preventing the woman from working or attending social events at study entry, AT population, Switzerland |
| Table B-4.7.12 | Disabling endometriosis associated pain preventing the woman from working or attending social events at study entry, AT population, Russia |



Supporting document SOP BMT 01.09 – Doc 5002.02 – Effective date 21.03.2017

#### Section B-4.8 Severity of endometriosis associated pain at study entry

Table B-4.8.1 Severity of endometriosis associated pain at study entry, ITT population, Complete cohort

| | DNG | OAED | | | NAED | | | Allocation<br>unknown | Total |
|---|---|---|---|---|---|---|---|---|---|
| | | GnRH-a | Danazol | All OAED | CC | Other progestin | All NAED | | |
| Number (%) of women | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) |
| Pain severity score* | | | | | | | | | |
| Mild (0-3) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderate (4-7) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Severe (8-10) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Missing | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

Note: \*Pain severity score is defined from 0 (no pain) up to 10 (unbearable pain).



| Table B-4.8.2 | Severity of endometriosis associated pain at study entry, AT population, Complete cohort |
|---|---|
| Table B-4.8.3 | Severity of endometriosis associated pain at study entry, AT population, Starter |
| Table B-4.8.4 | Severity of endometriosis associated pain at study entry, AT population, Switcher |
| Table B-4.8.5 | Severity of endometriosis associated pain at study entry, AT population, Restarter |
| Table B-4.8.6 | Severity of endometriosis associated pain at study entry, AT population, Diagnosis confirmed by surgery |
| Table B-4.8.7 | Severity of endometriosis associated pain at study entry, AT population, Diagnosis based on clinical symptoms |
| Table B-4.8.8 | Severity of endometriosis associated pain at study entry, AT population, Germany |
| Table B-4.8.9 | Severity of endometriosis associated pain at study entry, AT population, Poland |
| Table B-4.8.10 | Severity of endometriosis associated pain at study entry, AT population, Hungary |
| Table B-4.8.11 | Severity of endometriosis associated pain at study entry, AT population, Switzerland |
| Table B-4.8.12 | Severity of endometriosis associated pain at study entry, AT population, Russia |
| Table B-4.8.13 | Severity of endometriosis associated pain at study entry, AT population, Ukraine |



Supporting document SOP BMT 01.09 - Doc 5002.02 - Effective date 21.03.2017

#### Section B-5 Medical history

Section B-5.1 Self-reported history of selected risk factors at study entry

Table B-5.1.1 Self-reported history of selected risk factors at study entry, ITT population, Complete cohort

| | DNG | OAED | | | NAED | | | Allocation<br>unknown | Total |
|---|---|---|---|---|---|---|---|---|---|
| | ****** | GnRH-a | Danazol | All OAED | CC | Other progestin | All NAED | | |
| Number (%) of women | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) |
| Endometriosis of relatives* | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Depression of relatives* | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Thrombosis or pulmonary embolism of relatives* | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| BMI >= 25.0 to <30.0 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| BMI >=30.0 to <35.0 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| BMI >= 35.0 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Smoker | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Heavy smoker (>15 cigarettes / day) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

Note: \* First-degree relatives only.



| Table B-5.1.2 | Self-reported history of selected risk factors at study entry, AT population, Complete cohort |
|---|---|
| Table B-5.1.3 | Self-reported history of selected risk factors at study entry, AT population, Starter |
| Table B-5.1.4 | Self-reported history of selected risk factors at study entry, AT population, Switcher |
| Table B-5.1.5 | Self-reported history of selected risk factors at study entry, AT population, Restarter |
| Table B-5.1.6 | Self-reported history of selected risk factors at study entry, AT population, Diagnosis confirmed by surgery |
| Table B-5.1.7 | Self-reported history of selected risk factors at study entry, AT population, Diagnosis based on clinical symptoms |
| Table B-5.1.8 | Self-reported history of selected risk factors at study entry, AT population, Germany |
| Table B-5.1.9 | Self-reported history of selected risk factors at study entry, AT population, Poland |
| Table B-5.1.10 | Self-reported history of selected risk factors at study entry, AT population, Hungary |
| Table B-5.1.11 | Self-reported history of selected risk factors at study entry, AT population, Switzerland |
| Table B-5.1.12 | Self-reported history of selected risk factors at study entry, AT population, Russia |
| Table B-5.1.13 | Self-reported history of selected risk factors at study entry, AT population, Ukraine |

Supporting document SOP BMT 01.09 – Doc 5002.02 – Effective date 21.03.2017

#### Section B-5.2 Self-reported history of selected diseases at study entry

Table B-5.2.1 Self-reported history of selected diseases at study entry, ITT population, Complete cohort

| | DNG | OAED | | | NAED | | | Allocation<br>unknown | Total |
|---|---|---|---|---|---|---|---|---|---|
| | | GnRH-a | Danazol | All OAED | CC | Other progestin | All NAED | | |
| Number (%) of women | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) |
| Depression* | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Anemia* | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Myocardial infarction* | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Stroke* | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Clotting lung (pulmonary embolism) * | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Deep venous thrombosis* | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Cancer* | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Other serious diseases* | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Any none endometriosis related surgery | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

Note: \* Treated by HCP only



| Self-reported history of selected diseases at study entry, AT population, Complete cohort |
|---|
| Self-reported history of selected diseases at study entry, AT population, Starter |
| Self-reported history of selected diseases at study entry, AT population, Switcher |
| Self-reported history of selected diseases at study entry, AT population, Restarter |
| Self-reported history of selected diseases at study entry, AT population, Diagnosis confirmed by surgery |
| Self-reported history of selected diseases at study entry, AT population, Diagnosis based on clinical symptoms |
| Self-reported history of selected diseases at study entry, AT population, Germany |
| Self-reported history of selected diseases at study entry, AT population, Poland |
| Self-reported history of selected diseases at study entry, AT population, Hungary |
| Self-reported history of selected diseases at study entry, AT population, Switzerland |
| Self-reported history of selected diseases at study entry, AT population, Russia |
| Self-reported history of selected diseases at study entry, AT population, Ukraine |

Supporting document SOP BMT 01.09 - Doc 5002.02 - Effective date 21.03.2017

#### Section B-6 Medication and other procedures for endometriosis treatment

Section B-6.1 Medication prescribed for the treatment of endometriosis during the past two years before study entry

Table B-6.1.1 Medication prescribed for the treatment of endometriosis during the past two years before study entry, ITT population, Complete cohort

| | DNG | OAED | | | NAED | | | Allocation<br>unknown | Total |
|---|---|---|---|---|---|---|---|---|---|
| | | GnRH-a | Danazol | All OAED | CC | Other progestin | All NAED | | |
| Number (%) of women | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) |
| Endometriosis medication | | | | | | | | | |
| Thereof* | | | | | | | | | |
| Category 1 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Category 2 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Category 3 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Categories <1% | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Missing | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

Note: \* Multiple answers possible



| Table B-6.1.2 | Medication prescribed for the treatment of endometriosis during the past two years before study entry, AT population, Complete cohort |
|---|---|
| Table B-6.1.3 | Medication prescribed for the treatment of endometriosis during the past two years before study entry, AT population, Starter |
| Table B-6.1.4 | Medication prescribed for the treatment of endometriosis during the past two years before study entry, AT population, Switcher |
| Table B-6.1.5 | Medication prescribed for the treatment of endometriosis during the past two years before study entry, AT population, Restarter |
| Table B-6.1.6 | Medication prescribed for the treatment of endometriosis during the past two years before study entry, AT population, Diagnosis confirmed by surgery |
| Table B-6.1.7 | Medication prescribed for the treatment of endometriosis during the past two years before study entry, AT population, Diagnosis based on clinical |
| symptom | S |
| Table B-6.1.8 | Medication prescribed for the treatment of endometriosis during the past two years before study entry, AT population, Germany |
| Table B-6.1.9 | Medication prescribed for the treatment of endometriosis during the past two years before study entry, AT population, Poland |
| Table B-6.1.10 | Medication prescribed for the treatment of endometriosis during the past two years before study entry, AT population, Hungary |
| Table B-6.1.11 | Medication prescribed for the treatment of endometriosis during the past two years before study entry, AT population, Switzerland |
| Table B-6.1.12 | Medication prescribed for the treatment of endometriosis during the past two years before study entry, AT population, Russia |
| Table B-6.1.13 | Medication prescribed for the treatment of endometriosis during the past two years before study entry, AT population, Ukraine |
Supporting document SOP BMT 01.09 – Doc 5002.02 – Effective date 21.03.2017

### Section B-6.2 Medication and other procedures for endometriosis treatment at study entry

Table B-6.2.1 Medication and other procedures for endometriosis treatment at study entry, ITT population, Complete cohort

| | DNG | | OAED | | NAED | | | Allocation<br>unknown | Total |
|---|---|---|---|---|---|---|---|---|---|
| | | GnRH-a | Danazol | All OAED | CC | Other progestin | All NAED | | |
| Number (%) of women | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) |
| Other measures taken for treatment of endometriosis Thereof* | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Non-prescription pain killers | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Natural/herbal products | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Acupuncture | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Dietary modification | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Massage/manual therapy | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Home remedies | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Other | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Nothing else | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Missing | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

Note: \* Multiple answers possible



| Table B-6.2.2 | Medication and other procedures for endometriosis treatment at study entry, AT population, Complete cohort |
|---|---|
| Table B-6.2.3 | Medication and other procedures for endometriosis treatment at study entry, AT population, Starter |
| Table B-6.2.4 | Medication and other procedures for endometriosis treatment at study entry, AT population, Switcher |
| Table B-6.2.5 | Medication and other procedures for endometriosis treatment at study entry, AT population, Restarter |
| Table B-6.2.6 | Medication and other procedures for endometriosis treatment at study entry, AT population, Diagnosis confirmed by surgery |
| Table B-6.2.7 | Medication and other procedures for endometriosis treatment at study entry, AT population, Diagnosis based on clinical symptoms |
| Table B-6.2.8 | Medication and other procedures for endometriosis treatment at study entry, AT population, Germany |
| Table B-6.2.9 | Medication and other procedures for endometriosis treatment at study entry, AT population, Poland |
| Table B-6.2.10 | Medication and other procedures for endometriosis treatment at study entry, AT population, Hungary |
| Table B-6.2.11 | Medication and other procedures for endometriosis treatment at study entry, AT population, Switzerland |
| Table B-6.2.12 | Medication and other procedures for endometriosis treatment at study entry, AT population, Russia |
| Table B-6.2.13 | Medication and other procedures for endometriosis treatment at study entry, AT population, Ukraine |

Supporting document SOP BMT 01.09 – Doc 5002.02 – Effective date 21.03.2017

### Section B-6.3 Regular use of other than endometriosis treatment medication at study entry

Table B-6.3.1 Regular use of other than endometriosis treatment medication at study entry, ITT population, Complete cohort

| | DNG | OAED | | NAED | | | Allocation<br>unknown | Total | |
|---|---|---|---|---|---|---|---|---|---|
| | | GnRH-a | Danazol | All OAED | CC | Other progestin | All NAED | | |
| Number (%) of women | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100% |
| Regular use of medication | | | | | | | | | |
| Any | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x% |
| Thereof* | | | | | | | | | |
| Category 1 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x% |
| Category 2 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x% |
| Category 3 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x% |
| Categories <1% | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x% |
| Missing | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x% |

Note: \*ATC (version: 2010), 1st level. Women may appear in more than one category.



| Table B-6.3.2 | Regular use of other than endometriosis treatment medication at study entry, AT population, Complete cohort |
|---|---|
| Table B-6.3.3 | Regular use of other than endometriosis treatment medication at study entry, AT population, Starter |
| Table B-6.3.4 | Regular use of other than endometriosis treatment medication at study entry, AT population, Switcher |
| Table B-6.3.5 | Regular use of other than endometriosis treatment medication at study entry, AT population, Restarter |
| Table B-6.3.6 | Regular use of other than endometriosis treatment medication at study entry, AT population, Diagnosis confirmed by surgery |
| Table B-6.3.7 | Regular use of other than endometriosis treatment medication at study entry, AT population, Diagnosis based on clinical symptoms |
| Table B-6.3.8 | Regular use of other than endometriosis treatment medication at study entry, AT population, Germany |
| Table B-6.3.9 | Regular use of other than endometriosis treatment medication at study entry, AT population, Poland |
| Table B-6.3.10 | Regular use of other than endometriosis treatment medication at study entry, AT population, Hungary |
| Table B-6.3.11 | Regular use of other than endometriosis treatment medication at study entry, AT population, Switzerland |
| Table B-6.3.12 | Regular use of other than endometriosis treatment medication at study entry, AT population, Russia |
| Table B-6.3.13 | Regular use of other than endometriosis treatment medication at study entry, AT population, Ukraine |



Supporting document SOP BMT 01.09 – Doc 5002.02 – Effective date 21.03.2017

### Section B-6.4 Psychotropic medication at study entry

Table B-6.4.1 Psychotropic medication at study entry, ITT population, Complete cohort

| | DNG | OAED | | NAED | | | Allocation<br>unknown | Total | |
|---|---|---|---|---|---|---|---|---|---|
| | | GnRH-a | Danazol | All OAED | CC | Other progestin | All NAED | | |
| Number (%) of women | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) |
| Psychotropic medication | | | | | | | | | |
| Category 1 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Category 2 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Category 3 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | ( 0() | ( 0() | ( 0() | / 0/) | 4 04) | / 0/) | ( 0() | 4 04) | ( 0() |
| Categories <1% | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Missing | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

Note: \*ATC (version: 2010), 3<sup>rd</sup> level. Women may appear in more than one category.



| Table B-6.4.2 | Psychotropic medication at study entry, AT population, Complete cohort |
|---|---|
| Table B-6.4.3 | Psychotropic medication at study entry, AT population, Starter |
| Table B-6.4.4 | Psychotropic medication at study entry, AT population, Switcher |
| Table B-6.4.5 | Psychotropic medication at study entry, AT population, Restarter |
| Table B-6.4.6 | Psychotropic medication at study entry, AT population, Diagnosis confirmed by surgery |
| Table B-6.4.7 | Psychotropic medication at study entry, AT population, Diagnosis based on clinical symptoms |
| Table B-6.4.8 | Psychotropic medication at study entry, AT population, Germany |
| Table B-6.4.9 | Psychotropic medication at study entry, AT population, Poland |
| Table B-6.4.10 | Psychotropic medication at study entry, AT population, Hungary |
| Table B-6.4.11 | Psychotropic medication at study entry, AT population, Switzerland |
| Table B-6.4.12 | Psychotropic medication at study entry, AT population, Russia |
| Table B-6.4.13 | Psychotropic medication at study entry, AT population, Ukraine |



Supporting document SOP BMT 01.09 – Doc 5002.02 – Effective date 21.03.2017

### Section B-7 Distribution and selected baseline characteristics of Visanne long-term user

#### Section B-7.1 Duration of Visanne use

Table B-7.1.1 Duration of Visanne use

| | DNG long-term user* |
|--------------------------|---------------------|
| Number (%) of women | xx ( 100%) |
| Duration of DNG use | |
| 15 months to < 24 months | xx ( xx.x%) |
| 24 months to < 30 months | xx ( xx.x%) |
| 30 months to < 36 months | xx ( xx.x%) |
| 36 months to < 42 months | xx ( xx.x%) |
| 42 months to < 48 months | xx ( xx.x%) |
| 48 months to < 54 months | xx ( xx.x%) |
| 54 months to < 60 months | xx ( xx.x%) |
| 60 months to < 66 months | xx ( xx.x%) |
| 66 months to < 72 months | xx ( xx.x%) |
| 72 months to < 78 months | xx ( xx.x%) |
| 78 months to < 84 months | xx ( xx.x%) |
| 84 months and more | xx ( xx.x%) |

Note: \*Long-term: defined as continuous use for >= 15 months. They may have started with other than DNG treatment.



| Table B-7.1.2 | Duration of Visanne use, Starter |
|---|---|
| Table B-7.1.3 | Duration of Visanne use, Switcher |
| Table B-7.1.4 | Duration of Visanne use, Restarter |
| Table B-7.1.5 | Duration of Visanne use, Diagnosis confirmed by surgery |
| Table B-7.1.6 | Duration of Visanne use, Diagnosis based on clinical symptoms |
| Table B-7.1.7 | Duration of Visanne use, Germany |
| Table B-7.1.8 | Duration of Visanne use, Poland |
| Table B-7.1.9 | Duration of Visanne use, Hungary |
| Table B-7.1.10 | Duration of Visanne use, Switzerland |
| Table B-7.1.11 | Duration of Visanne use, Russia |
| Table B-7.1.12 | Duration of Visanne use. Ukraine |



Supporting document SOP BMT 01.09 – Doc 5002.02 – Effective date 21.03.2017

#### Section B-7.2 Regional distribution

Table B-7.2.1 Regional distribution

| | DNG long-term user* |
|---------------------|---------------------|
| Number (%) of women | xx (100 %) |
| Germany | xx ( xx.x%) |
| Poland | xx ( xx.x%) |
| Russia | xx ( xx.x%) |
| Hungary | xx ( xx.x%) |
| Switzerland | xx ( xx.x%) |
| Ukraine | xx ( xx.x%) |

Note: \*Long-term: defined as continuous use for >= 15 months. They may have started with other than DNG treatment



| Table B-7.2.2 | Regional distribution, Starter |
|---------------|-------------------------------------------------------------|
| Table B-7.2.3 | Regional distribution, Switcher |
| Table B-7.2.4 | Regional distribution, Restarter |
| Table B-7.2.5 | Regional distribution, Diagnosis confirmed by surgery |
| Table B-7.2.6 | Regional distribution, Diagnosis based on clinical symptoms |



Supporting document SOP BMT 01.09 – Doc 5002.02 – Effective date 21.03.2017

#### Section B-7.3 Diagnosis classification at study entry

Table B-7.3.1 Diagnosis classification at study entry

| | DNG long-term user* |
|--------------------------------|---------------------|
| Number (%) of women | xx ( 100%) |
| Surgically confirmed diagnosis | xx ( xx.x%) |
| Clinically confirmed diagnosis | xx ( xx.x%) |

Note: \*Long-term: defined as continuous use for >= 15 months. They may have started with other than

DNG treatment Date of analysis:



| Table B-7.3.2 | Diagnosis classification at study entry, Starter |
|----------------|------------------------------------------------------|
| Table B-7.3.3 | Diagnosis classification at study entry, Switcher |
| Table B-7.3.4 | Diagnosis classification at study entry, Restarter |
| Table B-7.3.5 | Diagnosis classification at study entry, Germany |
| Table B-7.3.6 | Diagnosis classification at study entry, Poland |
| Table B-7.3.7 | Diagnosis classification at study entry, Hungary |
| Table B-7.3.8 | Diagnosis classification at study entry, Switzerland |
| Table B-7.3.9 | Diagnosis classification at study entry, Russia |
| Table B-7.3.10 | Diagnosis classification at study entry, Ukraine |



Supporting document SOP BMT 01.09 – Doc 5002.02 – Effective date 21.03.2017

### Section B-7.4 Age (years) at study entry

Table B-7.4.1 Age (years) at study entry

| | DNG long-term user* |
|--------------------------------------|---------------------|
| Number (%) of Visanne long-term user | xx ( 100%) |
| Age (years) | |
| n | xx ( xx.x%) |
| Missing | 0 ( 0.00%) |
| Mean | xx.x |
| SD | xx.xx |
| Min | XX |
| Q1 | XX.X |
| Median | XX.X |
| Q3 | XX.X |
| Max | xx |
| Adolescents <18 years | xx ( xx.x%) |
| Age category | |
| <20 years | xx ( xx.x%) |
| 20 to <30 years | xx ( xx.x%) |
| 30 to <40 years | xx ( xx.x%) |
| ≥40 years | xx ( xx.x%) |
| Missing | 0 ( 0.00%) |

Note: \*Long-term user: defined as continuous use for >= 15 months. They may have started with other than DNG treatment



| Table B-7.4.2 | Age (years) at study entry, Starter |
|---|---|
| Table B-7.4.3 | Age (years) at study entry, Switcher |
| Table B-7.4.4 | Age (years) at study entry, Restarter |
| Table B-7.4.5 | Age (years) at study entry, Diagnosis confirmed by surgery |
| Table B-7.4.6 | Age (years) at study entry, Diagnosis based on clinical symptoms |
| Table B-7.4.7 | Age (years) at study entry, Germany |
| Table B-7.4.8 | Age (years) at study entry, Poland |
| Table B-7.4.9 | Age (years) at study entry, Hungary |
| Table B-7.4.10 | Age (years) at study entry, Switzerland |
| Table B-7.4.11 | Age (years) at study entry, Russia |
| Table B-7.4.12 | Age (years) at study entry, Ukraine |



Supporting document SOP BMT 01.09 – Doc 5002.02 – Effective date 21.03.2017

### Section B-7.5 Body Mass Index (BMI) at study entry

Table B-7.5.1 Body Mass Index (BMI) at study entry

| | DNG long-term user* |
|--------------------------------------|---------------------|
| Number (%) of Visanne long-term user | xx ( 100%) |
| BMI (kg/m²) | |
| n | xx ( xx.x%) |
| Missing | xx ( xx.x%) |
| Mean | xx.x |
| SD | XX.XX |
| Min | XX |
| Q1 | XX.X |
| Median | XX.X |
| Q3 | XX.X |
| Max | xx |
| BMI category | |
| <20 | xx ( xx.x%) |
| 20 to <25 | xx ( xx.x%) |
| 25 to <30 | xx ( xx.x%) |
| 30 to <35 | xx ( xx.x%) |
| ≥35 | xx ( xx.x%) |
| Missing | xx ( xx.x%) |

Note: \*Long-term user: defined as continuous use for >= 15 months. They may have started with other than DNG treatment



| Table B-7.5.2 | Body Mass Index (BMI) at study entry, Starter |
|---|---|
| Table B-7.5.3 | Body Mass Index (BMI) at study entry, Switcher |
| Table B-7.5.4 | Body Mass Index (BMI) at study entry, Restarter |
| Table B-7.5.5 | Body Mass Index (BMI) at study entry, Diagnosis confirmed by surgery |
| Table B-7.5.6 | Body Mass Index (BMI) at study entry, Diagnosis based on clinical symptoms |
| Table B-7.5.7 | Body Mass Index (BMI) at study entry, Germany |
| Table B-7.5.8 | Body Mass Index (BMI) at study entry, Poland |
| Table B-7.5.9 | Body Mass Index (BMI) at study entry, Hungary |
| Table B-7.5.10 | Body Mass Index (BMI) at study entry, Switzerland |
| Table B-7.5.11 | Body Mass Index (BMI) at study entry, Russia |
| Table B-7.5.12 | Body Mass Index (BMI) at study entry, Ukraine |

Supporting document SOP BMT 01.09 - Doc 5002.02 - Effective date 21.03.2017

#### Section B-7.6 Endometriosis associated symptoms at study entry

Table B-7.6.1 Endometriosis associated symptoms at study entry

| | DNG long-term user* |
|-----------------------------------------|---------------------|
| Number (%) of women | xx ( 100%) |
| Endometriosis associated symptoms ** | |
| Pelvic pain | xx ( xx.x%) |
| Pain during or after sexual intercourse | xx ( xx.x%) |
| Difficulty conceiving / infertility | xx ( xx.x%) |
| Painful periods | xx ( xx.x%) |
| Heavy or irregular bleeding | xx ( xx.x%) |
| Pain when passing urine | xx ( xx.x%) |
| Pain during bowel movement | xx ( xx.x%) |
| Constipation or diarrhea | xx ( xx.x%) |
| Tiredness / weakness | xx ( xx.x%) |
| Other | xx ( xx.x%) |
| Missing | xx ( xx.x%) |
| At least one pain symptom*** | xx ( xx.x%) |
| All three pain symptoms*** | xx ( xx.x%) |

Note: \*Long-term user: defined as continuous use for >= 15 months. They may have started with other than DNG treatment

Note: \*\* Multiple answers possible

Note: Multiple answers possible

Note: \*\*\* Apply to pelvic pain, pain during or after sexual intercourse and painful periods



| Table B-7.6.2 | Endometriosis associated symptoms at study entry, Starter |
|---|---|
| Table B-7.6.3 | Endometriosis associated symptoms at study entry, Switcher |
| Table B-7.6.4 | Endometriosis associated symptoms at study entry, Restarter |
| Table B-7.6.5 | Endometriosis associated symptoms at study entry, Diagnosis confirmed by surgery |
| Table B-7.6.6 | Endometriosis associated symptoms at study entry, Diagnosis based on clinical symptoms |
| Table B-7.6.7 | Endometriosis associated symptoms at study entry, Germany |
| Table B-7.6.8 | Endometriosis associated symptoms at study entry, Poland |
| Table B-7.6.9 | Endometriosis associated symptoms at study entry, Hungary |
| Table B-7.6.10 | Endometriosis associated symptoms at study entry, Switzerland |
| Table B-7.6.11 | Endometriosis associated symptoms at study entry, Russia |
| Table B-7.6.12 | Endometriosis associated symptoms at study entry, Ukraine |



Supporting document SOP BMT 01.09 – Doc 5002.02 – Effective date 21.03.2017

#### Section B-7.7 Endometriosis associated pain severity score at study entry

Table B-7.7.1 Endometriosis associated pain severity score at study entry

| | DNG long-term user* |
|-----------------------|---------------------|
| Number (%) of women | xx ( 100%) |
| Pain severity score** | |
| Mild (0-3) | xx ( xx.x%) |
| Moderate (4-7) | xx ( xx.x%) |
| Severe (8-10) | xx ( xx.x%) |
| Missing | xx ( xx.x%) |

Note: \*Long-term user: defined as continuous use for >= 15 months. They may have started with other than DNG treatment

Note: \*\* Pain severity score is defined from 0 (no pain) up to 10 (unbearable pain) Date of analysis:



| Table B-7.7.2 | Endometriosis associated pain severity score at study entry, Starter |
|---|---|
| Table B-7.7.3 | Endometriosis associated pain severity score at study entry, Switcher |
| Table B-7.7.4 | Endometriosis associated pain severity score at study entry, Restarter |
| Table B-7.7.5 | Endometriosis associated pain severity score at study entry, Diagnosis confirmed by surgery |
| Table B-7.7.6 | Endometriosis associated pain severity score at study entry, Diagnosis based on clinical symptoms |
| Table B-7.7.7 | Endometriosis associated pain severity score at study entry, Germany |
| Table B-7.7.8 | Endometriosis associated pain severity score at study entry, Poland |
| Table B-7.7.9 | Endometriosis associated pain severity score at study entry, Hungary |
| Table B-7.7.10 | Endometriosis associated pain severity score at study entry, Switzerland |
| Table B-7.7.11 | Endometriosis associated pain severity score at study entry, Russia |
| Table B-7.7.12 | Endometriosis associated pain severity score at study entry, Ukraine |



Supporting document SOP BMT 01.09 – Doc 5002.02 – Effective date 21.03.2017

### Section B-8 Follow-up characteristics

Section B-8.1 Mood symptoms at study entry

Table B-8.1.1 Mood symptoms at study entry, ITT population, Complete cohort

| | DNG | | OAED | | | NAED | Allocation unknown | Total | |
|---|---|---|---|---|---|---|---|---|---|
| | | GnRH-a | Danazol | All OAED | CC | Other progestin | All NAED | | |
| Number (%) of women* | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) |
| Feeling down, depressed or | | | | | | | | | |
| hopeless | | | | | | | | | |
| Never | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Rarely | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Sometimes | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Often | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Always | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Missing | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Feeling like being a failure and | | | | | | | | | |
| have let down friends and/or | | | | | | | | | |
| family | | | | | | | | | |
| ··· | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Feeling happy or optimistic | | | | | | | | | |
| about the future | | | | | | | | | |
| | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Mood Score** | | | | | | | | | |
| Mean (± SD) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) |

Note: \* Allocation to user cohorts is defined according to current EMT use.



Supporting document SOP BMT 01.09 – Doc 5002.02 – Effective date 21.03.2017

Note:  $^{**}$  Mood score is calculated as described in the SAP Appendix IV Date of analysis:

| Table B-8.1.2 | Mood symptoms at study entry, AT population, Complete cohort |
|---|---|
| Table 0-0.1.2 | wood symptoms at study entry, AT population, complete conort |
| Table B-8.1.3 | Mood symptoms at study entry, AT population, Starter |
| Table B-8.1.4 | Mood symptoms at study entry, AT population, Switcher |
| Table B-8.1.5 | Mood symptoms at study entry, AT population, Restarter |
| Table B-8.1.6 | Mood symptoms at study entry, AT population, Diagnosis confirmed by surgery |
| Table B-8.1.7 | Mood symptoms at study entry, AT population, Diagnosis based on clinical symptoms |
| Table B-8.1.8 | Mood symptoms at study entry, AT population, Germany |
| Table B-8.1.9 | Mood symptoms at study entry, AT population, Poland |
| Table B-8.1.10 | Mood symptoms at study entry, AT population, Hungary |
| Table B-8.1.11 | Mood symptoms at study entry, AT population, Switzerland |
| Table B-8.1.12 | Mood symptoms at study entry, AT population, Russia |
| Table B-8.1.13 | Mood symptoms at study entry, AT population, Ukraine |



Supporting document SOP BMT 01.09 - Doc 5002.02 - Effective date 21.03.2017

Section B-8.2 Mood symptoms at 6 months after study entry

Table B-8.2.1 Mood symptoms at 6 months after study entry, ITT population, Complete cohort

Table B-8.2.2 Mood symptoms at 6 months after study entry, AT population, Complete cohort

| | DNG | | OAED | | | NAED | | Ex-use | Allocation<br>unknown | Total |
|---|---|---|---|---|---|---|---|---|---|---|
| | | GnRH-a | Danazol | All OAED | CC | Other<br>progestin | All NAED | | | |
| Number (%) of women* | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) |
| Feeling down, depressed or | | | | | | | | | | |
| hopeless | | | | | | | | | | |
| Never | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Rarely | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Sometimes | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Often | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Always | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Missing | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Feeling like being a failure and | | | | | | | | | | |
| have let down friends and/or | | | | | | | | | | |
| family | | | | | | | | | | |
| | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Feeling happy or optimistic | | | | | | | | | | |
| about the future | | | | | | | | | | |
| | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| ** | | | | | | | | | | |
| Mood Score** | | | | 4. | | 4. | | | | 4. |
| Mean (± SD) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) |

Note: \* Allocation to user cohorts is defined according to current EMT use.

Note: \*\* Mood score is calculated as described in the SAP Appendix IV.



Supporting document SOP BMT 01.09 – Doc 5002.02 – Effective date 21.03.2017

| Table B-8.2.3 | Mood symptoms at 6 months after study entry, AT population, Starter |
|---|---|
| Table B-8.2.4 | Mood symptoms at 6 months after study entry, AT population, Switcher |
| Table B-8.2.5 | Mood symptoms at 6 months after study entry, AT population, Restarter |
| Table B-8.2.6 | Mood symptoms at 6 months after study entry, AT population, Diagnosis confirmed by surgery |
| Table B-8.2.7 | Mood symptoms at 6 months after study entry, AT population, Diagnosis based on clinical symptoms |
| Table B-8.2.8 | Mood symptoms at 6 months after study entry, AT population, Germany |
| Table B-8.2.9 | Mood symptoms at 6 months after study entry, AT population, Poland |
| Table B-8.2.10 | Mood symptoms at 6 months after study entry, AT population, Hungary |
| Table B-8.2.11 | Mood symptoms at 6 months after study entry, AT population, Switzerland |
| Table B-8.2.12 | Mood symptoms at 6 months after study entry, AT population, Russia |
| Table B-8.2.13 | Mood symptoms at 6 months after study entry, AT population, Ukraine |



| Section B-8.3 | Mood symptoms at 12 months after study entry |
|---|---|
| Table B-8.3.1 | Mood symptoms at 12 months after study entry, ITT population, Complete cohort |
| Table B-8.3.2 | Mood symptoms at 12 months after study entry, AT population, Complete cohort |
| Table B-8.3.3 | Mood symptoms at 12 months after study entry, AT population, Starter |
| Table B-8.3.4 | Mood symptoms at 12 months after study entry, AT population, Switcher |
| Table B-8.3.5 | Mood symptoms at 12 months after study entry, AT population, Restarter |
| Table B-8.3.6 | Mood symptoms at 12 months after study entry, AT population, Diagnosis confirmed by surgery |
| Table B-8.3.7 | Mood symptoms at 12 months after study entry, AT population, Diagnosis based on clinical symptoms |
| Table B-8.3.8 | Mood symptoms at 12 months after study entry, AT population, Germany |
| Table B-8.3.9 | Mood symptoms at 12 months after study entry, AT population, Poland |
| Table B-8.3.10 | Mood symptoms at 12 months after study entry, AT population, Hungary |
| Table B-8.3.11 | Mood symptoms at 12 months after study entry, AT population, Switzerland |
| Table B-8.3.12 | Mood symptoms at 12 months after study entry, AT population, Russia |
| Table B-8.3.13 | Mood symptoms at 12 months after study entry, AT population, Ukraine |
| Section B-8.4 | Mood symptoms at 24 months after study entry |
| Table B-8.4.1 | Mood symptoms at 24 months after study entry, ITT population, Complete cohort |
| Table B-8.4.2 | Mood symptoms at 24 months after study entry, AT population, Complete cohort |
| Table B-8.4.3 | Mood symptoms at 24 months after study entry, AT population, Starter |
| Table B-8.4.4 | Mood symptoms at 24 months after study entry, AT population, Switcher |
| Table B-8.4.5 | Mood symptoms at 24 months after study entry, AT population, Restarter |
| Table B-8.4.6 | Mood symptoms at 24 months after study entry, AT population, Diagnosis confirmed by surgery |
| Table B-8.4.7 | Mood symptoms at 24 months after study entry, AT population, Diagnosis based on clinical symptoms |
| Table B-8.4.8 | Mood symptoms at 24 months after study entry, AT population, Germany |



| Table B-8.4.9 | Mood symptoms at 24 months after study entry, AT population, Poland |
|---|---|
| Table B-8.4.10 | Mood symptoms at 24 months after study entry, AT population, Hungary |
| Table B-8.4.11 | Mood symptoms at 24 months after study entry, AT population, Switzerland |
| Table B-8.4.12 | Mood symptoms at 24 months after study entry, AT population, Russia |
| Table B-8.4.13 | Mood symptoms at 24 months after study entry, AT population, Ukraine |
| Section B-8.5 | Mood symptoms at 36 months after study entry |
| Table B-8.5.1 | Mood symptoms at 36 months after study entry, ITT population, Complete cohort |
| Table B-8.5.2 | Mood symptoms at 36 months after study entry, AT population, Complete cohort |
| Table B-8.5.3 | Mood symptoms at 36 months after study entry, AT population, Starter |
| Table B-8.5.4 | Mood symptoms at 36 months after study entry, AT population, Switcher |
| Table B-8.5.5 | Mood symptoms at 36 months after study entry, AT population, Restarter |
| Table B-8.5.6 | Mood symptoms at 36 months after study entry, AT population, Diagnosis confirmed by surgery |
| Table B-8.5.7 | Mood symptoms at 36 months after study entry, AT population, Diagnosis based on clinical symptoms |
| Table B-8.5.8 | Mood symptoms at 36 months after study entry, AT population, Germany |
| Table B-8.5.9 | Mood symptoms at 36 months after study entry, AT population, Poland |
| Table B-8.5.10 | Mood symptoms at 36 months after study entry, AT population, Hungary |
| Table B-8.5.11 | Mood symptoms at 36 months after study entry, AT population, Switzerland |
| Table B-8.5.12 | Mood symptoms at 36 months after study entry, AT population, Russia |
| Table B-8.5.13 | Mood symptoms at 36 months after study entry, AT population, Ukraine |
| Section B-8.6 | Mood symptoms at 48 months after study entry |
| Table B-8.6.1 | Mood symptoms at 48 months after study entry, ITT population, Complete cohort |
| Table B-8.6.2 | Mood symptoms at 48 months after study entry, AT population, Complete cohort |



| Table B-8.6.3 | Mood symptoms at 48 months after study entry, AT population, Starter |
|---|---|
| Table B-8.6.4 | Mood symptoms at 48 months after study entry, AT population, Switcher |
| Table B-8.6.5 | Mood symptoms at 48 months after study entry, AT population, Restarter |
| Table B-8.6.6 | Mood symptoms at 48 months after study entry, AT population, Diagnosis confirmed by surgery |
| Table B-8.6.7 | Mood symptoms at 48 months after study entry, AT population, Diagnosis based on clinical symptoms |
| Table B-8.6.8 | Mood symptoms at 48 months after study entry, AT population, Germany |
| Table B-8.6.9 | Mood symptoms at 48 months after study entry, AT population, Poland |
| Table B-8.6.10 | Mood symptoms at 48 months after study entry, AT population, Hungary |
| Table B-8.6.11 | Mood symptoms at 48 months after study entry, AT population, Switzerland |
| Table B-8.6.12 | Mood symptoms at 48 months after study entry, AT population, Russia |
| Table B-8.6.13 | Mood symptoms at 48 months after study entry, AT population, Ukraine |
| Section B-8.7 | Mood symptoms at 60 months after study entry |
| Table B-8.7.1 | Mood symptoms at 60 months after study entry, ITT population, Complete cohort |
| Table B-8.7.2 | Mood symptoms at 60 months after study entry, AT population, Complete cohort |
| Table B-8.7.3 | Mood symptoms at 60 months after study entry, AT population, Starter |
| Table B-8.7.4 | Mood symptoms at 60 months after study entry, AT population, Switcher |
| Table B-8.7.5 | Mood symptoms at 60 months after study entry, AT population, Restarter |
| Table B-8.7.6 | Mood symptoms at 60 months after study entry, AT population, Diagnosis confirmed by surgery |
| Table B-8.7.7 | Mood symptoms at 60 months after study entry, AT population, Diagnosis based on clinical symptoms |
| Table B-8.7.8 | Mood symptoms at 60 months after study entry, AT population, Germany |
| Table B-8.7.9 | Mood symptoms at 60 months after study entry, AT population, Poland |
| Table B-8.7.10 | Mood symptoms at 60 months after study entry, AT population, Hungary |
| Table B-8.7.11 | Mood symptoms at 60 months after study entry, AT population, Switzerland |
| Table R-8 7 12 | Mood symptoms at 60 months after study entry. AT population, Russia |



Supporting document SOP BMT 01.09 – Doc 5002.02 – Effective date 21.03.2017

### Table B-8.7.13 Mood symptoms at 60 months after study entry, AT population, Ukraine

| Section B-8.8 | Mood symptoms at 72 months after study entry |
|---|---|
| Table B-8.8.1 | Mood symptoms at 72 months after study entry, ITT population, Complete cohort |
| Table B-8.8.2 | Mood symptoms at 72 months after study entry, AT population, Complete cohort |
| Table B-8.8.3 | Mood symptoms at 72 months after study entry, AT population, Starter |
| Table B-8.8.4 | Mood symptoms at 72 months after study entry, AT population, Switcher |
| Table B-8.8.5 | Mood symptoms at 72 months after study entry, AT population, Restarter |
| Table B-8.8.6 | Mood symptoms at 72 months after study entry, AT population, Diagnosis confirmed by surgery |
| Table B-8.8.7 | Mood symptoms at 72 months after study entry, AT population, Diagnosis based on clinical symptoms |
| Table B-8.8.8 | Mood symptoms at 72 months after study entry, AT population, Germany |
| Table B-8.8.9 | Mood symptoms at 72 months after study entry, AT population, Poland |
| Table B-8.8.10 | Mood symptoms at 72 months after study entry, AT population, Hungary |
| Table B-8.8.11 | Mood symptoms at 72 months after study entry, AT population, Switzerland |
| Table B-8.8.12 | Mood symptoms at 72 months after study entry, AT population, Russia |
| Table B-8.8.13 | Mood symptoms at 72 months after study entry, AT population, Ukraine |
| Section B-8.9 | Mood symptoms at 84 months after study entry |
| Table B-8.9.1 | Mood symptoms at 84 months after study entry, ITT population, Complete cohort |
| Table B-8.9.2 | Mood symptoms at 84 months after study entry, AT population, Complete cohort |
| Table B-8.9.3 | Mood symptoms at 84 months after study entry, AT population, Starter |
| Table B-8.9.4 | Mood symptoms at 84 months after study entry, AT population, Switcher |
| Table B-8.9.5 | Mood symptoms at 84 months after study entry, AT population, Restarter |
| Table B-8.9.6 | Mood symptoms at 84 months after study entry, AT population, Diagnosis confirmed by surgery |



| Table B-8.9.7 | Mood symptoms at 84 months after study entry, AT population, Diagnosis based on clinical symptoms |
|---|---|
| Table B-8.9.8 | Mood symptoms at 84 months after study entry, AT population, Germany |
| Table B-8.9.9 | Mood symptoms at 84 months after study entry, AT population, Poland |
| Table B-8.9.10 | Mood symptoms at 84 months after study entry, AT population, Hungary |
| Table B-8.9.11 | Mood symptoms at 84 months after study entry, AT population, Switzerland |
| Table B-8.9.12 | Mood symptoms at 84 months after study entry, AT population, Russia |
| Table B-8.9.13 | Mood symptoms at 84 months after study entry, AT population, Ukraine |

Supporting document SOP BMT 01.09 – Doc 5002.02 – Effective date 21.03.2017

Section B-8.10 Change of Mood Score after study entry, constant user only

Table B-8.10.1 Change of Mood Score after study entry, constant user only\*, AT population, Complete cohort

| | DNG | | OAED | OAED | | NAED | Allocation<br>unknown | Total | |
|---|---|---|---|---|---|---|---|---|---|
| | | GnRH-a | Danazol | All OAED | СС | Other<br>progestin | All NAED | | |
| Number (%) of women | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) |
| Change of Mood Score** | | | | | | | | | |
| N | | | | | | | | | |
| Mean (± SD) | | | | | | | | | |
| Change from Baseline to 6 | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| months follow up | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) |
| Change from Baseline to 12 | xx | xx | XX | xx | XX | xx | xx | XX | xx |
| months follow up | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) |
| Change from Baseline to 24 | XX | XX | XX | xx | XX | xx | xx | XX | xx |
| months follow up | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) |
| Change from Baseline to 36 | xx | xx | XX | xx | XX | xx | xx | XX | xx |
| months follow up | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) |
| Change from Baseline to 48 | XX | XX | XX | xx | XX | xx | xx | XX | xx |
| months follow up | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) |
| Change from Baseline to 60 | XX | XX | XX | xx | XX | xx | xx | XX | xx |
| months follow up | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) |
| Change from Baseline to 72 | xx | xx | XX | xx | XX | xx | xx | XX | xx |
| months follow up | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) |
| Change from Baseline to 84 | xx | xx | xx | xx | XX | xx | xx | XX | XX |
| months follow up | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) |

Note:\* Only women who continuously used their baseline prescription are considered



Supporting document SOP BMT 01.09 – Doc 5002.02 – Effective date 21.03.2017

Note: \*\* Mood score is calculated as described in the SAP Appendix IV.

Date of analysis:

| Table B-8.10.2 | Change of Mood Score after study entry, constant user only*, AT population, Starter |
|---|---|
| Table B-8.10.3 | Change of Mood Score after study entry, constant user only *, AT population, Switcher |
| Table B-8.10.4 | Change of Mood Score after study entry, constant user only *, AT population, Restarter |
| Table B-8.10.5 | Change of Mood Score after study entry, constant user only *, AT population, Diagnosis confirmed by surgery |
| Table B-8.10.6 | Change of Mood Score after study entry, constant user only *, AT population, Diagnosis based on clinical symptoms |
| Table B-8.10.7 | Change of Mood Score after study entry, constant user only *, AT population, Germany |
| Table B-8.10.8 | Change of Mood Score after study entry, constant user only *, AT population, Poland |
| Table B-8.10.9 | Change of Mood Score after study entry, constant user only *, AT population, Hungary |
| Table B-8.10.10 | Change of Mood Score after study entry, constant user only *, AT population, Switzerland |
| Table B-8.10.11 | Change of Mood Score after study entry, constant user only *, AT population, Russia |
| Table B-8.10.12 | Change of Mood Score after study entry, constant user only *, AT population, Ukraine |

Supporting document SOP BMT 01.09 - Doc 5002.02 - Effective date 21.03.2017

Section B-8.11 Change of Mood Score after study entry, switcher only

Table B-8.11.1 Change of Mood Score after study entry, switcher only \*, AT population, Complete cohort

| | DNG | | OAED | | | NAED | Allocation<br>unknown | Total | |
|---|---|---|---|---|---|---|---|---|---|
| | | GnRH-a | Danazol | All OAED | CC | Other<br>progestin | All NAED | | |
| Number (%) of women | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) |
| Change of Mood Score** | | | | | | | | | |
| N | | | | | | | | | |
| Mean (± SD) | | | | | | | | | |
| Change from Baseline to 6 | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| months follow up | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) |
| Change from Baseline to 12 | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| months follow up | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) |
| Change from Baseline to 24 | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| months follow up | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) |
| Change from Baseline to 36 | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| months follow up | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) |
| Change from Baseline to 48 | XX | XX | XX | xx | XX | xx | xx | xx | xx |
| months follow up | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) |
| Change from Baseline to 60 | XX | XX | XX | xx | XX | xx | xx | xx | xx |
| months follow up | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) |
| Change from Baseline to 72 | xx | xx | XX | xx | XX | xx | xx | XX | xx |
| months follow up | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) |
| Change from Baseline to 84 | xx | xx | xx | xx | XX | xx | xx | XX | xx |
| months follow up | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) | xx.x (± xx.xx) |

Note: Only women who switched or stopped baseline prescription are considered with their first treatment episode.

Note: \*\* Mood score is calculated as described in the SAP Appendix IV.



- Table B-8.11.2 Change of Mood Score after study entry, switcher only \*, AT population, Starter
- Table B-8.11.3 Change of Mood Score after study entry, switcher only \*, AT population, Switcher
- Table B-8.11.4 Change of Mood Score after study entry, switcher only \*, AT population, Restarter
- Table B-8.11.5 Change of Mood Score after study entry, switcher only \*, AT population, Diagnosis confirmed by surgery
- Table B-8.11.6 Change of Mood Score after study entry, switcher only \*, AT population, Diagnosis based on clinical symptoms
- Table B-8.11.7 Change of Mood Score after study entry, switcher only \*, AT population, Germany
- Table B-8.11.8 Change of Mood Score after study entry, switcher only \*, AT population, Poland
- Table B-8.11.9 Change of Mood Score after study entry, switcher only \*, AT population, Hungary
- Table B-8.11.10 Change of Mood Score after study entry, switcher only \*, AT population, Switzerland
- Table B-8.11.11 Change of Mood Score after study entry, switcher only \*, AT population, Russia
- Table B-8.11.12 Change of Mood Score after study entry, switcher only \*, AT population, Ukraine



Supporting document SOP BMT 01.09 – Doc 5002.02 – Effective date 21.03.2017

### Section B-8.12 Cohort status/switch of women during follow-up

Table B-8.12.1 Cohort status/switch of women during follow-up, AT population, Complete cohort

| | DNG | OAED | | | | NAED | Allocation<br>unknown | Total | |
|---|---|---|---|---|---|---|---|---|---|
| | | GnRH-a | Danazol | All OAED | CHC | Other progestin | All NAED | | |
| Number (%) of women | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) |
| Switched or stopped EMT* | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Thereof | | | | | | | | | |
| Switch to DNG | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| of which | | | | | | | | | |
| Within 6 months | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Within 7 and 12 months | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| After 12 months | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Switch to GnRH-a | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| of which | | | | | | | | | |
| Within 6 months | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Within 7 and 12 months | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| After 12 months | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Switch to Danazol of which | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Switch to CHC of which | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Switch to Other progestins of which | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

...



Supporting document SOP BMT 01.09 – Doc 5002.02 – Effective date 21.03.2017

Switch to other EMT\*' xx (xx.x%) xx (xx.x%

of which

•••

Note: \*Only the first switch or stop of the EMT prescribed at study entry is considered.

Note: "Women switched to other NAED, unspecific treatment (Multi-use, allocation unknown) or stopped EMT use (Ex-use).

Date of analysis:

Table B-8.12.2 Cohort status/switch of women during follow-up, AT population, Starter

Table B-8.12.3 Cohort status/switch of women during follow-up, AT population, Switcher

Table B-8.12.4 Cohort status/switch of women during follow-up, AT population, Restarter

Table B-8.12.5 Cohort status/switch of women during follow-up, AT population, Diagnosis confirmed by surgery

Table B-8.12.6 Cohort status/switch of women during follow-up, AT population, Diagnosis based on clinical symptoms

Table B-8.12.7 Cohort status/switch of women during follow-up, AT population, Germany

Table B-8.12.8 Cohort status/switch of women during follow-up, AT population, Poland

Table B-8.12.9 Cohort status/switch of women during follow-up, AT population, Hungary

Table B-8.12.10 Cohort status/switch of women during follow-up, AT population, Switzerland

Table B-8.12.11 Cohort status/switch of women during follow-up, AT population, Russia

Table B-8.12.12 Cohort status/switch of women during follow-up, AT population, Ukraine



Supporting document SOP BMT 01.09 – Doc 5002.02 – Effective date 21.03.2017

### Section B-9 Summary tables of selected baseline characteristics

#### Section B-9.1 Selected baseline characteristics

Table B-9.1.1 Selected baseline characteristics, ITT population, Complete cohort

| | DNG | | OAED | OAED | | NAED | | Allocation unknown | Total |
|---|---|---|---|---|---|---|---|---|---|
| | | GnRH-a | Danazol | All OAED | CC | Other progestin | All NAED | | |
| Number (%) of women | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) |
| Age (years) | | | | | | | | | |
| Mean | xx.x | xx.x | xx.x | xx.x | XX.X | xx.x | XX.X | xx.x | xx.x |
| SD | xx.xx | xx.xx | xx.xx | XX.XX | xx.xx | XX.XX | xx.xx | xx.xx | xx.xx |
| BMI | | | | | | | | | |
| <20 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 20 to <25 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 25 to <30 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 30 to <35 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| ≥35 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Missing | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Education | | | | | | | | | |
| Lower than university entrance level | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| University entrance level | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Higher than university entrance level | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Missing | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Diagnosis classification | | | | | | | | | |
| Surgically confirmed diagnosis | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |


Supporting document SOP BMT 01.09 – Doc 5002.02 – Effective date 21.03.2017

| Clinically confirmed diagnosis | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
|---|---|---|---|---|---|---|---|---|---|
| Parity | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Gravidity | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Pain severity score | | | | | | | | | |
| Mild (0-3) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderate (4-7) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Severe (8-10) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Missing | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Pain symptoms | | | | | | | | | |
| Pelvic pain | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Pain during or after<br>sexual intercourse | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Painful periods | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Personal history of Depression | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Personal history of Anemia | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Use of Antidepressants/SSRI | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |



| Table B-9.1.2 | Selected baseline characteristics, AT population, Complete cohort |
|---|---|
| Table B-9.1.3 | Selected baseline characteristics, AT population, Starter |
| Table B-9.1.4 | Selected baseline characteristics, AT population, Switcher |
| Table B-9.1.5 | Selected baseline characteristics, AT population, Restarter |
| Table B-9.1.6 | Selected baseline characteristics, AT population, Diagnosis confirmed by surgery |
| Table B-9.1.7 | Selected baseline characteristics, AT population, Diagnosis based on clinical symptoms |
| Table B-9.1.8 | Selected baseline characteristics, AT population, Germany |
| Table B-9.1.9 | Selected baseline characteristics, AT population, Poland |
| Table B-9.1.10 | Selected baseline characteristics, AT population, Hungary |
| Table B-9.1.11 | Selected baseline characteristics, AT population, Switzerland |
| Table B-9.1.12 | Selected baseline characteristics, AT population, Russia |
| Table B-9.1.13 | Selected baseline characteristics, AT population, Ukraine |



| Section B-9.2 | Selected baseline characteristics by age categories |
|---|---|
| Table B-9.2.1 | Selected baseline characteristics, Adolescence, ITT population |
| Table B-9.2.2 | Selected baseline characteristics, Adolescence, AT population |
| Table B-9.2.3 | Selected baseline characteristics, Women <20 years, ITT population |
| Table B-9.2.4 | Selected baseline characteristics, Women <20 years, AT population |
| Table B-9.2.5 | Selected baseline characteristics Women >=20 and < 30 years, ITT population |
| Table B-9.2.6 | Selected baseline characteristics Women >=20 and < 30 years, AT population |
| Table B-9.2.7 | Selected baseline characteristics, Women >=30 and < 40 years, ITT population |
| Table B-9.2.8 | Selected baseline characteristics, Women >= 30 and < 40 years, AT population |
| Table B-9.2.9 | Selected baseline characteristics, Women >=40 years, ITT population |
| Table B-9.2.10 | Selected baseline characteristics, Women >=40 years, AT population |
| Table B-9.2.11 | Selected baseline characteristics, age-standardized, ITT population |
| Table B-9.2.12 | Selected baseline characteristics, age-standardized, AT population |



Section B-9.3 Selected baseline characteristics for women with treatment failure

Table B-9.3.1 Selected baseline characteristics for women with treatment failure, AT population, Complete cohort

| | DNG | | OAED | | | NAED | | Allocation<br>unknown | Total |
|---|---|---|---|---|---|---|---|---|---|
| | | GnRH-a | Danazol | All OAED | CC | Other progestin | All NAED | | |
| Number (%) of women | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) |
| Medication ineffective as a reason<br>for stopping or switching<br>treatment*<br>Age (years) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Mean | xx.x | xx.x | xx.x | xx.x | XX.X | xx.x | xx.x | xx.x | xx.x |
| SD | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx | XX.XX |
| Diagnosis classification | | | | | | | | | |
| Surgically confirmed diagnosis | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Clinically confirmed diagnosis | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Pain severity score | | | | | | | | | |
| Mild (0-3) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderate (4-7) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Severe (8-10) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Side effects of medication as a reason for stopping or switching treatment Age (years) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Mean | XX.X | XX.X | xx.x | xx.x | xx.x | xx.x | XX.X | xx.x | xx.x |
| SD | XX.X<br>XX.XX | XX.X<br>XX.XX | XX.XX<br>XX.XX | XX.XX<br>XX.XX | XX.X<br>XX.XX | | XX.XX<br>XX.XX | XX.X<br>XX.XX | XX.XX |
| Diagnosis classification | ***** | ***** | AA.XX | AA.AX | AX.XX | | ***** | ***** | AX.XX |
| Surgically confirmed diagnosis | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Surgically confinition diagnosis | ^^ ( ^^.^/0) | ^^ ( ^^.^/0) | ^^ ( ^^.^/0) | ^^ ( ^^.^/0) | ^^ ( ^^.7/0) | ^^ ( ^^.^/0) | ^^ ( ^^.^/0) | ^^ ( ^^.^/0) | ^^ ( ^^.7/0) |



Supporting document SOP BMT 01.09 – Doc 5002.02 – Effective date 21.03.2017

| Clinically confirmed diagnosis | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
|---|---|---|---|---|---|---|---|---|---|
| Pain severity score | | | | | | | | | |
| Mild (0-3) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderate (4-7) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Severe (8-10) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

Note: \* Only the first stop or switch from baseline prescription is considered Date of analysis:

Table B-9.3.2 Selected baseline characteristics for women with treatment failure, AT population, Starter

Table B-9.3.3 Selected baseline characteristics for women with treatment failure, AT population, Switcher

Table B-9.3.4 Selected baseline characteristics for women with treatment failure, AT population, Restarter



Section B-9.4 Selected baseline characteristics for women who switched

Table B-9.4.1 Selected baseline characteristics for women who switched, AT population

| | DNG | | OAED | | | NAED | | Allocation<br>unknown | |
|---|---|---|---|---|---|---|---|---|---|
| | | GnRH-a | Danazol | All OAED | CHC | Other progestin | All NAED | | |
| Number (%) of women | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) | xx ( 100%) |
| Switched to DNG* | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Age (years) | | | | | | | | | |
| Mean | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |
| SD | XX.XX | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx |
| Diagnosis classification | | | | | | | | | |
| Surgically confirmed diagnosis | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Clinically confirmed diagnosis | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Pain severity score | | | | | | | | | |
| Mild (0-3) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderate (4-7) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Severe (8-10) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Switched to GnRH-a* | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Age (years) | | | | | | | | | |
| Mean | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |
| SD | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx |
| Diagnosis classification | | | | | | | | | |
| Surgically confirmed diagnosis | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Clinically confirmed diagnosis | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Pain severity score | | | | | | | | | |
| Mild (0-3) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |



Supporting document SOP BMT 01.09 – Doc 5002.02 – Effective date 21.03.2017

| Moderate (4-7) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
|---|---|---|---|---|---|---|---|---|---|
| Severe (8-10) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Switched to Danazol* | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Age (years) | | | | | | | | | |
| Mean | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |
| SD | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx |
| Diagnosis classification | | | | | | | | | |
| Surgically confirmed diagnosis | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Clinically confirmed diagnosis | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Pain severity score | | | | | | | | | |
| Mild (0-3) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderate (4-7) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Severe (8-10) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Switched to CHC* | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Switched to Other progestins* | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| <br>Switched to other EMT* | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

Note: \* Only the first stop or switch from baseline prescription is considered

Date of analysis:

Table B-9.4.2 Selected baseline characteristics for women who switched, Starter

Table B-9.4.3 Selected baseline characteristics for women who switched, Switcher

Table B-9.4.4 Selected baseline characteristics for women who switched, Restarter



Supporting document SOP BMT 01.09 - Doc 5002.02 - Effective date 21.03.2017

Section C Clinical Outcome

Section C-1 Primary outcomes

Section C-1.1 Incidence rate of clinically relevant anemia

Table C-1.1.1 Incidence rate of clinically relevant anemia, ITT population, Complete cohort

| | DNG | | OAED | | | NAED | | Allocation<br>unknown | Total |
|---|---|---|---|---|---|---|---|---|---|
| | | GnRH-a | Danazol | All OAED | СНС | Other<br>progestin | All NAED | | |
| Number of women years | xx | XX | xx | XX | xx | xx | XX | xx | xx |
| Confirmed anemia | xx | xx | xx | xx | xx | xx | xx | XX | xx |
| IR* (95% CI) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |
| Thereof | | | | | | | | | |
| Treated with iron | xx | xx | xx | XX | XX | XX | XX | xx | xx |
| tablets | xx.x (xx.x–x.x) | xx.x (xx.x-x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |
| Treated with iron | xx | xx | xx | xx | xx | XX | xx | xx | xx |
| infusions/injections | xx.x (xx.x–x.x) | xx.x (xx.x-x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x-x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x-x.x) |
| Treated with blood | XX | xx | xx | xx | XX | XX | xx | XX | xx |
| transfusions | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) |

Note: \* Incidence rate is shown per 10<sup>4</sup> women years.



| Table C-1.1.2 | Incidence rate of newly diagnosed or reoccurrence of anemia, AT population, Complete cohort |
|---|---|
| Table C-1.1.3 | Incidence rate of newly diagnosed or reoccurrence of anemia, AT population, Starter |
| Table C-1.1.4 | Incidence rate of newly diagnosed or reoccurrence of anemia, AT population, Switcher |
| Table C-1.1.5 | Incidence rate of newly diagnosed or reoccurrence of anemia, AT population, Restarter |
| Table C-1.1.6 | Incidence rate of newly diagnosed or reoccurrence of anemia, AT population, Diagnosis confirmed by surgery |
| Table C-1.1.7 | Incidence rate of newly diagnosed or reoccurrence of anemia, AT population, Diagnosis based on clinical symptoms |
| Table C-1.1.8 | Incidence rate of newly diagnosed or reoccurrence of anemia, AT population, Germany |
| Table C-1.1.9 | Incidence rate of newly diagnosed or reoccurrence of anemia, AT population, Poland |
| Table C-1.1.10 | Incidence rate of newly diagnosed or reoccurrence of anemia, AT population, Hungary |
| Table C-1.1.11 | Incidence rate of newly diagnosed or reoccurrence of anemia, AT population, Switzerland |
| Table C-1.1.12 | Incidence rate of newly diagnosed or reoccurrence of anemia, AT population, Russia |
| Table C-1.1.13 | Incidence rate of newly diagnosed or reoccurrence of anemia, AT population, Ukraine |

Supporting document SOP BMT 01.09 – Doc 5002.02 – Effective date 21.03.2017

### Section C-1.2 Incidence rate of new depression or worsening of existing depression

Table C-1.2.1 Incidence rate of new depression or worsening of existing depression, ITT population, Complete cohort

| DI | NG | | OAED | | | NAED | | Allocation<br>unknown | Total |
|---|---|---|---|---|---|---|---|---|---|
| | | GnRH-a | Danazol | All OAED | CC | Other<br>progestin | All NAED | | |
| of women years | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| ed depression | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| (CI) XX.X (X | xx.x–x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |
| ed by psychiatrist xx.x (x | xx.x–x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x–x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) |
| | xx | XX | xx | xx | xx | XX | xx | xx | XX |
| al admission xx.x (x | xx.x–x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x–x.x) | xx.x (xx.x-x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) |
| | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| e attempt xx.x (x | xx.x–x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x–x.x) | xx.x (xx.x-x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) |
| | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| nitted suicide xx.x (x | xx.x–x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x–x.x) | xx.x (xx.x-x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) |
| nal history of | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| ssion xx.x (x | xx.x–x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x–x.x) | xx.x (xx.x-x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) |
| history of | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| ssion xx.x (x | xx.x–x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |

Note: \* Incidence rate is shown per 10<sup>4</sup> women years.



| Table C-1.2.2 | Incidence rate of new depression or worsening of existing depression, AT population, Complete cohort |
|---|---|
| Table C-1.2.3 | Incidence rate of new depression or worsening of existing depression, AT population, Starter |
| Table C-1.2.4 | Incidence rate of new depression or worsening of existing depression, AT population, Switcher |
| Table C-1.2.5 | Incidence rate of new depression or worsening of existing depression, AT population, Restarter |
| Table C-1.2.6 | Incidence rate of new depression or worsening of existing depression, AT population, Diagnosis confirmed by surgery |
| Table C-1.2.7 | Incidence rate of new depression or worsening of existing depression, AT population, Diagnosis based on clinical symptoms |
| Table C-1.2.8 | Incidence rate of new depression or worsening of existing depression, AT population, Germany |
| Table C-1.2.9 | Incidence rate of new depression or worsening of existing depression, AT population, Poland |
| Table C-1.2.10 | Incidence rate of new depression or worsening of existing depression, AT population, Hungary |
| Table C-1.2.11 | Incidence rate of new depression or worsening of existing depression, AT population, Switzerland |
| Table C-1.2.12 | Incidence rate of new depression or worsening of existing depression, AT population, Russia |
| Table C-1.2.13 | Incidence rate of new depression or worsening of existing depression, AT population, Ukraine |



Supporting document SOP BMT 01.09 - Doc 5002.02 - Effective date 21.03.2017

#### Section C-1.3 Incidence proportions of treatment discontinuation due to treatment failure

Table C-1.3.1 Incidence proportions of treatment discontinuation due to treatment failure, AT population, Complete cohort

| | DNG | | OAED | | | NAED | | Allocation<br>unknown | Total |
|---|---|---|---|---|---|---|---|---|---|
| | | GnRH-a | Danazol | All OAED | СНС | Other<br>progestin | All NAED | | |
| Number of treatment starts | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| Treatment failure | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| <b>IP* (95% CI)</b><br>Thereof** | xx.x (xx.x–x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x-x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) |
| Medication ineffective | xx<br>xx.x (xx.x–x.x) | | | xx<br>xx.x (xx.x–x.x) | xx<br>xx.x (xx.x-x.x) | | xx<br>xx.x (xx.x-x.x) | | |
| Side effects Thereof*** | xx<br>xx.x (xx.x-x.x) | | xx<br>xx.x (xx.x–x.x) | | xx<br>xx.x (xx.x–x.x) | | | xx<br>xx.x (xx.x-x.x) | |
| Depression / Depressive mood | xx<br>xx.x (xx.x-x.x) | | xx<br>xx.x (xx.x-x.x) | xx<br>xx.x (xx.x–x.x) | xx<br>xx.x (xx.x–x.x) | | | xx<br>xx.x (xx.x–x.x) | |
| <category>&gt;</category> | xx<br>xx.x (xx.x–x.x) | | xx<br>xx.x (xx.x-x.x) | xx<br>xx.x (xx.x–x.x) | xx<br>xx.x (xx.x–x.x) | | | xx<br>xx.x (xx.x–x.x) | |

Note: \* Incidence proportion is shown per 10<sup>2</sup> treatment starts, including incident exposure at study entry, switches between exposure groups and/or restarts within exposure groups.

Note: \*\* Multiple answers possible.

Note: "Multiple answers possible. Only side effect categories with a proportion > 1% were displayed



| Table C-1.3.2 | Incidence proportions of treatment discontinuation due to treatment failure, AT population, Starter |
|---|---|
| Table C-1.3.3 | Incidence proportions of treatment discontinuation due to treatment failure, AT population, Switcher |
| Table C-1.3.4 | Incidence proportions of treatment discontinuation due to treatment failure, AT population, Restarter |
| Table C-1.3.5 | Incidence proportions of treatment discontinuation due to treatment failure, AT population, Diagnosis confirmed by surgery |
| Table C-1.3.6 | Incidence proportions of treatment discontinuation due to treatment failure, AT population, Diagnosis based on clinical symptoms |
| Table C-1.3.7 | Incidence proportions of treatment discontinuation due to treatment failure, AT population, Germany |
| Table C-1.3.8 | Incidence proportions of treatment discontinuation due to treatment failure, AT population, Poland |
| Table C-1.3.9 | Incidence proportions of treatment discontinuation due to treatment failure, AT population, Hungary |
| Table C-1.3.10 | Incidence proportions of treatment discontinuation due to treatment failure, AT population, Switzerland |
| Table C-1.3.11 | Incidence proportions of treatment discontinuation due to treatment failure, AT population, Russia |
| Table C-1.3.12 | Incidence proportions of treatment discontinuation due to treatment failure, AT population, Ukraine |



Supporting document SOP BMT 01.09 - Doc 5002.02 - Effective date 21.03.2017

#### Section C-2 Secondary outcomes

#### Section C-2.1 Incidence proportions of treatment discontinuation unrelated to treatment failure

Table C-2.1.1 Incidence proportions of treatment discontinuation unrelated to treatment failure, AT population, Complete cohort

| | DNG | | OAED | | | NAED | | Allocation<br>unknown | Total |
|---|---|---|---|---|---|---|---|---|---|
| | | GnRH-a | Danazol | All OAED | СНС | Other<br>progestin | All NAED | | |
| Number of treatment starts | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| Treatment | | | | | | | | | |
| discontinuation | XX | XX | XX | XX | XX | xx | xx | xx | xx |
| IP* (95% CI) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x–x.x) | xx.x (xx.x-x.x) |
| Thereof** | | | | | | | | | |
| Trying to become | XX | xx | xx | XX | xx | xx | XX | xx | xx |
| pregnant | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x–x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |
| Treatment duration | xx | xx | xx | XX | xx | xx | XX | xx | xx |
| finished | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x–x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |
| Other | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |
| Thereof** | | | | | | | | | |
| Physician's advice | xx | xx | xx | xx | XX | xx | xx | xx | xx |
| | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |
| < <category>&gt;</category> | xx | xx | xx | xx | XX | xx | xx | xx | xx |
| | xx.x (xx.x–x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x–x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |

Note: 'Incidence proportion is shown per 102 treatment starts, including incident exposure at study entry, switches between exposure groups and/or restarts within exposure groups.

Note: \*\*Multiple answers possible.



| Table C-2.1.2 | Incidence proportions of treatment discontinuation unrelated to treatment failure, AT population, Starter |
|---|---|
| Table C-2.1.3 | Incidence proportions of treatment discontinuation unrelated to treatment failure, AT population, Switcher |
| Table C-2.1.4 | Incidence proportions of treatment discontinuation unrelated to treatment failure, AT population, Restarter |
| Table C-2.1.5 | Incidence proportions of treatment discontinuation unrelated to treatment failure, AT population, Diagnosis confirmed by surgery |
| Table C-2.1.6 | Incidence proportions of treatment discontinuation unrelated to treatment failure, AT population, Diagnosis based on clinical symptoms |
| Table C-2.1.7 | Incidence proportions of treatment discontinuation unrelated to treatment failure, AT population, Germany |
| Table C-2.1.8 | Incidence proportions of treatment discontinuation unrelated to treatment failure, AT population, Poland |
| Table C-2.1.9 | Incidence proportions of treatment discontinuation unrelated to treatment failure, AT population, Hungary |
| Table C-2.1.10 | Incidence proportions of treatment discontinuation unrelated to treatment failure, AT population, Switzerland |
| Table C-2.1.11 | Incidence proportions of treatment discontinuation unrelated to treatment failure, AT population, Russia |
| Table C-2.1.12 | Incidence proportions of treatment discontinuation unrelated to treatment failure, AT population, Ukraine |

Supporting document SOP BMT 01.09 – Doc 5002.02 – Effective date 21.03.2017

### Section C-2.2 Incidence rate of clinically relevant anemia for adolescence

Table C-2.2.1 Incidence rate of clinically relevant anemia for adolescence\*, AT population, Complete cohort

| | DNG | | OAED | | NAED | | | Ex-use | Allocation<br>unknown | Total |
|---|---|---|---|---|---|---|---|---|---|---|
| | | GnRH-a | Danazol | All OAED | СНС | Other<br>progestin | All NAED | | | |
| Number of women years | xx | xx | xx | xx | xx | XX | xx | xx | xx | xx |
| Confirmed anemia | xx | xx | XX | xx | XX | xx | xx | xx | xx | xx |
| IR** (95% CI) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |
| Thereof | | | | | | | | | | |
| Treated with iron | xx | xx | xx | xx | XX | xx | XX | xx | xx | xx |
| tablets | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x–x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) |
| Treated with iron | xx | xx | xx | xx | xx | XX | XX | XX | xx | xx |
| infusions/injections | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |
| Treated with blood | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| transfusions | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x–x.x) |

Note: \* Adolescent at study entry.

Note: \*\* Incidence rate is shown per 10<sup>4</sup> women years.



| Table C-2.2.2 | Incidence rate of clinically relevant anemia for adolescence*, AT population, Starter |
|---|---|
| Table C-2.2.3 | Incidence rate of clinically relevant anemia for adolescence*, AT population, Switcher |
| Table C-2.2.4 | Incidence rate of clinically relevant anemia for adolescence*, AT population, Restarter |
| Table C-2.2.5 | Incidence rate of clinically relevant anemia for adolescence*, AT population, Diagnosis confirmed by surgery |
| Table C-2.2.6 | $Incidence\ rate\ of\ clinically\ relevant\ anemia\ for\ adolescence^*,\ AT\ population,\ Diagnosis\ based\ on\ clinical\ symptoms$ |
| Table C-2.2.7 | Incidence rate of clinically relevant of anemia for adolescence*, AT population, Germany |
| Table C-2.2.8 | Incidence rate of clinically relevant of anemia for adolescence*, AT population, Poland |
| Table C-2.2.9 | Incidence rate of clinically relevant anemia for adolescence*, AT population, Hungary |
| Table C-2.2.10 | Incidence rate of clinically relevant anemia for adolescence*, AT population, Switzerland |
| Table C-2.2.11 | Incidence rate of clinically relevant anemia for adolescence*, AT population, Russia |
| Table C-2.2.12 | Incidence rate of clinically relevant anemia for adolescence*, AT population, Ukraine |

Supporting document SOP BMT 01.09 – Doc 5002.02 – Effective date 21.03.2017

### Section C-2.3 Incidence rate of new depression or worsening of existing depression for adolescence

Table C-2.3.1 Incidence rate of new depression or worsening of existing depression for adolescence\*, AT population, Complete cohort

| | DNG | | OAED | | | NAED | | | Allocation<br>unknown | Total |
|---|---|---|---|---|---|---|---|---|---|---|
| | | GnRH-a | Danazol | All OAED | СНС | Other<br>progestin | All NAED | | | |
| Number of women years | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| Confirmed depression | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| IR** (95% CI)<br>Thereof | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x–x.x) | xx.x (xx.x-x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x-x.x) |
| Treated by psychiatrist | XX | xx | xx | XX | XX | xx | XX | xx | xx | xx |
| | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x–x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |
| Hospital admission | xx | xx | xx | xx | xx | xx | XX | xx | xx | xx |
| | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) |
| Suicide attempt | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| | xx.x (xx.x-x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) |
| Committed suicide | xx | xx | xx | xx | xx | xx | XX | xx | xx | xx |
| | xx.x (xx.x-x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) |
| Personal history | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| of depression | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x–x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |
| Family history | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| of depression | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x–x.x) |

Note: \* Adolescent at study entry.

Note: \*\* Incidence rate is shown per 10<sup>4</sup> women years.



| Table C-2.3.2 | Incidence rate of new depression or worsening of existing depression for adolescence*, AT population, Starter |
|---|---|
| Table C-2.3.3 | Incidence rate of new depression or worsening of existing depression for adolescence*, AT population, Switcher |
| Table C-2.3.4 | Incidence rate of new depression or worsening of existing depression for adolescence*, AT population, Restarter |
| Table C-2.3.5 | Incidence rate of new depression or worsening of existing depression for adolescence*, AT population, Diagnosis confirmed by surgery |
| Table C-2.3.6 | Incidence rate of new depression or worsening of existing depression for adolescence*, AT population, Diagnosis based on clinical symptoms |
| Table C-2.3.7 | Incidence rate of new depression or worsening of existing depression for adolescence*, AT population, Germany |
| Table C-2.3.8 | Incidence rate of new depression or worsening of existing depression for adolescence*, AT population, Poland |
| Table C-2.3.9 | Incidence rate of new depression or worsening of existing depression for adolescence*, AT population, Hungary |
| Table C-2.3.10 | Incidence rate of new depression or worsening of existing depression for adolescence*, AT population, Switzerland |
| Table C-2.3.11 | Incidence rate of new depression or worsening of existing depression for adolescence*, AT population, Russia |
| Table C-2.3.12 | Incidence rate of new depression or worsening of existing depression for adolescence*, AT population, Ukraine |

Supporting document SOP BMT 01.09 - Doc 5002.02 - Effective date 21.03.2017

#### Section C-2.4 Incidence proportions of treatment discontinuation for adolescence

Table C-2.4.1 Incidence proportions of treatment discontinuation for adolescence\*, AT population, Complete cohort

| | DNG | | OAED | | | NAED | Allocation<br>unknown | Total | |
|---|---|---|---|---|---|---|---|---|---|
| | • | GnRH-a | Danazol | All OAED | СНС | Other<br>progestin | All NAED | | |
| Number of treatment starts | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| Treatment failure | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| <b>IP** (95% CI)</b><br>Thereof*** | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x-x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x-x.x) |
| Medication ineffective | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| | xx.x (xx.x–x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x–x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x–x.x) | xx.x (xx.x-x.x) |
| Side effects | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| | xx.x (xx.x–x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x–x.x) | xx.x (xx.x-x.x) |

Note: \* Adolescent at study entry

Note: \*\* Incidence proportion is shown per 102 treatment starts, including incident exposure at study entry, switches between exposure groups and/or restarts within exposure groups.

Note: \*\*\* Multiple answers possible.



| Table C-2.4.2 | Incidence proportions of treatment discontinuation for adolescence*, AT population, Starter |
|---|---|
| Table C-2.4.3 | Incidence proportions of treatment discontinuation for adolescence*, AT population, Switcher |
| Table C-2.4.4 | Incidence proportions of treatment discontinuation for adolescence*, AT population, Restarter |
| Table C-2.4.5 | Incidence proportions of treatment discontinuation for adolescence*, AT population, Diagnosis confirmed by surgery |
| Table C-2.4.6 | Incidence proportions of treatment discontinuation for adolescence*, AT population, Diagnosis based on clinical symptoms |
| Table C-2.4.7 | Incidence proportions of treatment discontinuation for adolescence*, AT population, Germany |
| Table C-2.4.8 | Incidence proportions of treatment discontinuation for adolescence*, AT population, Poland |
| Table C-2.4.9 | Incidence proportions of treatment discontinuation for adolescence*, AT population, Hungary |
| Table C-2.4.10 | Incidence proportions of treatment discontinuation for adolescence*, AT population, Switzerland |
| Table C-2.4.11 | Incidence proportions of treatment discontinuation for adolescence*, AT population, Russia |
| Table C-2.4.12 | Incidence proportions of treatment discontinuation for adolescence*, AT population, Ukraine |



Table C-2.6.8

### INAS-VIPOS Statistical Analysis Plan V02-00

Supporting document SOP BMT 01.09 - Doc 5002.02 - Effective date 21.03.2017

| Section C-2.5 | Incidence rate of clinically relevant anemia for long-term use, AT population, Complete cohort |
|---|---|
| Table C-2.5.1 | Incidence rate of clinically relevant anemia for long-term use, AT population, Starter |
| Table C-2.5.2 | Incidence rate of clinically relevant anemia for long-term use, AT population, Switcher |
| Table C-2.5.3 | Incidence rate of clinically relevant anemia for long-term use, AT population, Restarter |
| Table C-2.5.4 | Incidence rate of clinically relevant anemia for long-term use, AT population, Diagnosis confirmed by surgery |
| Table C-2.5.5 | Incidence rate of clinically relevant anemia for long-term use, AT population, Diagnosis based on clinical symptoms |
| Table C-2.5.6 | Incidence rate of clinically relevant anemia for long-term use, AT population, Germany |
| Table C-2.5.7 | Incidence rate of clinically relevant anemia for long-term use, AT population, Poland |
| Table C-2.5.8 | Incidence rate of clinically relevant anemia for long-term use, AT population, Hungary |
| Table C-2.5.9 | Incidence rate of clinically relevant anemia for long-term use, AT population, Switzerland |
| Table C-2.5.10 | Incidence rate of clinically relevant anemia for long-term use, AT population, Russia |
| Table C-2.5.11 | Incidence rate of clinically relevant anemia for long-term use, AT population, Ukraine |
| Section C-2.6 | Incidence rate of new depression or worsening of existing depression for long-term use |
| Table C-2.6.1 | Incidence rate of new depression or worsening of existing depression for long-term use, AT population, Complete cohort |
| Table C-2.6.2 | Incidence rate of new depression or worsening of existing depression for long-term use, AT population, Starter |
| Table C-2.6.3 | Incidence rate of new depression or worsening of existing depression for long-term use, AT population, Switcher |
| Table C-2.6.4 | Incidence rate of new depression or worsening of existing depression for long-term use, AT population, Restarter |
| Table C-2.6.5 | Incidence rate of new depression or worsening of existing depression for long-term use, AT population, Diagnosis confirmed by surgery |
| Table C-2.6.6 | Incidence rate of new depression or worsening of existing depression for long-term use, AT population, Diagnosis based on clinical symptoms |
| Table C-2.6.7 | Incidence rate of new depression or worsening of existing depression for long-term use, AT population, Germany |

Incidence rate of new depression or worsening of existing depression for long-term use, AT population, Poland

Table C-2.6.9 Incidence rate of new depression or worsening of existing depression for long-term use, AT population, Hungary



| Table C-2.6.10 Incidence rate of new depression or worsening of existing depression for long-term use, AT population, Switzerland |
|---|
| Table C-2.6.11 Incidence rate of new depression or worsening of existing depression for long-term use, AT population, Russia |
| Table C-2.6.12 Incidence rate of new depression or worsening of existing depression for long-term use, AT population, Ukraine |
| Section C-2.7 Incidence proportions of treatment discontinuation for long-term use |
| Table C-2.7.1 Incidence proportions of treatment discontinuation for long-term use, AT population, Complete cohort |
| Table C-2.7.2 Incidence proportions of treatment discontinuation for long-term use, AT population, Starter |
| Table C-2.7.3 Incidence proportions of treatment discontinuation for long-term use, AT population, Switcher |
| Table C-2.7.4 Incidence proportions of treatment discontinuation for long-term use, AT population, Restarter |
| Table C-2.7.5 Incidence proportions of treatment discontinuation for long-term use, AT population, Diagnosis confirmed by surgery |
| Table C-2.7.6 Incidence proportions of treatment discontinuation for long-term use, AT population, Diagnosis based on clinical symptoms |
| Table C-2.7.7 Incidence proportions of treatment discontinuation for long-term use, AT population, Germany |
| Table C-2.7.8 Incidence proportions of treatment discontinuation for long-term use, AT population, Poland |
| Table C-2.7.9 Incidence proportions of treatment discontinuation for long-term use, AT population, Hungary |
| Table C-2.7.10 Incidence proportions of treatment discontinuation for long-term use, AT population, Switzerland |
| Table C-2.7.11 Incidence proportions of treatment discontinuation for long-term use, AT population, Russia |
| Table C-2.7.12 Incidence proportions of treatment discontinuation for long-term use, AT population, Ukraine |



Supporting document SOP BMT 01.09 – Doc 5002.02 – Effective date 21.03.2017

### Section C-3 Other safety outcomes

#### Section C-3.1 Incidence rate of confirmed thromboembolic events

Table C-3.1.1 Incidence rate of confirmed thromboembolic events, AT population, Complete cohort

| | DNG | | OAED | | | NAED | | | Allocation<br>unknown | Total |
|---|---|---|---|---|---|---|---|---|---|---|
| | •••• | GnRH-a | Danazol | All OAED | СНС | Other<br>progestin | All NAED | | | |
| Number of women years | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| ALL VTE & ATE | xx | xx | xx | xx | xx | XX | xx | xx | xx | xx |
| IR* (95% CI) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |
| Thereof | | | | | | | | | | |
| All VTE | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |
| Thereof | | | | | | | | | | |
| PE | xx | xx | xx | xx | XX | xx | xx | xx | xx | xx |
| | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |
| ALL ATE (TIAs included) | XX | xx | xx | XX | xx | XX | XX | xx | XX | xx |
| | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |
| Thereof | | | | | | | | | | |
| AMI | | | | | | | | | | |
| Ischemic stroke | | | | | | | | | | |
| TIA | | | | | | | | | | |
| ALL ATE (TIAs excluded) | | | | | | | | | | |

Note: \* Incidence rate is shown per 10<sup>4</sup> women years.



| Table C-3.1.2 | Incidence rate of confirmed thromboembolic events, AT population, Starter |
|---|---|
| Table C-3.1.3 | Incidence rate of confirmed thromboembolic events, AT population, Switcher |
| Table C-3.1.4 | Incidence rate of confirmed thromboembolic events, AT population, Restarter |
| Table C-3.1.5 | Incidence rate of confirmed thromboembolic events, AT population, Diagnosis confirmed by surgery |
| Table C-3.1.6 | Incidence rate of confirmed thromboembolic events, AT population, Diagnosis based on clinical symptoms |
| Table C-3.1.7 | Incidence rate of confirmed thromboembolic events, AT population, Germany |
| Table C-3.1.8 | Incidence rate of confirmed thromboembolic events, AT population, Poland |
| Table C-3.1.9 | Incidence rate of confirmed thromboembolic events, AT population, Hungary |
| Table C-3.1.10 | Incidence rate of confirmed thromboembolic events, AT population, Switzerland |
| Table C-3.1.11 | Incidence rate of confirmed thromboembolic events, AT population, Russia |
| Table C-3.1.12 | Incidence rate of confirmed thromboembolic events, AT population, Ukraine |



Supporting document SOP BMT 01.09 – Doc 5002.02 – Effective date 21.03.2017

### Section C-3.2 Incidence rate of fatal cases (all deaths)

Table C-3.2.1 Incidence rate of fatal cases (all deaths), AT population, Complete cohort

| | DNG | | OAED | | NAED | | Ex-use | Allocation<br>unknown | Total | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | GnRH-a | Danazol | All OAED | СНС | Other<br>progestin | All NAED | | | |
| Number of women years | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| All deaths IR* (95% CI) | xx<br>xx.x (xx.x–x.x) | xx<br>xx.x (xx.x–x.x) | xx<br>xx.x (xx.x–x.x) | xx<br>xx.x (xx.x–x.x) | xx<br>xx.x (xx.x–x.x) | xx<br>xx.x (xx.x–x.x) | xx<br>xx.x (xx.x–x.x) | xx<br>xx.x (xx.x–x.x) | xx<br>xx.x (xx.x–x.x) | xx<br>xx.x (xx.x–x.x) |
| Reason << Category >> | xx<br>xx.x (xx.x–x.x) | xx<br>xx.x (xx.x–x.x) | | xx<br>xx.x (xx.x–x.x) | xx<br>xx.x (xx.x–x.x) | xx<br>xx.x (xx.x–x.x) | xx<br>xx.x (xx.x-x.x) | xx<br>xx.x (xx.x–x.x) | xx<br>xx.x (xx.x–x.x) | xx<br>xx.x (xx.x–x.x) |

Note: \* Incidence rate is shown per 10<sup>4</sup> women years.



| Table C-3.2.2 | Incidence rate of fatal cases (all deaths), AT population, Starter |
|---|---|
| Table C-3.2.3 | Incidence rate of fatal cases (all deaths), AT population, Switcher |
| Table C-3.2.4 | Incidence rate of fatal cases (all deaths), AT population, Restarter |
| Table C-3.2.5 | Incidence rate of fatal cases (all deaths), AT population, Diagnosis confirmed by surgery |
| Table C-3.2.6 | Incidence rate of fatal cases (all deaths), AT population, Diagnosis based on clinical symptoms |
| Table C-3.2.7 | Incidence rate of fatal cases (all deaths), AT population, Germany |
| Table C-3.2.8 | Incidence rate of fatal cases (all deaths), AT population, Poland |
| Table C-3.2.9 | Incidence rate of fatal cases (all deaths), AT population, Hungary |
| Table C-3.2.10 | Incidence rate of fatal cases (all deaths), AT population, Switzerland |
| Table C-3.2.11 | Incidence rate of fatal cases (all deaths), AT population, Russia |
| Table C-3.2.12 | Incidence rate of fatal cases (all deaths), AT population, Ukraine |



Supporting document SOP BMT 01.09 – Doc 5002.02 – Effective date 21.03.2017

### Section C-3.3 Incidence rate of serious adverse events by organ system

Table C-3.3.1 Incidence rate of serious adverse events by organ system, AT population, Complete cohort

| | DNG | | OAED | | NAED | | Ex-use | Allocation<br>unknown | Total | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | GnRH-a | Danazol | All OAED | СНС | Other<br>progestin | All NAED | | | |
| Number of women years | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| Serious adverse events* | xx | xx | xx | xx | xx | xx | XX | xx | xx | xx |
| <b>IR** (95% CI)</b><br>Thereof*** | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x–x.x) |
| Infectious diseases | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |
| Neoplasms, malignant | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |
| Neoplasms, benign | xx | XX | XX | XX | XX | xx | XX | xx | xx | xx |
| | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |
| Blood | xx | xx | xx | XX | XX | xx | XX | xx | xx | xx |
| and blood-forming organs | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) |
| Endocrine diseases | XX | xx | XX | xx | XX | xx | XX | xx | XX | xx |
| | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |
| Mental and | xx | xx | xx | XX | XX | xx | XX | xx | xx | xx |
| behavioral disorders | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |
| Disease of the nervous system | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |
| Eye | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |
| Ear | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |



Supporting document SOP BMT 01.09 – Doc 5002.02 – Effective date 21.03.2017

| Cardiovascular system | xx | xx | xx | xx | xx | XX | xx | xx | xx | XX |
|---|---|---|---|---|---|---|---|---|---|---|
| caratovascatar system | | | | | xx.x (xx.x–x.x) | | | | | |
| Respiratory system | XX | | XX (XX.X X.X) | XX | XX | XX (XX.X X.X) | XX (XX.X X.X) | XX | XX (XX.X X.X) | XX (XX.X X.X) |
| Respiratory system | | | | | | | | | | |
| | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) |
| Digestive system | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |
| Skin | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |
| Musculoskeletal | xx | xx | xx | xx | XX | xx | xx | xx | xx | xx |
| system and connective | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |
| tissue | | | | | | | | | | |
| tissac | | | | | | | | | | |
| Genitourinary system | XX | XX | xx | xx | xx | xx | XX | xx | xx | xx |
| | | | | | xx<br>xx.x (xx.x–x.x) | | | | | |
| | | xx.x (xx.x-x.x) | | | | xx.x (xx.x-x.x) | | | | |
| Genitourinary system | xx.x (xx.x-x.x)<br>xx | xx.x (xx.x-x.x)<br>xx | xx.x (xx.x-x.x)<br>xx | xx.x (xx.x–x.x)<br>xx | xx.x (xx.x-x.x) | xx.x (xx.x–x.x)<br>xx | xx.x (xx.x–x.x)<br>xx | xx.x (xx.x-x.x)<br>xx | xx.x (xx.x–x.x)<br>xx | xx.x (xx.x–x.x)<br>xx |
| Genitourinary system Pregnancy, delivery | xx.x (xx.x-x.x)<br>xx | xx.x (xx.x-x.x)<br>xx<br>xx.x (xx.x-x.x) | xx.x (xx.x-x.x)<br>xx | xx.x (xx.x–x.x)<br>xx | xx.x (xx.x–x.x)<br>xx | xx.x (xx.x-x.x)<br>xx<br>xx.x (xx.x-x.x) | xx.x (xx.x–x.x)<br>xx | xx.x (xx.x-x.x)<br>xx | xx.x (xx.x–x.x)<br>xx | xx.x (xx.x–x.x)<br>xx |
| Genitourinary system Pregnancy, delivery and puerperium* | xx.x (xx.x-x.x)<br>xx<br>xx.x (xx.x-x.x)<br>xx | xx.x (xx.x-x.x)<br>xx<br>xx.x (xx.x-x.x)<br>xx | xx.x (xx.x-x.x)<br>xx<br>xx.x (xx.x-x.x)<br>xx | xx.x (xx.x-x.x)<br>xx<br>xx.x (xx.x-x.x)<br>xx | xx.x (xx.x–x.x)<br>xx<br>xx.x (xx.x–x.x) | xx.x (xx.x-x.x)<br>xx<br>xx.x (xx.x-x.x)<br>xx | xx.x (xx.x-x.x)<br>xx<br>xx.x (xx.x-x.x)<br>xx | xx.x (xx.x-x.x)<br>xx<br>xx.x (xx.x-x.x)<br>xx | xx.x (xx.x-x.x)<br>xx<br>xx.x (xx.x-x.x)<br>xx | xx.x (xx.x-x.x)<br>xx<br>xx.x (xx.x-x.x)<br>xx |
| Genitourinary system Pregnancy, delivery and puerperium* Malformations, | xx.x (xx.x-x.x)<br>xx<br>xx.x (xx.x-x.x)<br>xx | xx.x (xx.x-x.x)<br>xx<br>xx.x (xx.x-x.x)<br>xx | xx.x (xx.x-x.x)<br>xx<br>xx.x (xx.x-x.x)<br>xx | xx.x (xx.x-x.x)<br>xx<br>xx.x (xx.x-x.x)<br>xx | xx.x (xx.x-x.x)<br>xx<br>xx.x (xx.x-x.x)<br>xx | xx.x (xx.x-x.x)<br>xx<br>xx.x (xx.x-x.x)<br>xx | xx.x (xx.x-x.x)<br>xx<br>xx.x (xx.x-x.x)<br>xx | xx.x (xx.x-x.x)<br>xx<br>xx.x (xx.x-x.x)<br>xx | xx.x (xx.x-x.x)<br>xx<br>xx.x (xx.x-x.x)<br>xx | xx.x (xx.x-x.x)<br>xx<br>xx.x (xx.x-x.x)<br>xx |
| Genitourinary system Pregnancy, delivery and puerperium* Malformations, deformations and | xx.x (xx.x-x.x)<br>xx<br>xx.x (xx.x-x.x)<br>xx | xx.x (xx.x-x.x)<br>xx<br>xx.x (xx.x-x.x)<br>xx | xx.x (xx.x-x.x)<br>xx<br>xx.x (xx.x-x.x)<br>xx | xx.x (xx.x-x.x)<br>xx<br>xx.x (xx.x-x.x)<br>xx | xx.x (xx.x-x.x)<br>xx<br>xx.x (xx.x-x.x)<br>xx | xx.x (xx.x-x.x)<br>xx<br>xx.x (xx.x-x.x)<br>xx | xx.x (xx.x-x.x)<br>xx<br>xx.x (xx.x-x.x)<br>xx | xx.x (xx.x-x.x)<br>xx<br>xx.x (xx.x-x.x)<br>xx | xx.x (xx.x-x.x)<br>xx<br>xx.x (xx.x-x.x)<br>xx | xx.x (xx.x-x.x)<br>xx<br>xx.x (xx.x-x.x)<br>xx |
| Genitourinary system Pregnancy, delivery and puerperium* Malformations, deformations and chromosomal | xx.x (xx.x-x.x)<br>xx<br>xx.x (xx.x-x.x)<br>xx | xx.x (xx.x-x.x)<br>xx<br>xx.x (xx.x-x.x)<br>xx<br>xx.x (xx.x-x.x) | xx.x (xx.x-x.x)<br>xx<br>xx.x (xx.x-x.x)<br>xx<br>xx.x (xx.x-x.x) | xx.x (xx.x-x.x)<br>xx<br>xx.x (xx.x-x.x)<br>xx | xx.x (xx.x-x.x)<br>xx<br>xx.x (xx.x-x.x)<br>xx | xx.x (xx.x-x.x)<br>xx<br>xx.x (xx.x-x.x)<br>xx<br>xx.x (xx.x-x.x) | xx.x (xx.x-x.x)<br>xx<br>xx.x (xx.x-x.x)<br>xx | xx.x (xx.x-x.x)<br>xx<br>xx.x (xx.x-x.x)<br>xx | xx.x (xx.x-x.x)<br>xx<br>xx.x (xx.x-x.x)<br>xx<br>xx.x (xx.x-x.x) | xx.x (xx.x-x.x)<br>xx<br>xx.x (xx.x-x.x)<br>xx<br>xx.x (xx.x-x.x) |

Note: \* SAEs, which occurred within 3 months after stop of EMT, were attributed to the last EMT used by the women. Therefore, pregnancy-related SAEs in XXX cohorts does not necessarily reflect unwanted pregnancies during EMT use.

Note: \*\* Incidence rate is shown per 104 women years.

Note: \*\*\* Women may appear in more than one category. ICD10 Codes Version 2009.



| Table C-3.3.2 | Incidence rate of serious adverse events by organ system, AT population, Starter |
|---|---|
| Table C-3.3.3 | Incidence rate of serious adverse events by organ system, AT population, Switcher |
| Table C-3.3.4 | Incidence rate of serious adverse events by organ system, AT population, Restarter |
| Table C-3.3.5 | Incidence rate of serious adverse events by organ system, AT population, Diagnosis confirmed by surgery |
| Table C-3.3.6 | Incidence rate of serious adverse events by organ system, AT population, Diagnosis based on clinical symptoms |
| Table C-3.3.7 | Incidence rate of serious adverse events by organ system, AT population, Germany |
| Table C-3.3.8 | Incidence rate of serious adverse events by organ system, AT population, Poland |
| Table C-3.3.9 | Incidence rate of serious adverse events by organ system, AT population, Hungary |
| Table C-3.3.10 | Incidence rate of serious adverse events by organ system, AT population, Switzerland |
| Table C-3.3.11 | Incidence rate of serious adverse events by organ system, AT population, Russia |
| Table C-3.3.12 | Incidence rate of serious adverse events by organ system, AT population, Ukraine |



Supporting document SOP BMT 01.09 – Doc 5002.02 – Effective date 21.03.2017

### Section C-3.4 Incidence rate of serious adverse events by organ system for long-term use

Table C-3.4.1 Incidence rate of serious adverse events by organ system for long-term use, AT population, Complete cohort

| | DNG | | OAED | | | NAED | | Ex-use | Allocation<br>unknown | Total |
|---|---|---|---|---|---|---|---|---|---|---|
| | | GnRH-a | Danazol | All OAED | СНС | Other<br>progestin | All NAED | | | |
| Number of women years* | XX | XX | XX | xx | xx | XX | xx | xx | xx | xx |
| Serious adverse events** | xx | xx | xx | XX | xx | xx | XX | XX | xx | xx |
| <b>IR (95% CI)</b><br>Thereof*** | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x–x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) |
| Infectious diseases | XX | | XX | XX | XX | | XX | XX | XX | XX |
| Neoplasms, malignant | xx | xx | xx.x (xx.x–x.x) | xx | XX | XX | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx | xx |
| Neoplasms, benign | xx | xx | xx.x (xx.x–x.x) | xx | xx | | xx | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx |
| Diseases of the blood | xx.x (xx.x–x.x) | , | xx.x (xx.x–x.x) | xx.x (xx.x–x.x)<br>xx | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x)<br>xx | xx.x (xx.x–x.x)<br>xx | xx.x (xx.x–x.x) |
| and blood-forming organs<br>Endocrine diseases | xx.x (xx.x–x.x) | | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x-x.x) | xx.x (xx.x–x.x) |
| | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x–x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |
| Psychiatric and neurological disorders | xx xx.x (xx.x-x.x) | xx<br>xx.x (xx.x–x.x) | xx<br>xx.x (xx.x–x.x) | xx<br>xx.x (xx.x–x.x) | xx xx.x (xx.x-x.x) | | xx<br>xx.x (xx.x–x.x) | xx<br>xx.x (xx.x–x.x) | xx<br>xx.x (xx.x–x.x) | xx.x (xx.x–x.x) |
| Eye | xx xx.x (xx.x-x.x) | | xx<br>xx.x (xx.x–x.x) | xx<br>xx.x (xx.x–x.x) | xx<br>xx.x (xx.x–x.x) | xx<br>xx.x (xx.x–x.x) | xx<br>xx.x (xx.x–x.x) | xx<br>xx.x (xx.x–x.x) | xx<br>xx.x (xx.x–x.x) | xx.x (xx.x-x.x) |
| Ear | xx<br>xx.x (xx.x–x.x) | xx<br>xx.x (xx.x–x.x) | xx<br>xx.x (xx.x–x.x) | xx<br>xx.x (xx.x–x.x) | xx<br>xx.x (xx.x–x.x) | xx<br>xx.x (xx.x–x.x) | xx<br>xx.x (xx.x–x.x) | xx<br>xx.x (xx.x–x.x) | xx<br>xx.x (xx.x–x.x) | xx<br>xx.x (xx.x–x.x) |
| Cardiovascular system | xx | xx | xx<br>xx.x (xx.x–x.x) | xx | xx | , | xx | xx<br>xx.x (xx.x–x.x) | xx | xx |
| Respiratory system | xx | xx | xx (xx.x-x.x) | xx | XX | xx | xx<br>xx.x (xx.x-x.x) | xx (xx.x-x.x) | xx | xx |



Supporting document SOP BMT 01.09 - Doc 5002.02 - Effective date 21.03.2017

| Digestive system | xx | XX | xx | XX | xx | xx | xx | xx | xx | xx |
|---|---|---|---|---|---|---|---|---|---|---|
| | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |
| Skin | XX | xx | xx | xx | XX | XX | XX | xx | xx | xx |
| | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |
| Musculoskeletal system | xx | xx | xx | xx | XX | xx | XX | xx | xx | xx |
| and connective tissue | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |
| Genitourinary system | xx | xx | XX | XX | XX | xx | XX | xx | xx | xx |
| | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |
| Pregnancy, delivery and | xx | xx | xx | xx | XX | xx | XX | xx | xx | XX |
| Puerperium | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |
| Injury, poisoning, | xx | xx | xx | xx | XX | xx | XX | xx | xx | XX |
| accidents etc. | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |

Note: \* Only women with 15 months or more of continuous EMT intake were considered. Incidence rates are calculated based on an observation time of 15 months or more

Note: \*\* Incidence rate is shown per 104 women years.

SAEs, which occurred within 3 months after stop of EMT, were attributed to the last EMT used by the women. Therefore, pregnancy-related SAEs in XXX cohorts does not necessarily reflect unwanted pregnancies during

Note: \*\*\* Women may appear in more than one category. ICD10 Codes Version 2009.

| Table C-3.4.2 | Incidence rate of serious adverse events by organ system for long-term use, AT population, Starter |
|---|---|
| Table C-3.4.3 | Incidence rate of serious adverse events by organ system for long-term use, AT population, Switcher |
| Table C-3.4.4 | Incidence rate of serious adverse events by organ system for long-term use, AT population, Restarter |
| Table C-3.4.5 | Incidence rate of serious adverse events by organ system for long-term use, AT population, Diagnosis confirmed by surgery |
| Table C-3.4.6 | Incidence rate of serious adverse events by organ system for long-term use, AT population, Diagnosis based on clinical symptoms |
| Table C-3.4.7 | Incidence rate of serious adverse events by organ system for long-term use, AT population, Germany |
| Table C-3.4.8 | Incidence rate of serious adverse events by organ system for long-term use, AT population, Poland |
| Table C-3.4.9 | Incidence rate of serious adverse events by organ system for long-term use, AT population, Hungary |



- Table C-3.4.10 Incidence rate of serious adverse events by organ system for long-term use, AT population, Switzerland
- Table C-3.4.11 Incidence rate of serious adverse events by organ system for long-term use, AT population, Russia
- Table C-3.4.12 Incidence rate of serious adverse events by organ system for long-term use, AT population, Ukraine



Supporting document SOP BMT 01.09 – Doc 5002.02 – Effective date 21.03.2017

### Section C-3.5 Incidence rate of malignant neoplasms by organ system

Table C-3.5.1 Incidence rate of malignant neoplasms by organ system, AT population, Complete cohort

| | DNG | | OAED | | NAED | | Ex-use | Allocation unknown | Total | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | GnRH-a | Danazol | All OAED | СНС | Other<br>progestin | All NAED | | | |
| Number of women years | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| Malignant neoplasms | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| IR* (95% CI) | xx.x (xx.x–x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x–x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x–x.x) |
| Breast | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |
| Cervix uteri | XX | xx | xx | XX | XX | xx | XX | xx | xx | XX |
| | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |
| Corpus uteri and uterus | xx | xx | xx | xx | XX | xx | XX | xx | xx | xx |
| unspecified | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |
| Ovary | xx | xx | xx | xx | XX | xx | xx | XX | xx | xx |
| | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |
| Fallopian tube | XX | XX | xx | XX | XX | xx | XX | xx | xx | XX |
| | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x-x.x) | xx.x (xx.x–x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |
| Vagina | XX | XX | xx | XX | XX | xx | XX | xx | xx | XX |
| | xx.x (xx.x–x.x) | xx.x (xx.x-x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x-x.x) | xx.x (xx.x–x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |
| Vulva | XX | XX | XX | XX | XX | | XX | XX | XX | XX |
| | xx.x (xx.x–x.x) | xx.x (xx.x-x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x-x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) |
| Unspecified genital | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x-x.x) | xx.x (xx.x–x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x–x.x) |
| Placenta | XX | | XX | XX | XX | XX | XX | XX | XX | XX |
| | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x-x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) |
| Subtotal of gyn. cancer | XX | XX | XX | XX | XX | XX | хх | XX | XX | XX |



Supporting document SOP BMT 01.09 – Doc 5002.02 – Effective date 21.03.2017

| | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | хх.х (хх.х–х.х) | xx.x (xx.x–x.x) | xx.x (xx.x-x.x) | хх.х (хх.х–<br>х.х) | xx.x (xx.x–<br>x.x) | хх.х (хх.х–х.х) |
|---|---|---|---|---|---|---|---|---|---|---|
| Lip, oral cavity and | xx | xx | xx | xx | xx | xx | xx | xx | XX | xx |
| pharynx | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |
| Digestive organs | xx | xx | xx | xx | XX | xx | xx | xx | xx | xx |
| | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |
| Respiratory and | xx | xx | xx | xx | XX | xx | xx | xx | xx | xx |
| intrathoracic organs | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |
| Bone and articular | XX | XX | XX | XX | XX | xx | XX | xx | xx | xx |
| cartilage organs | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |
| Skin | XX | XX | XX | XX | XX | xx | XX | xx | XX | xx |
| | xx.x (xx.x–x.x) | xx.x (xx.x-x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x-x.x) | xx.x (xx.x–x.x) | xx.x (xx.x-x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) |
| Mesothelial and | XX | XX | XX | XX | XX | xx | XX | XX | XX | XX |
| soft tissue | xx.x (xx.x-x.x) | xx.x (xx.x–x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x–x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x–x.x) |
| Urinary tract | XX | XX | xx | XX | XX | xx | XX | xx | XX | xx |
| | xx.x (xx.x-x.x) | xx.x (xx.x–x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x–x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x–x.x) |
| Eye, brain and other | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| parts of central<br>nervous system | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) |
| Thyroid and other | XX | XX | xx | xx | XX | xx | XX | xx | xx | xx |
| endocrine glands | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |
| III-defined, secondary | xx | XX | xx | XX | XX | xx | XX | xx | xx | xx |
| and unspecified sites | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |
| Lymphoid, | xx | XX | xx | XX | XX | xx | XX | xx | xx | xx |
| hematopoietic and related tissue | xx.x (xx.x-x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x-x.x) |
| Subtotal of none | хх | хх | хх | хх | хх | xx | хх | xx | хх | хх |
| gyn. cancer | xx.x (xx.x–x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x–<br>x.x) | xx.x (xx.x–<br>x.x) | xx.x (xx.x-x.x) |

Note: \* Incidence rate is shown per 10<sup>4</sup> women years.




| Table C-3.5.2 | Incidence rate of malignant neoplasms by organ system, AT population, Starter |
|---|---|
| Table C-3.5.3 | Incidence rate of malignant neoplasms by organ system, AT population, Switcher |
| Table C-3.5.4 | Incidence rate of malignant neoplasms by organ system, AT population, Restarter |
| Table C-3.5.5 | Incidence rate of malignant neoplasms by organ system, AT population, Diagnosis confirmed by surgery |
| Table C-3.5.6 | Incidence rate of malignant neoplasms by organ system, AT population, Diagnosis based on clinical symptoms |
| Table C-3.5.7 | Incidence rate of malignant neoplasms by organ system, AT population, Germany |
| Table C-3.5.8 | Incidence rate of malignant neoplasms by organ system, AT population, Poland |
| Table C-3.5.9 | Incidence rate of malignant neoplasms by organ system, AT population, Hungary |
| Table C-3.5.10 | Incidence rate of malignant neoplasms by organ system, AT population, Switzerland |
| Table C-3.5.11 | Incidence rate of malignant neoplasms by organ system, AT population, Russia |
| Table C-3.5.12 | Incidence rate of malignant neoplasms by organ system, AT population, Ukraine |



Supporting document SOP BMT 01.09 - Doc 5002.02 - Effective date 21.03.2017

### Section C-3.6 Incidence proportion of malformations

Table C-3.6.1 Incidence proportion of malformations, AT population, Complete cohort

| | DNG | | OAED | | | NAED | | Allocation<br>unknown | Total |
|---|---|---|---|---|---|---|---|---|---|
| | | GnRH-a | Danazol | All OAED | СНС | Other<br>progestin | All NAED | | |
| Number of deliveries | xx | xx | xx | xx | xx | XX | xx | xx | xx |
| Malformations | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| IP** (95% CI) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x–x.x) |
| Thereof last<br>endometriosis treatment<br>exposure | | | | | | | | | |
| At conception | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |
| One cycle before | xx | xx | xx | XX | XX | xx | XX | xx | xx |
| conception | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |
| More than one cycle | xx | xx | xx | XX | XX | xx | XX | xx | xx |
| before conception | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) |

Note: \* Cohort allocation is based on the intake of the last endometriosis treatment before delivery.

Note: \*\*Incidence proportion is shown per 10<sup>2</sup> deliveries.



| Table C-3.6.2 | Incidence proportion of malformations, AT population, Starter |
|---|---|
| Table C-3.6.3 | Incidence proportion of malformations, AT population, Switcher |
| Table C-3.6.4 | Incidence proportion of malformations, AT population, Restarter |
| Table C-3.6.5 | Incidence proportion of malformations, AT population, Diagnosis confirmed by surgery |
| Table C-3.6.6 | Incidence proportion of malformations, AT population, Diagnosis based on clinical symptoms |
| Table C-3.6.7 | Incidence proportion of malformations, AT population, Germany |
| Table C-3.6.8 | Incidence proportion of malformations, AT population, Poland |
| Table C-3.6.9 | Incidence proportion of malformations, AT population, Hungary |
| Table C-3.6.10 | Incidence proportion of malformations, AT population, Switzerland |
| Table C-3.6.11 | Incidence proportion of malformations, AT population, Russia |
| Table C-3.6.12 | Incidence proportion of malformations, AT population, Ukraine |



Supporting document SOP BMT 01.09 - Doc 5002.02 - Effective date 21.03.2017

Section C-3.7 Other outcomes of interest

Section C-3.8 Incidence rate of surgery / laparoscopy because of endometriosis

Section C-3.1 Incidence rate of surgery / laparoscopy because of endometriosis, ITT population, Complete cohort

| | DNG | | OAED | | | NAED | | Ex-use | Allocation unknown | Total |
|---|---|---|---|---|---|---|---|---|---|---|
| | | GnRH-a | Danazol | All OAED | СНС | Other<br>progestin | All NAED | | | |
| Number of women years | XX | XX | XX | xx | xx | xx | XX | XX | xx | xx |
| Diagnostic surgical | | | | | | | | | | |
| intervention | xx | xx | xx | xx | XX | xx | xx | xx | xx | xx |
| IR* (95% CI) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |
| Therapeutic surgery | xx | xx | xx | XX | xx | XX | XX | XX | xx | XX |
| (laparoscopic) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |
| Thereof | | | | | | | | | | |
| Excisions of lesions / | xx | xx | xx | xx | XX | xx | xx | xx | xx | xx |
| adhesions | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |
| Removal of ovarian | xx | xx | xx | XX | XX | xx | XX | xx | xx | xx |
| cysts | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |
| Removal of ovary / | xx | xx | xx | XX | XX | xx | XX | xx | xx | xx |
| fallopian tubes | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |
| Hysterectomy | xx | xx | xx | XX | XX | xx | XX | xx | xx | xx |
| Hysterectority | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |
| Other | xx | XX | xx | xx | XX | xx | xx | xx | xx | xx |
| Other | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x-x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |
| Therapeutic surgery | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| (open abdominal) Thereof | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x–x.x) |



Supporting document SOP BMT 01.09 – Doc 5002.02 – Effective date 21.03.2017

| Excisions of lesions / | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx |
|---|---|---|---|---|---|---|---|---|---|---|
| adhesions | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |
| Removal of ovarian | xx | xx | xx | XX | xx | xx | XX | XX | xx | xx |
| cysts | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |
| Removal of ovary / | xx | xx | xx | xx | XX | xx | xx | xx | xx | xx |
| fallopian tubes | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |
| I liveta va eta va. | xx | xx | xx | xx | XX | xx | xx | xx | xx | xx |
| Hysterectomy | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |
| Othor | xx | xx | xx | xx | XX | xx | xx | xx | xx | xx |
| Other | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |
| Therapeutic surgery | | | | | | | | | | |
| (other, incl type | xx | xx | xx | xx | XX | xx | xx | XX | xx | xx |
| unknown) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |
| Thereof | | | | | | | | | | |
| Excisions of lesions / | xx | xx | xx | xx | XX | xx | xx | xx | xx | xx |
| adhesions | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |
| Removal of ovarian | xx | xx | xx | xx | XX | xx | xx | XX | xx | xx |
| cysts | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |
| Removal of ovary / | xx | xx | xx | xx | XX | xx | xx | XX | xx | xx |
| fallopian tubes | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |
| I liveta va eta va. | xx | xx | xx | xx | XX | xx | xx | xx | xx | xx |
| Hysterectomy | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |
| Out | xx | xx | xx | xx | XX | xx | xx | xx | xx | xx |
| Other | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |

Note: \* Incidence rate is shown per 10<sup>4</sup> women years.



| Table C-3.8.2 | Incidence rate of surgery / laparoscopy because of endometriosis, AT population, Starter |
|---|---|
| Table C-3.8.3 | Incidence rate of surgery / laparoscopy because of endometriosis, AT population, Switcher |
| Table C-3.8.4 | Incidence rate of surgery / laparoscopy because of endometriosis, AT population, Restarter |
| Table C-3.8.5 | Incidence rate of surgery / laparoscopy because of endometriosis, AT population, Diagnosis confirmed by surgery |
| Table C-3.8.6 | Incidence rate of surgery / laparoscopy because of endometriosis, AT population, Diagnosis based on clinical symptoms |
| Table C-3.8.7 | Incidence rate of surgery / laparoscopy because of endometriosis, AT population, Germany |
| Table C-3.8.8 | Incidence rate of surgery / laparoscopy because of endometriosis, AT population, Poland |
| Table C-3.8.9 | Incidence rate of surgery / laparoscopy because of endometriosis, AT population, Hungary |
| Table C-3.8.10 | Incidence rate of surgery / laparoscopy because of endometriosis, AT population, Switzerland |
| Table C-3.8.11 | Incidence rate of surgery / laparoscopy because of endometriosis, AT population, Russia |
| Table C-3.8.12 | Incidence rate of surgery / laparoscopy because of endometriosis, AT population, Ukraine |



Supporting document SOP BMT 01.09 – Doc 5002.02 – Effective date 21.03.2017

### Section C-3.9 Incidence rate of self-reported anemia

Table C-3.9.1 Incidence rate of self-reported anemia, AT population, Complete cohort

| | DNG | | OAED | | | NAED | | Ex-use | Allocation<br>unknown | Total |
|---|---|---|---|---|---|---|---|---|---|---|
| | | GnRH-a | Danazol | All OAED | CC | Other<br>progestin | All NAED | | | |
| Number of women years | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| Self-reported anemia | xx | xx | xx | XX | xx | xx | xx | xx | xx | xx |
| IR* (95% CI) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |
| Thereof | | | | | | | | | | |
| Confirmed | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |
| Not confirmed | XX | XX | xx | xx | xx | xx | XX | xx | xx | xx |
| | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |
| Thereof | | | | | | | | | | |
| Recurrent anemia | xx | XX | xx | xx | XX | xx | XX | xx | xx | xx |
| | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |
| Potential anemia, | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| no further clarification possible | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x-x.x) | xx.x (xx.x–x.x) | xx.x (xx.x–x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x–x.x) |
| Anemia caused by | XX | xx | xx | xx | XX | xx | XX | xx | xx | xx |
| other reason** | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |
| Anemia not confirmed | XX | xx | xx | xx | XX | xx | XX | xx | xx | xx |
| by diagnostic measures | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |
| Anemia not treated by | XX | xx | xx | XX | XX | xx | XX | xx | xx | xx |
| НСР | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |
| "No event" - before | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| study, repetition | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |

Note: \* Incidence rate is shown per 10<sup>4</sup> women years.

Note: \*\* Includes e.g. other primary disease, surgery



Supporting document SOP BMT 01.09 – Doc 5002.02 – Effective date 21.03.2017

| Table C-3.9.2 | Incidence rate of self-reported anemia, AT population, Starter |
|---|---|
| Table C-3.9.3 | Incidence rate of self-reported anemia, AT population, Switcher |
| Table C-3.9.4 | Incidence rate of self-reported anemia, AT population, Restarter |
| Table C-3.9.5 | Incidence rate of self-reported anemia, AT population, Diagnosis confirmed by surgery |
| Table C-3.9.6 | Incidence rate of self-reported anemia, AT population, Diagnosis based on clinical symptoms |
| Table C-3.9.7 | Incidence rate of self-reported anemia, AT population, Germany |
| Table C-3.9.8 | Incidence rate of self-reported anemia, AT population, Poland |
| Table C-3.9.9 | Incidence rate of self-reported anemia, AT population, Hungary |
| Table C-3.9.10 | Incidence rate of self-reported anemia, AT population, Switzerland |
| Table C-3.9.11 | Incidence rate of self-reported anemia, AT population, Russia |
| Table C-3.9.12 | Incidence rate of self-reported anemia, AT population, Ukraine |



Supporting document SOP BMT 01.09 – Doc 5002.02 – Effective date 21.03.2017

### Section C-3.10 Incidence rate of self-reported depression

Table C-3.10.1 Incidence rate of self-reported depression, AT population, Compete cohort

| | DNG | | OAED | | | NAED | | Allocation<br>unknown | Total |
|---|---|---|---|---|---|---|---|---|---|
| | | GnRH-a | Danazol | All OAED | CC | Other<br>progestin | All NAED | | |
| Number of women years | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| Self-reported depression | xx | xx | xx | XX | xx | xx | XX | XX | XX |
| IR* (95% CI) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x–x.x) |
| Thereof | | | | | | | | | |
| Confirmed | xx | xx | xx | xx | xx | xx | xx | xx | XX |
| | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |
| Not confirmed | xx | xx | xx | xx | xx | xx | xx | xx | XX |
| | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x |
| Thereof | | | | | | | | | |
| Recurrent depression | xx | xx | xx | xx | xx | xx | xx | xx | XX |
| | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |
| Potential depression, | xx | xx | xx | xx | xx | xx | xx | xx | XX |
| no further clarification | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |
| possible | | | | | | | | | |
| Depression treated by | xx | xx | xx | XX | XX | xx | xx | xx | XX |
| GP | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |
| Depressive disorders | xx | xx | xx | XX | XX | XX | XX | xx | XX |
| treated by psychologist | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |
| Other psychiatric | xx | xx | xx | XX | XX | XX | XX | xx | XX |
| disorders** | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |
| Other psychic | xx | xx | xx | XX | XX | xx | xx | XX | xx |
| problems*** | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |
| "No event" - before | xx | xx | XX | xx | xx | xx | xx | XX | xx |
| study, repetition | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) | xx.x (xx.x-x.x) |



Supporting document SOP BMT 01.09 – Doc 5002.02 – Effective date 21.03.2017

Note: \* Incidence rate is shown per 10<sup>4</sup> women years.

Note: \*\* Includes e.g. schizophrenia, bipolar, anxiety, eating disorders.

Note: \*\*\* Includes e.g. mood changes, psychosomatic disorders, no HCP visited.

| Table C-3.10.2 Incidence rate of self-reported depression, AT population, Starter |
|---|
| Table C-3.10.3 Incidence rate of self-reported depression, AT population, Switcher |
| Table C-3.10.4 Incidence rate of self-reported depression, AT population, Restarter |
| Table C-3.10.5 Incidence rate of self-reported depression, AT population, Diagnosis confirmed by surgery |
| Table C-3.10.6 Incidence rate of self-reported depression, AT population, Diagnosis based on clinical symptoms |
| Table C-3.10.7 Incidence rate of self-reported depression, AT population, Germany |
| Table C-3.10.8 Incidence rate of self-reported depression, AT population, Poland |
| Table C-3.10.9 Incidence rate of self-reported depression, AT population, Hungary |
| Table C-3.10.10 Incidence rate of self-reported depression, AT population, Switzerland |
| Table C-3.10.11 Incidence rate of self-reported depression, AT population, Russia |
| Table C-3.10.12 Incidence rate of self-reported depression, AT population, Ukraine |

Supporting document SOP BMT 01.09 - Doc 5002.02 - Effective date 21.03.2017

### Section D Comparisons and Inferential Statistics of Primary Outcomes

#### Section D-1 New anemia and reoccurrence of anemia

Table D-1.1.1 Incidence rate ratio of new anemia and reoccurrence of anemia between EMT user cohorts, AT population

| Comparison | Cohort | No. of | WY | Incidence | Incidence Rate Ratio |
|---|---|---|---|---|---|
| Group | | events | | rate* | (95% CI) |
| | DNG | xx | xxxxx | x.xxxx | x.xxxx |
| 1 | OAED | xx | XXXXX | x.xxxx | (x.xxxx - x.xxxx) |
| 2 | DNG<br>NAED | xx<br>xx | xxxxx | x.xxxx<br>x.xxxx | x.xxxx<br>(x.xxxx - x.xxxx) |
| 3 | DNG | xx | xxxxx | x.xxxx | x.xxxx |
| 3 | Ex-use | XX | XXXXX | x.xxxx | (x.xxxx - x.xxxx) |

Note: \*Incidence rate per 10<sup>4</sup> women years



Supporting document SOP BMT 01.09 – Doc 5002.02 – Effective date 21.03.2017

Table D-1.1.2 Risk of new anemia and reoccurrence of anemia obtained from Cox model (HR), AT population

| Cohort | No. of | No. of WYs Incidence | | Hazard Ratio (95% CI) | |
|---|---|---|---|---|---|
| | events | | | Crude HR | Adjusted HR |
| DNG | xx | xxxxx | x.xxxx | x.xxxx | x.xxxx |
| OAED | XX | xxxxx | x.xxxx | (x.xxxx - x.xxxx) | (x.xxxx - x.xxxx) |
| DNG | xx | xxxxx | X.XXXX | x xxxx | X.XXXX |
| NAED | xx | xxxxx | x.xxxx | (x.xxxx - x.xxxx) | (x.xxxx - x.xxxx) |
| DNG | VV | | V VVVV | V VVVV | V |
| Ex-use | xx<br>xx | XXXXX | x.xxxx<br>x.xxxx | x.xxxx<br>(x.xxxx - x.xxxx) | x.xxxx<br>(x.xxxx - x.xxxx) |
| | DNG OAED DNG NAED | DNG XX DNG XX DNG XX DNG XX NAED XX | DNG XX XXXXX DNG XX XXXXX DNG XX XXXXX DNG XX XXXXX DNG XX XXXXX | DNG XX XXXXX X.XXXX OAED XX XXXXX X.XXXX DNG XX XXXXX X.XXXX NAED XX XXXXX X.XXXX DNG XX XXXXX X.XXXX | DNG XX XXXXXX XXXXXX XXXXXX OAED XX XXXXXX XXXXXX XXXXXX DNG XX XXXXXX XXXXXX XXXXXX NAED XX XXXXXX XXXXXX XXXXXX DNG XX XXXXXX XXXXXX XXXXXX |

Note: \*Adjusted for age, history of bleeding and history of anemia.



| Section D-2 | New depression or deterioration of existing depression |
|---|---|
| | Incidence rate ratio of new depression or deterioration of existing depression between EMT user cohorts, AT population Risk of new depression or deterioration of existing depression obtained from the Cox model (HR), AT population |
| Section D-3 | Treatment failure |
| Section D-3.1 | Incidence rate ratio of treatment failure between EMT user cohorts, AT population |
| Section D-3.2 | Risk of treatment failure obtained from the Cox model (HR), AT population |